

# **CLINICAL INVESTIGATIONAL PLAN**

# A RANDOMISED, CONTROLLED, OPEN-LABEL, MULTI-CENTRE STUDY TO EVALUATE THE EFFICACY OF FEETME® HOME-BASED REHABILITATION PROGRAM IN COMPARISON TO CONVENTIONAL PHYSIOTHERAPY IN PATIENTS WITH PARKINSON'S DISEASE USING CONNECTED INSOLES

Clinical investigational plan Number: 2023-A00150-45

Clinical investigational plan Version: Version 0.2

Date: May 2023

Principal Investigator: Prof DR Caroline MOREAU

Neurologue - CHRU de Lille

Directrice Medicale FeetMe

Sponsor: Feetme

157 bd MacDonald75019 Paris, France

#### **CONFIDENTIAL**

This clinical investigational plan is the property of FeetMe. The clinical investigational plan can only be applied in connection with the current clinical trial. No part of this document may be reproduced or utilised for any purpose other than the designated trial without prior written consent of FeetMe. This document is confidential and no information about its content may be disclosed to third parties not participating in the current trial.

#### 1 CLINICAL INVESTIGATIONAL PLAN APPROVAL SIGNATURES

#### Sponsor's Approval

Clinical investigational plan Number: 2023-A00150-45

Clinical investigational plan Title: A randomised, controlled, open-label, multi-center study to evaluate the efficacy of FeetMe® Home-Based rehabilitation program in comparison to conventional physiotherapy in patients with Parkinson's disease using connected insoles.

I agree with the content of this clinical investigational plan and the confidential nature of the documentation made as part of this study. I also acknowledge that the Investigator of the study has the right to discontinue the study at any time. I have read the clinical investigational plan, understand it, and will conduct the study in agreement with it and according to the principles of Good Clinical Practice, applicable laws and regulations and the Declaration of Helsinki.

#### Sponsor's representative

| Name: Arango-Lievano Margarita |
|--------------------------------|
| Title: Program Diretor |
| Address: Feetme |
| 157 bd MacDonald |
| 75019 Paris, France |
| Signature |
| Date |


#### Coordinating Principal Investigator's Approval

Clinical investigational plan Number: 2023-A00150-45

Clinical investigational plan Title: A randomised, controlled, open-label, multi-center study to evaluate the efficacy of FeetMe® Home-Based rehabilitation program in comparison to conventional physiotherapy in patients with Parkinson's disease using connected insoles.

I agree with the content of this clinical investigational plan and the confidential nature of the documentation made as part of this study. I also acknowledge that the Sponsor of the study has the right to discontinue the study at any time. I have read the clinical investigational plan, understand it, and will work in agreement with it and according to the principles of Good Clinical Practice, applicable laws and regulations and the Declaration of Helsinki.

#### **Coordinating Principal Investigator**

| Name: Caroline Moreau |
|-----------------------------------------------------|
| Title: Neurologist, FeetMe Chief Medical<br>Officer |
| Address: CHRU Lille |
| Signature |
| Date |

# 1 TABLE OF CONTENTS

| 1 | Table | of Contents | 4 |
|---|-------------|----------------------------------------|----|
| | List of fig | gures | 8 |
| | List of Ta | ables | 8 |
| 2 | List of | Abbreviations and Definitions of Terms | 9 |
| 3 | Synop | sis | 11 |
| 4 | Backg | ound Information | 19 |
| | 4.1 D | isease to be Assessed | 19 |
| | 4.1.1 | Parkinson's Disease | 19 |
| | 4.1.2 | Rehabilitation in Parkinson's Disease | 19 |
| | 4.2 S1 | tudy Background and Rationale | 20 |
| | 4.2.1 | Study Background | 20 |
| | 4.2.2 | Study Rationale | 20 |
| | 4.3 In | vestigational Medical Device | 21 |
| | 4.4 Fe | eetMe Rehabilitation Service | 21 |
| | 4.5 C | onventional physiotherapy | 23 |
| | 4.6 B | enefit-Risk Considerations | 23 |
| | 4.7 N | on-investigational Medical Device | 25 |
| 5 | Study | Objectives and Endpoints | 26 |
| | 5.1 A | ppropriateness of Measurements | 28 |
| 6 | Investi | gational Plan | 28 |
| | 6.1 St | audy design and rationale | 28 |
| | 6.2 Se | chedule of Assessments | 30 |
| | 6.3 St | udy Population | 33 |
| | 6.3.1 | Sample Size | 33 |
| | 6.3.2 | Inclusion Criteria | 33 |
| | 6.3.3 | Exclusion Criteria | 33 |
| | 6.3.4 | Patient Replacement | 34 |
| | 6.4 In | vestigational Medical Device | 34 |
| | 6.4.1 | Device Description | 34 |
| | 6.4.2 | Data collection | 35 |
| | Uniț | pedal parameters collected | 35 |
| | Bala | nce data and pressure data | 35 |
| | Exe | cises data | 35 |
| | 6.4.3 | Packaging and Labelling | 35 |

| | | nber 2023-A00150-45<br>rsion 0.2 | CONFIDENTIAL<br>May 2023 |
|---|---|---|---|
| | 6.4.4 | 4 Blinding | 36 |
| | 6.4.5 | 5 Supply and Accountability | 36 |
| 7 | Stud | dy Assessments by Visit | 37 |
| | 7.1 | Introduction and reflection period | 37 |
| | 7.2 | Screening | 37 |
| | 7.2.1 | 1.1 Screening | 37 |
| | 7.2.1 | 1.2 Randomisation | 37 |
| | 7.2.2 | 2 Re-Screening | 37 |
| | 7.2.3 | 3 Screen Failure | 37 |
| | 7.3 | Baseline Visit | 37 |
| | 7.4 | Primary Intervention Period | 38 |
| | 7.4.1 | 1 Remote Gait Monitoring 1 | 38 |
| | 7.4.2 | 2 Visits 1 and 2 | 39 |
| | 7.4.3 | 3 Visit 3 | 39 |
| | 7.5 | Long Term Intervention Period | 39 |
| | 7.5.1 | 1 Remote Gait Monitoring 2 | 40 |
| | 7.5.2 | 2 Visits 1.2 and 2.2 | 40 |
| | 7.5.3 | 3 Visit 4 | 40 |
| | 7.5.4 | 4 Remote Gait Monitoring 3 | 41 |
| | 7.6 | End of Study Visit | 41 |
| | 7.7 | Withdrawal / Early Termination Visit | 41 |
| 8 | Stud | dy Assessments | 41 |
| | 8.1 | Gait Assessments | 41 |
| | 8.1.1 | 1 6 Minutes Walk Test (6MWT) | 41 |
| | 8.1.2 | 2 Remote 6 Minutes Walk Test (6MWT) | 42 |
| | 8.1.3 | 3 Mini Balance Evaluation Systems Test (Mini-BESTest (Appendix L)) | ) 42 |
| | 8.2 | Medical History | 42 |
| | 8.3 | Prior- and Concomitant Medication | 42 |
| | 8.4 | Rehabilitation | 43 |
| | 8.5 | Device Deficiencies and Complaints | 43 |
| | 8.6 | Clinical Scales | 43 |
| | 8.6.1 | 1 Montreal Cognitive Assessment (MoCA) | 43 |
| | 8.6.2 | 2 Modified Hoehn and Yahr staging (mH&Y) | 44 |
| | 8.6.3<br>Dise | The Movement Disorder Society sponsored Revision of the Unified Pease Rating Scale (MDS-UPDRS) | Parkinson's 44 |
| | 8.6.4 | 4 Parkinson's Disease Questionnaire (PDQ-39) | 44 |
| | 8.6.5 | 5 Parkinson's Disease Questionnaire (PDQ-8) | 44 |

| CIP Numb<br>Final version | er 2023-A00150-45<br>on 0.2 | CONFIDENTIAL<br>May 2023 |
|---|---|---|
| 8.6.6 | Clinical Global Impression of Severity (CGI-S) | 45 |
| 8.6.7 | Patient Global Impression of Severity (PGI-S) | 45 |
| 8.6.8 | Clinical Global Impression of Improvement (CGI-I) | 45 |
| 8.6.9 | Patient Global Impression of Improvement (PGI-I) | 45 |
| 8.6.10 | Parkinson Disease Sleep Scale 2 (PDSS-2) | 45 |
| 8.6.11 | Pain Visual Analog scale (VAS) | 46 |
| 8.6.12 | 2 Freezing of gait questionnaire (FOG-Q) | 46 |
| 8.7 F | Falls Diary | 46 |
| 8.8 | Conventional Physiotherapy tracking | 46 |
| 8.9 S | Safety Assessments | 46 |
| 8.9.1 | Adverse Events | 46 |
| 8.9.2 | Serious Adverse Events (SAE) | 46 |
| 8.9.3 | AEs of Special Interest | 47 |
| 8.9.4 | Adverse Device Effect (ADE) | 47 |
| 8.9.5 | Serious Adverse Device Effect (SADE) | 47 |
| 8.9.6 | Assessment Definitions | 47 |
| 9 Statist | tical Methods and Considerations | 49 |
| 9.1 A | Analysis sets | 49 |
| 9.1.1 | Usage of the analysis sets | 49 |
| 9.1.2 | Short description of endpoints and time periods | 49 |
| 9.2 I | Description of statistical analysis | 49 |
| 9.2.1 | Estimands for primary and key secondary objectives | 49 |
| 9.2.2 | Overall testing strategy | 50 |
| 9.2.3 | Analysis of the primary efficacy outcome | 51 |
| 9.2.4 | Analysis of the key secondary efficacy outcome | 51 |
| 9.2.5 | Analysis of other secondary efficacy outcomes | 51 |
| 9.2.6 | Analysis of exploratory efficacy outcomes | 51 |
| 9.2.7 | Analysis of safety outcomes | 51 |
| 9.3 I | nterim analysis | 51 |
| 9.4 I | Determination of sample size | 51 |
| 9.5 S | Statistical analysis | 52 |
| 9.5.1 | Analysis for the primary endpoint | 52 |
| 9.5.2 | Analysis for the secondary endpoints | 53 |
| 9.5.3 | Exploratory analysis | 53 |
| 10 Data I | Handling | 54 |
| 10.1 I | Data Monitoring Committee | 54 |
| 10.2 | Gait Data Collection and Management | 54 |

| CIP Number 2023-A00150-45<br>Final version 0.2 | CONFIDENTIAL<br>May 2023 |
|---|---|
| 10.3 Clinical Data Collection and Monitoring | 54 |
| 10.4 Record Retention | 54 |
| 10.5 Reporting and Publication | 55 |
| 11 Quality Assurance and Quality Control | 56 |
| 12 Ethics | 56 |
| 12.1 Independent Ethics Committee or Institutional Review Board | d 56 |
| 12.2 Regulatory Authorities | 56 |
| 12.3 Ethical Conduct of the Study | 56 |
| 12.4 Informed Consent | 56 |
| 12.5 Patient Confidentiality | 57 |
| 12.6 Data Protection | 57 |
| 12.7 Financing and Insurance | 57 |
| 13 Study Personnel and Administrative Structure | 58 |
| 14 Appendices | 59 |
| 14.1 Appendix A – Rehabilitation Exercises | 59 |
| 14.1.1 Static Exercises | 59 |
| 14.1.1.1 Balance | 59 |
| 14.1.1.2 Muscle strengthening | 59 |
| 14.1.2 Dynamic Exercises | 60 |
| 14.1.2.1 Gait Quality | 60 |
| 14.1.2.2 Endurance | 60 |
| 14.2 Appendix B – Rehabilitation Program | 61 |
| 14.2.1 Decision Tree for Initial Program | 61 |
| 14.2.2 Program Adaptation Principles | 62 |
| 14.2.3 Program A | 63 |
| 14.2.4 Program B | 63 |
| 14.2.5 Program C | 63 |
| 14.3 Appendix C – FeetMe Satisfaction Questionnaire for Initial l | Patient Training 64 |
| 14.4 Appendix D – FeetMe Satisfaction Questionnaire – Patient V | Version 65 |
| 14.5 Appendix E – Satisfaction Questionnaire – Investigator Vers | sion 67 |
| 14.5.1 Application FeetMe Evaluation application et semelles | FeetMe Monitor 67 |
| 14.6 Appendix F – Conventional Physiotherapy Tracking Sheet | 70 |
| 14.7 Appendix G – Falls Diary | 72 |
| 14.8 Appendix H – Visual analog scale | 74 |
| 14.9 Appendix I – Parkinson disease questionnaire-39 | 75 |
| 14.10 Appendix J – Parkinson disease questionnaire 8 | 81 |
| 14.11 Appendix K – MOCA | 83 |

| CIP Number 2023-A00150-45<br>Final version 0.2 | CONFIDENTIAL<br>May 2023 |
|---|---|
| 14.12 Appendix L – MiniBEST | 84 |
| 14.13 Appendix M – MDS-UPDRS | 87 |
| 14.14 Appendix N – Hoehn and Yahr stage | 104 |
| 14.15 Appendix O – Freezing of gait questionnaire. | 105 |
| 14.16 Appendix P – PDSS 2 | 107 |
| 14.17 Appendix Q – Patient global impression of severity (PGI-S) and impro | ovement (PGI-I) 108 |
| 14.17.1 PGI-S: patient global impression of severity | 108 |
| 14.17.2 PGI-I: patient global impression of improvement | 108 |
| 14.18 Appendix R – Clinical global impression of severity (CGI-S) and impr | ovement (CGI-I) 109 |
| 14.18.1 Clinical global impression of severity | 109 |
| 14.18.2 Clinical global impression of improvement | 109 |
| 14.19 Appendix S – User guides | 110 |
| 14.19.1 User guide for patient in the conventional physiotherapy arm | 110 |
| 14.19.2 User guide for patient in the FeetMe Rehabilitation arm | 111 |
| 15 References | 114 |
| List of figures | |
| Figure 1. Example of a rehabilitation program - Program A | 24 |
| Figure 2. Rehabilitation Program Follow up schedule | 25 |
| Figure 3. Schematic of the study design Figure 4. Picture of a FeetMe Insole with charger and related smartphone applica | 32<br>ation 39 |
| List of Tables | |
| Table 5.1 Study Objectives and Endpoints | 27 |
| Table 6.1 Schedule of Assessments Table 9.1 Combination of patient cohorts, patient treatment groups and analysis s | 33<br>sets 58 |
| Table 9.1 Treatment policy estimands for the primary and key secondary objective | |
| Table 9.3 Hypothetical estimands for primary and key secondary objectives | 59 |
| Table 9.4 Number of patients per arm for various scenarios | 62 |

# 2 LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| 6MWT | 6 Minutes Walk Test |
|-----------|------------------------------------------------|
| ADE | Adverse Device Effect |
| ADL | Activities of Daily Living |
| AE | Adverse Event |
| ANOVA | Analysis of Variance |
| BL | Baseline |
| BMI | Body Mass Index |
| CGI-I | Clinical Global Impression of Improvement |
| CGI-S | Clinical Global Impression of Severity |
| cm/s | Centimeters per second |
| CP or CPt | Conventional Physiotherapy |
| CRA | Clinical Research Associate |
| CRO | Clinical Research Organization |
| DT | Dual Task |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| ePRO | Electronic Patient Reported Outcome |
| FDA | Food and Drug Administration |
| FM | FeetMe Rehabilitation |
| FNA | FeetMe Rehabilitation No Access |
| FOG | Freezing Of Gait |
| FOG-Q | Freezing of gait questionnaire |
| GAD-7 | Global Anxiety Disorder Questionnaire |
| GCP | Good Clinical Practice |
| H&Y | Hoehn and Yahr staging |
| HAS | Haute Autorité de Santé |
| HS | Heel Strike |
| ICF | Informed Consent Form |
| IEC | Independent Ethical Committee |
| IMU | Inertial Measurement Unit |
| IRB | Institutional Review Board |
| ISO | International Organization for Standardization |
| IxRS | Interactive Voice/Web Response System |
| LARS | The Lille Apathy Rating Scale |

| LPLO | Last Patient Last Observation |
|---|---|
| LSVT | Lee Silverman Voice Treatment |
| MDS-UPDRS | The Movement Disorder Society sponsored Revision of the Unified Parkinson's Disease Rating Scale |
| MiniBESTest | Mini Balance Evaluation Systems Test |
| MoCA | Montreal Cognitive Assessment |
| NA | Not Applicable |
| NI | Non Intervention |
| NSAE | Non-serious Adverse Event |
| PD | Parkinson's Disease |
| PDQ-39 | Parkinson's Disease Questionnaire |
| PDQ-8 | Parkinson Disease Questionnaire short form |
| PDSS2 | Parkinson Disease Sleep Scale 2 |
| PGI-I | Patient Global Impression of Improvement |
| PGI-S | Patient Global Impression of Severity |
| PGI-S | Patient Global Impression of Severity |
| QIDS SR | Quick Inventory of Depressive Symptomatology, self-report questionnaire |
| SADE | Serious Adverse Device Effect |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SE-ADL | Schwab and England Activities of Daily Living |
| SoA | Schedule of Assessments |
| ТО | Toe Off |
| VAS | Visual Analog Scale |

## 3 SYNOPSIS

| GRONGOR | |
|---|---|
| SPONSOR: | CLINICAL INVESTIGATIONAL PLAN NUMBER: |
| FeetMe | |
| TITLE | A randomised, controlled, open-label, multi-centre study to evaluate the efficacy of FeetMe® home-based rehabilitation program in comparison to conventional physiotherapy in patients with Parkinson's Disease using connected insoles. |
| ACRONYM | RE-CONNECT |
| NAME OF DEVICES | FeetMe Monitor (insoles) and FeetMe Rehabilitation (application) |
| RATIONALE | Parkinson's disease (PD) is characterised by a range of motor- and non-motor symptoms which define the quality of life (QoL) of the PD patients. Physical rehabilitation is an essential part of the care complementing pharmacological treatment and it is recommended by the French Health Authority (Haute Autorité de Santé [HAS]) to support disease management. Despite demonstrated benefits of rehabilitation programs on gait and balance and consequently on risk of falls and QoL, only a fraction of PD patients benefit from conventional physiotherapy (CPt) due to multiple factors including the limited number of practices and rising demand. Thus, identifying an effective rehabilitation program that is readily accessible for PD patients remains a pressing unmet need. FeetMe Rehabilitation is an innovative technology solution that combines connected insoles with a mobile application containing rehabilitation exercises specific for PD patients, focusing on endurance, muscle strength and postural stability. The device is complemented by a remote rehabilitation service provided by a rehabilitation professional to follow progression and to adapt training needs based on results. Since patients can train remotely and in their home environment, FeetMe Rehabilitation ensures equal access to this essential therapy, which is currently strongly limited by local availability of rehabilitation centres and personnel. |
| | This study aims to evaluate the effectiveness of the FeetMe home-based rehabilitation program compared to CPt in participants with PD. The outcome measures of efficacy are defined according to the expected benefits of improving gait and balance, number of falls and QoL. |
| OBJECTIVES | Primary Objective |
| | To evaluate the efficacy of FeetMe home-based rehabilitation program compared to conventional physiotherapy at Week 12 in PD patients assessed by gait velocity. |
| | Key Secondary Objective |

| | To evaluate the efficacy of FeetMe home-based rehabilitation program compared to conventional physiotherapy at Week 12 in PD patients assessed by stance time variability. |
|---|---|
| | Secondary Objectives |
| | To evaluate the efficacy of FeetMe home-based rehabilitation program compared to conventional physiotherapy at Week 12 in PD patients assessed by: |
| | • rate of falls |
| | standard gait and balance exercises |
| | MDS-UPDRS Part III |
| | • quality of life |
| | <b>Exploratory Objectives</b> |
| | • To explore the long-term efficacy of FeetMe home-based rehabilitation program compared to conventional physiotherapy in patients who continue to Week 24. |
| | • To explore the maintenance of the effect after 3 months in patients who stop physiotherapy at Week 12. |
| | • To explore the efficacy in patients who switch from one treatment to the other at Week 12. |
| | • To explore the compliance with training, acceptability, and patient's engagement throughout the study. |
| | To explore the satisfaction with the service. |
| | • To explore the safety of FeetMe home-based rehabilitation program. |
| PLANNED<br>DURATION | The estimated recruitment period is approximately 18 months. The total duration of the study for each patient will be up to 26.5 weeks divided as follows: |
| | Screening: up to one month |
| | Primary Intervention period: 12 weeks |
| | Long Term Intervention Period: 12 weeks |
| | The end of the study is defined as the date when the last participant's last observation (LPLO) occurs, upon completion of the End of Study Visit. |
| SITES | 6 sites (Nîmes, Nice, Nantes, Toulouse, Lille and Avicennes) |
| POPULATION | All patients must fulfil the following criteria: |
| | Inclusion criteria |
| | 1. Written informed consent to participate in the study. |
| | 2. Male or female patients between 40 to 70 years of age, inclusive. |

- 3. Body weight range of 40 kg to 120 kg and a body mass index (BMI) of 18 to 34 kg/m2.
- 4. Diagnosis of Idiopathic Parkinson's disease (PD) according to UK Brain Bank Criteria (2/3 symptoms), with Hoehn and Yahr (H&Y) staging level 2, 2.5 or 3.
- 5. Disease onset of at least 3 years prior to enrolment.
- 6. Patients with a history of 50% of levodopa responsiveness based on motor signs.
- 7. On stable treatment of PD medication for at least 30 days before screening and with no expected major changes during the first 3 months of the study.
- 8. Prescription for physiotherapy available.
- 9. Ability to walk without aid for at least 6 minutes.
- 10. Shoe size between 35 46 (European Standard).
- 11. Intact skin on feet.
- 12. Adequate visual and auditory acuity to perform the rehabilitation program and the assessments in the Investigator's judgement.
- 13. Comfortable with the use of a smartphone. If assistance is required for the use of FeetMe technology, a caregiver or volunteer is fully available to assist the patient.
- 14. Willingness to be regularly contacted via phone-calls.
- 15. Willingness to suspend conventional physiotherapy treatment and start the FeetMe rehabilitation program, if applicable.
- 16. French speaker.

Patients must **not** fulfil the following criteria:

#### **Exclusion criteria**

- 1. Medical history indicating a Parkinsonian syndrome other than idiopathic PD.
- 2. Unable to walk without walking aid or presence of an injury preventing the patient to walk.
- 3. Any relevant comorbidity or vestibular/visual dysfunctions limiting locomotion or balance.
- 4. Clinically significant comorbidities which in the judgement of the investigator may preclude the reliable gait assessment of the patient.
- 5. Patients with poor wound healing or broken skin on the feet.
- 6. Patients with foot implants.
- 7. Montreal Cognitive Assessment (MoCA) score  $\leq 24/30$ .
- 8. Patients with dementia.
- 9. Patients with apathy.

- 10. Participation in another clinical trial with an investigational drug/ therapeutic within the three months before screening and during the study, unless agreed by the Sponsor.
- 11. Patients who had Lee Silverman Voice Treatment (LSVT) Big therapy within the past 12 months or have it planned during the course of the study.
- 12. Patients with Deep Brain Stimulation planned during the first 12 weeks of the study.
- 13. Patients with pacemakers.
- 14. Patients performing vigorous exercise > three times a week, 30 mins or more per session.

# STUDY DESIGN AND ASSESSMENTS

This is a multicentre, controlled, randomised in two parallel-groups, open-label, study designed to evaluate the efficacy of FeetMe home-based self-rehabilitation program in comparison to conventional physiotherapy, including no physiotherapy in patients with PD. The study consists of a screening period, a primary intervention period of 12 weeks and a long-term intervention period of 12 weeks.

#### **Screening**

During their routinely scheduled visit at the investigational site patients who express interest in participating in the study will be introduced to the device. If judged to be comfortable with and interested in the technology, patients will return to their home to consider their participation. There is a reflexion period that lasts at least fifteen days up to one month If the patient decides to participate in the study, they return to the site for the screening visit. Once the informed consent is signed the screening assessments will be performed by the investigator (the neurologist). If eligible, the patients will be randomised either into the conventional physiotherapy (CPt control group) or the FeetMe rehabilitation program (experimental group).

#### **Primary Intervention Period**

Once randomised patients will proceed to the Baseline Visit (BL). At the BL visit, all participants (experimental and CPt control group) will be trained to use the FeetMe devices and will wear the insoles as much as possible throughout the visit. Standard gait and balance assessments will performed (6 minute be walk test (6MWT), MiniBESTest). Additionally, patients will perform multiple clinical assessments designed to assess: disease severity, gait, balance, mobility, etc. by completing different surveys.

Following the BL visit, all patients will enter an initial 12 week period according to their patient group. Every patient in the study will be provided with a pair of insoles and will take the device to their homes. All patients, whatever the group of randomisation, will be asked to wear them as much as possible for 14 days after the BL visit to allow continuous gait data collection. This will permit the gathering of extensive data on a considerable number of gait parameters in a more familiar and natural setting reflecting real-life conditions. The FeetMe

patients will then continue to use the insoles according to the FeetMe rehabilitation program schedule.

During the Primary Intervention Period (PIP), all patients will participate in two remote visits: Visit 1 (four weeks after BL) and Visit 2 (eight weeks after BL). During these visits, all patients will perform a short battery of self-reported questionnaires.

At the end of the 12 week PIP, all patients will participate in a visit at their respective study centres (Visit 3). During the visit, they will perform the same gait and clinical assessments as during the BL visit allowing to record primary and secondary outcomes.

#### Open Label Extension period

Following Visit 3, patients will be asked whether they want to:

a) continue with their already assigned treatment;

Patients will continue with their respective rehabilitation programs.

b) switch to the other arm;

If patients on the conventional physiotherapy arm would like to start the FeetMe program they will be trained to use the devices and will start their 12 weeks program. Patients of FeetMe group wanting to switch from FeetMe to CPt will need to arrange the care themselves. Patients who switch will have the same visit schedule as during the first three months.

c) discontinue rehabilitation.

If a patient would like to discontinue rehabilitation they will still be asked to remain in the study for further data collection.

At Visit 3 every patient will again be provided with a pair of insoles to take to their homes. All patients will be asked to wear them as much as possible for 14 days. Patients on the FeetMe arm will also use their device according to their program schedule.

At the end of the second 12 weeks rehabilitation, all patients will participate in an additional in-clinic visit (Visit 4) at their respective study centres. During this visit, they will perform the same gait and clinical assessments as in the BL visit and Visit 3, wearing the insoles as much as possible throughout the visit. Following Visit 4, all patients will again take the insoles home to participate in an additional two-week remote gait monitoring.

All assessments performed at the designated visits by the patient must be performed in the ON-State.

Once the core 26 week period of the study is completed, an End of Study visit will be scheduled remotely and the patient's participation in the study will be considered concluded.

Based on the emerging data, the Sponsor may decide to ensure that participants have the option to continue or take part in the FeetMe rehabilitation program. Such extension will be described in a separate document.

#### **ENDPOINTS**

#### **Primary Endpoint**

Change from baseline to Week 12 (Visit 3) in gait velocity (cm/s) assessed during the 6 Minutes Walk-Test (6MWT).

#### **Key Secondary Endpoint**

Change from baseline to Week 12 (Visit 3) in Stance Time Variability assessed during the 6MWT.

#### **Secondary Endpoints**

- Rate of falls at Week 12 based on the results of the falls diary.
- Change from baseline to Week 12 (Visit 3) in the asymmetry of the swing duration assessed during the 6MWT.
- Change from baseline to Week 12 (Visit 3) in the Mini-BESTest.
- Change from baseline to Week 12 (Visit 3) in Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III sub-score.
- Change from baseline to Week 12 (Visit 3) in the results of the Parkinson Disease Questionnaire (PDQ-39).

#### **Exploratory Endpoints**

- Rate of falls at Week 24 based on the results of the falls diary.
- Change from Baseline to Week 24 (Visit 4) and from Week 12 (Visit 3) to Week 24 in:
  - Gait velocity (cm/s) assessed during the 6MWT
  - Stance Time Variability assessed during the 6MWT
  - Asymmetry of the swing duration assessed during 6MWT
  - the Mini-BESTest
  - MDS-UPDRS Part III sub-score
  - the results of the PDQ-39
- Change from Baseline to Week 12 (Visit 3) and to Week 24 (Visit 4) and from Week 12 to Week 24 in the:
  - gait parameters measured by the FeetMe Monitor during the 6MWTs other than ones of the primary and secondary endpoints
  - gait parameters measured by the FeetMe Monitor during remote gait monitoring
  - results of the pain VAS
  - results of the Parkinson Disease Sleep Scale 2 (PDSS2)
  - results of the Clinical and Patient Global Impression of Severity scales (CGI/PGI-S)
  - results of the Clinical and Patient Global Impression of Improvement scales (CGI/PGI-I)
- results of the MDS-UPDRS I, II and IV sub scores
- Actual versus prescribed time spent on physiotherapy at Week 12 and Week 24.

| Results of the Patient and Investigator satisfaction questionnaire. |
|---|
| • Number of device and protocol procedure related adverse events at Week 12 and at Week 24. |
| N=150 |
| The main objective of the RE-CONNECT study is to demonstrate the efficacy of FeetMe home-based rehabilitation program compared to conventional physiotherapy at Week 12 in PD patients. The primary endpoint is the change from baseline to Week 12 in gait velocity (cm/s) assessed during the 6 Minutes Walk-Test (6MWT). The sample size computation is based on the study of Chris J Hass et al. (Hass et, al, 2014.) aiming to determine the Minimal Clinically Important Difference (MCID) for the gait velocity in patients with idiopathic Parkinson's disease. In this study including 324 patients, MCID for gait velocity was classified as small, moderate and large with values of 6 cm/s, of 14 cm/s and 22 cm/s respectively (using a distribution-based analysis and the categorization defined by Cohen (Cohen et al, 1988)). We aim to show that the Feetme rehabilitation procedure will allow to improve the change in gait speed at least in a moderate range in comparison with that in standard rehabilitation group and we set the difference to be detected at 14cm/s. In the Chris J Hass et al, the standard deviation of gait velocity was estimated at 27 cm/s. To detect a difference of 14cm/s between the two groups for the change in velocity with a standard deviation of 27 cm/s for the change from baseline to Week 12 in gait speed (assuming a conservative correlation coefficient of 0.5 between the measures at baseline and at week 12), 60 patients per group are needed (two-sided Student's test, type I error of 0.05 and a power of 80%). To take into account a 20% rate of drop out for the measurement of the gait velocity at week 12 (15% of lost to follow up and 5% of deaths or injuries), we plan to recruit 75 patients per group (a total of 150 patients). |
| The primary outcome (the change in the gait velocity between baseline and week 12, assessed during the 6 Minutes Walk-Test) will be estimated and compared between Feetme rehabilitation and conventional physiotherapy groups using the constrained longitudinal data analysis (cLDA) model proposed by Liang and Zeger, including centre as random effect and adjusted for the covariable "already in rehabilitation" considered as stratification factor in the randomisation. The betweengroup mean differences in 12-week change in gait velocity will be estimated by the time-by-arm interaction as treatment effect size. The assumptions of the cLDA model will be checked. We will use the analysis of cDLA model residuals by examining graphically the normality of residuals (histogram and Quantile-quantile plot) and by using the Shapiro Wilk test. In case of strong departure from the normality assumptions (even after applying a logarithmic transformation), nonparametric analysis will be used as recommended by Vickers et al.; absolute changes between baseline and 12-week will be calculated and compared between the 2 treatments groups using non-parametric analysis of covariance |

g (standardized differences) computed on rank transformed data with its

| | 95% confidence interval (using the method based on noncentral Student distribution which is a corrected version of Cohen's d taking into account the sample size). |
|---|---|
| BENEFIT/RISK<br>CONSIDERATIONS | A risk analysis was carried out in accordance with ISO 14971 to identify the potential risks associated with the FeetMe Rehabilitation device. The residual risks are all at an acceptable level. |

#### 4 BACKGROUND INFORMATION

#### 4.1 Disease to be Assessed

#### 4.1.1 Parkinson's Disease

Parkinson's Disease (PD) is the second most common neurodegenerative disorder after Alzheimer's disease and is characterised by a variety of motor and non-motor symptoms, including bradykinesia, rigidity, gait disorders, tremor and falls. PD is pathologically characterised by the presence of Lewy bodies, composed of aggregated and phosphorylated alpha-synuclein in the subcortical regions of the brain (Spillantini et al., 1997). Nevertheless, the underlying causes of neuronal death and alpha-synuclein deposits are still unknown and subject to intense study (Poewe et al., 2017). PD has an incidence of 5-35 cases per 100,000 individuals, with an overall estimated global prevalence of 0.3%, increasing sharply up to 3% when considering people over 80 years of age (Poewe et al., 2017). PD has an adult onset and it is rarely diagnosed before the sixth decade of life; its incidence in the population however increases dramatically starting from that time point (Van Den Eeden et al., 2003).

Idiopathic PD is characterised by a continuous progression of clinical symptoms and can be preceded by a prodromal phase lasting years or even decades, defined by a specific set of non-motor symptoms such as Rapid Eye Movement (REM) sleep behaviour disorder, depression, constipation, and anxiety. At their onset, motor symptoms are usually unilateral, an asymmetry usually persists through the course of the disease. Bradykinesia, rigidity, and tremor are the typical motor abnormalities of early-stage PD, leading the patient to seek medical attention and guiding the first diagnosis. As the disease progresses, more debilitating symptoms emerge, as motor fluctuations (on/off phases) and dyskinesias manifest (Poewe et al., 2017). Slow walking is a common manifestation of PD that negatively affects patients' performance in daily living activities (Mehrholz et al., 2016; Muslimović et al., 2008). Among the most burdensome characteristics of late-stage PD are instability of posture and gait abnormalities, oftentimes causing falls that can be quite harmful, frequently leading to hospitalisation and reduction in life expectancy ((Verghese et al., 2009, Fasano et al., 2017). Some studies reported that approximately 35% to 90% of PD patients fall at least once a year, with an average rate of 60.5% (Fasano et al., 2017; Pickering et al., 2007; Wood et al., 2002). In another work, it was estimated that roughly 39% of patients sustain multiple falls and fall-related injuries over one year (Allen et al., 2013). Given the high rate of falls during walking in people with PD and the significant burden they impose on quality of life as well as on the health care system, identifying individuals at higher risk and developing rehabilitation programs to reduce such risk is crucial. Motor symptoms are also supplemented by a set of non-motor manifestations which can greatly affect the quality of life of the patients, such as pain, cognitive impairment, apathy and autonomic dysfunction (Chaudhuri and Schapira, 2009).

Motor symptoms of PD develop quite rapidly if untreated. However, the introduction of Levodopa has greatly prolonged the progression time and it could take up to 15 years until the patient is in need of extensive assistance from their caregiver (Poewe, 2006). The mortality ratio in PD patients is between 1.5 and 2.5 times higher than the normal population. The average survival from symptoms onset is 10 years; however, these values are highly dependent on the age at onset and on the individual course of the disease.

#### 4.1.2 Rehabilitation in Parkinson's Disease

The clinical management of PD has traditionally been centred on drug-based therapy (i.e. Levodopa) and surgical approaches (i.e., deep brain stimulation). Nonetheless, despite the undeniable usefulness of such treatments, PD patients still experience progressive motor deterioration and disability largely due to gait, balance and posture impairments (Abbruzzese et al., 2016).

A growing body of evidence highlights the effectiveness of physical therapy in PD and its positive effects on both motor and non-motor complications of PD (Abbruzzese et al., 2016; Tomlinson et al., 2013; van der Kolk and King, 2013). Due to these promising results and the amelioration of quality of

life, physiotherapy rehabilitation programs are currently considered an essential component of the management of patients with PD.

Importantly, rehabilitation was shown to have a positive effect on the risk of fall in a large metanalysis study (Shen et al., 2016), showing a significant overall fall rate reduction over both the short and long term, and supporting the application of exercise training to improve balance and gait ability and ultimately prevent falls in people with PD.

Although the evidence for a positive effect of physiotherapy rehabilitation treatments in PD is increasingly clear, some open questions remain to be further explored. One such question is which type of intervention yields the best results, and for how long the effect persists. Recent studies have shown that some forms of exercise such as balance training, gait training or complementary techniques such as Tai Chi can improve balance and mobility, as well as reduce fall frequency for up to six months after the end of training (Mak et al., 2017). This promising evidence highlights the necessity for structured and regular regimens of physiotherapy rehabilitation for every PD patient, a pressing need that is still unmet, due to the limited availability of physiotherapy practices (Benayoun et al., 2019) and the insufficient access to such services in remote and rural areas (Deane et al., 2002). Consequently, remote and web-based solutions for rehabilitation such as the one offered in this study can close this crucial gap and deliver this indispensable service in a capillary way.

#### 4.2 Study Background and Rationale

#### 4.2.1 Study Background

In France, physiotherapy is recommended by the French Health Authority (Haute Autorité de Santé [HAS]) to all PD patients to slow down the evolution of posture and motor disabilities (Haute Autorité de Santé, 2016). However, despite demonstrated benefits of rehabilitation programs in PD on gait parameters and several other aspects of life, only a fraction of PD patients are able to actually benefit from conventional physiotherapy rehabilitation sessions (Deane et al., 2002). This is due to the limited number of practices unable to meet the rising demand, as well as to their insufficient geographical coverage, de facto excluding patients residing in rural and remote areas (Benayoun et al., 2019). Recent data from the French Institute of Research and Statistics (Direction de la recherche, des études, de l'évaluation et des statistiques [DREES]) shows that up to 33% of the population in France resides in a municipality lacking a physiotherapy practice (Vergier and Chaput, 2017). Moreover, the recent COVID-19 pandemic has highlighted the fragility of the rehabilitation system for PD patients as it currently stands, with many countries discontinuing their in-person rehabilitation services during regional or national lockdowns (Bettger et al., 2020), often resulting in a total absence of physical activity (Cavallieri et al., 2021) and causing significant negative impacts on the functional abilities of PD patients (Braun et al., 2021). Telemedicine or remote rehabilitation services are therefore currently being considered to complement or as an alternative to in-person practices to overcome such limitations (Barbour et al., 2016; Vellata et al., 2021).

In this context, FeetMe Rehabilitation is an innovative technology combining connected insoles with a mobile application and a web platform to facilitate education and training on gait and mobility specifically for PD patients. Additionally, since patients can train in their home environment, FeetMe Rehabilitation ensures equal access to this essential service, overcoming constraints due to the place of residence of patients and the availability of rehabilitation centres in their area, therefore fulfilling the increasingly unmet need for physiotherapy in this patient population.

#### 4.2.2 Study Rationale

The use of wearables and their applications to remote care could complement the conventional medical practice in PD, creating a more pervasive and capillary distribution of rehabilitative care. The FeetMe devices are expected to have their major advantage by being able to encompass areas and segments of the population that traditional care cannot efficiently reach. The FeetMe home-based rehabilitation

program with it's targeted battery of rehabilitation exercises and personalised patient follow-up service has the long-term objective of slowing down disease progression, aims at improving patient mobility and consequently reducing the risk of falls - the ultimate driver of disability for patients and of the financial burden for the health system - and at improving overall quality of life. This study has the goal to evaluate the effectiveness of the FeetMe program compared to conventional physiotherapy in participants by assessing impact on both primary motor and secondary non-motor symptoms of PD patients and quality of life.

This study has the potential of informing clinicians and physiotherapists about how new remote medicine technologies could have an impact on ameliorating the progress of their patients, particularly those that would normally not have the possibility of following a consistent, well-structured regimen of rehabilitation. Lastly, the current study findings have the potential to inform about the usefulness of novel applications as FeetMe in the clinical settings, thus further promoting the integration of digital technologies in a range of areas that support primary care and essential public health functions.

#### 4.3 Investigational Medical Device

FeetMe® Monitor is a pair of connected insoles that measure spatio-temporal gait parameters and plantar pressure to support the mobility assessment of individuals. FeetMe® Rehabilitation is a mobile application used together with FeetMe Monitor Insoles. It has been specifically developed following the HAS recommendations for rehabilitation of PD patients. It consists of exercises which are widely used in physiotherapy practice of these patients, are clinically validated and are well described in literature (Ashburn et al., 2008; Caglar et al., 2005; Hirsch et al., 2003; Ridgel et al., 2009). It composes of static exercises for balance training and muscle strengthening and dynamic exercises to improve gait quality and endurance (Appendix A). The application allows patients to perform rehabilitation at home while receiving real-time biofeedback.

Additionally, the solution includes a web platform called the FeetMe® Mobility Dashboard that allows the healthcare professionals to remotely visualize and therefore track their patients' activity. The person in charge of the follow-up (a specialist in adapted physical activity (APA)) can adapt the rehabilitation program based on the patients' progress and compliance shown in the dashboard.

Depending on the user, the solution is not used in the same way. For Patients randomized in conventional physiotherapy group, they will use the FeetMe Evaluation application to import data stored within the insoles worn. For patients in the FeetMe arm, they will use the application FeetMe Rehabilitation to import their data and to perform exercises recommended on the program (Appendix S).

#### 4.4 FeetMe Rehabilitation Service

Feet-Me rehabilitation is a comprehensive program that includes several components, the insoles, the application that hosts the excercises and the service by an adapted physical activity (APA) specialist who collaborates with the patient's health care team. During exercises, the phone app guides the patient using the data from the insoles. Additionally, a direct biofeedback is given to the patient after each excercise based on the insole data. The insole data is also transmitted and visualized on an internal FeetMe webportal called Dashboard. This enables the APA to review the data coming from the insoles and make objective conclusions about e.g.: excercise time, frequency and efficiency. Using this data along with the patient's reported information, the APA can make informed decisions in adapting the rehabilitation program to suit the patient's needs.

There are three training programs developed of different intensity (Program A, B and C, program A being the most intensive (Appendix B)) to which a patient can be allocated during the first three months of the FeetMe rehabilitation. The programs differ in the combination and the amount of excercises. A decision tree (Appendix B) is put in place to define which program intensity is the most suitable for a

patient to begin with. To select the appropriate program the necessary information will be collected using a standardised form. The (APA) specialist assigned to the study will validate the content during an introductory phone call with the patient. Maximal walking time without pause (> or < to 30min), need of walking aid and/or a caregiver, amount of free time to practice a physical activity, active (> 30min/day) or sedentary (<30min/day) lifestyle are the parameters to be evaluated.

For example, for patients at the onset of their disease who are able to walk more than thirty minutes without break and have at least four hours per week to practice, program A will be scheduled. On the contrary, for sedentary patients with a more advanced disease stage and therefore more compromised balance and mobility, program C will be the most adapted. During the introductory phone call the initial training will also be scheduled.

The programs have been created based on the four principles the HAS recommendations: intensity, diversity, regularity and continuity and were co-developed with neurologists who are experts of the field. The practice sessions are composed of specifically selected exercises as well as free walking. The principle is to gradually increase the rehabilitation intensity throughout the three months by more and longer practice sessions and more free walking activity. The program have longer total weekly duration every three weeks, with the exception of Program A that reaches the highest intensity level at Week 7 (5 hours per week). Sessions are composed of balance exercises (5 to 10 minutes), muscle strengthening exercises (5 to 10 minutes), gait quality training (5 to 10 minutes) and endurance exercises (15 to 30 minutes), always the same order. This overall schedule follows literature recommendations (Ashburn et al., 2008; Caglar et al., 2005; Ellis et al., 2005; McGinley et al., 2011; Ridgel et al., 2009) of intensive therapies. It also ensures that the program remains dynamic and versatile in order to maintain the motivation through. In case a patient originally assigned to the FeetMe arm decides to continue up to 6 months, the patient pursues the exercises and the level of intensity recommended in week 12.

Nh Total weekly Duration Periods walking sessions of sessions time / week W1-W3 3x/week 30min 60min =2h30 W4-W6 4x/week 30min 60min =3h W7-W9 45min 60min 4x/week =4h Intensity \X/10-\X/12 60min 60min 4x/week =5h W12-W24 60min 60min 4x/week =5h

Figure 1. Example of a rehabilitation program - Program B

Once the patient has the devices available at their home the rehabilitation program starts with the initial remote training during which the APA specialist explains to the patient the usage of the devices, the safety instructions to follow for ensuring the security of the patient when practising and describes the program, the exercises and how to perform a walking test. Once these first steps are done, the recommended exercises are tested to check if they are well adapted and see if the safety instructions previously described are followed by the patient. During training the patient uses the application on the mobile device. Instructions are given on the screen on how the patient should move reaching a given target. After each exercise a direct biofeedback on the performance is visualised. At the end of the training a specific questionnaire is sent to evaluate the patient's satisfaction regarding the initial training (Appendix C).

Once the program has started regular follow-up calls are scheduled during which the APA specialist discusses with the patients their progress based on the data available in the Mobility Dashboard (e.g.: the patient has difficulties to start his walking with a heel strike) and the feedback of the patient. The calls are conducted in accordance with the Sponsor's internal standard operating procedure. They are initially more frequent (weekly and then bi-weekly). If a patient proceeds up to six months the calls become monthly. During the call a standard set of questions is always asked but the discussion is also adapted to the situation, focusing on motivation, resolving difficulties the patient might face, advising on the movements to be carried out and reviewing the results obtained. Each call is documented in a report and standard data are databased (e.g.: potential adverse events, reason for non-compliance, reported device deficiencies). The reports are also sent to the investigators. If it turns out that an adaptation to the rehabilitation program is needed (e.g. : the patient has difficulties to finish an exercise or/and session or it's easy for the patient to complete all sessions planed in a week) an increase or decrease in the intensity of the program will be applied to match the patient's needs (Appendix B). In addition, if the APA observes that the patient has a low success percentage on an exercise, he will guide them how to improve theresults. All modifications must be validated by the investigator before execution.

The patients' satisfaction is evaluated by the use of a questionnaire at 1, 3 (and 6 months, if applicable) (Appendix D). At the end of the program patients return the devices to the site. *Figure 2*. *Rehabilitation Program Follow up schedule* 



#### 4.5 Conventional physiotherapy

The control arm in the study consists of patients who have a prescription for conventional physiotherapy and did not get randomised into the FeetMe arm. Their rehabilitation should typically follow the HAS recommendations nevertheless, in order to make this group the most representative of real life the protocol will not standardise what is performed as part of the conventional physiotherapy. Patients who have no access to physiotherapy despite having a prescription will therefore also be part of the conventional physiotherapy arm.

The only restrictions are the ones specified in the eligibility criteria for both arms, i.e.: patients who had LSVT Big therapy within the past 12 months or are scheduled to have it during the course of the study or patients performing vigorous exercise more than 3 times a week, 30 mins or more per session either as part of their rehabilitation or otherwise, are excluded.

Patients will be asked to track their conventional physiotherapy using the weekly diary in Appendix F so the method and the time spent on rehabilitation can be evaluated and compared for analysis.

#### 4.6 Benefit-Risk Considerations

During the study, every patient will only use the FeetMe® Monitor device and patients in the FeetMe rehabilitation groups will use FeetMe Rehabilitation applications as well.

The current generation of the insoles, which is the improvement of the previous generations, have been on the market since 2019 and have been used by approximately 2530 people. Neither this nor previous generations of the insoles have had device-related adverse events reported. The insoles have been used

in a variety of populations. In a validation study, the gait parameters of 25 healthy volunteers aged 20 to 77 years were analysed to compare the FeetMe® insoles against the GAITRite® mat reference. The devices were concluded to be equivalent in estimating the mean and variability of gait parameters (Jacobs et al., 2021). The system was also validated against the GAITRite® with 205 Multiple Sclerosis patients (Domínguez et al., 2020) and 29 Stroke patients (Farid et al., 2021). In these studies, patients had to walk 8 meters (25 Foot Walk Test) multiple times. Agreement between the devices was almost perfect in both populations. Tests with 19 adults older than 65 years in good perceived health status were carried out during single- and motor-cognitive dual-task trials while outdoor walking, mimicking real-life situations. Patients had to perform 3-minute walking tests outdoors, altogether four times. The device proved to be capable of reliably capturing between condition differences in gait parameters transparently and accurately studying ecological walking activities. Additionally, it received an excellent usability feedback (Lunardini et al., 2021). To characterise and compare gait patterns in relapsing-remitting MS and secondary-progressive MS, 141 patients were enrolled in a study where they had to perform three gait assessments, a 6MWT, a 2-minute walk test and a 25 Foot Walk Test (Granja et al., 2019). The insoles were likewise successfully used in a spastic hemiparetic patient with foot drop (David et al., 2019).

Furthermore, the insoles have already been used together with the FeetMe Rehabilitation application as remote rehabilitation service in Parkinson's disease patients. A one month pilot study to test this solution was conducted with 13 PD patients during the first lockdown period of the COVID-19 pandemic. Patients showed a very high compliance, measured by the amount of practice time versus the prescribed practice time and reported overall satisfaction with the program. Patients were further given the option to continue with the rehabilitation program and the majority chose to do so, completing three month (9 patients) and six months (7 patients) of remote rehabilitation. Importantly, a positive trend was observed in the patient's quality of life (Laplanche et al, 2021). There have been several other individual use cases where the solution was successfully deployed and an initiative where the FeetMe solution will be used by thirty PD patients with apomorphine pump is currently being conducted. Further details are provided in the Investigator's Brochure.

In the current study, during the in person study visits on site well established gait measurements (6MWTs and the MiniBESTest) will be conducted using the insoles. The testing procedures will follow standard testing instructions. These assessments will be conducted under the direct supervision of a health care professional and therefore are not considered to put the study population at any risk.

Patients in their home will either use only the insoles or the combination of the insoles and the Rehabilitation application. Patients can encounter a minimal residual risk while using the insoles which can originate from inappropriately using the charging device by using an incompatible charging module. This risk is minimised by providing all patients with an adapter compatible with their location and clear instructions in the user manual. Regarding the application, theoretically it may occur that the instructions, movement targets during the exercises or the biofeedback would not be properly displayed on the patient' smartphone screen, resulting in movements of potentially excessive amplitude and consequently in loss of balance. This risk is considered to be at an acceptable level by the Sponsor as it has been reduced to the minimal technically possible level during the development of the software and will be further mitigated by adequate training of patients before use and regular follow-up.

The current population assessed is not considered to be more compromised and therefore at higher risk compared with patients who have previously used the insoles and the smartphone application without device-related side effects. Additionally, it is ensured throughout the eligibility criteria that the study population is cognitively and physically capable of respectively understanding and executing the prescribed rehabilitation. Regular follow-up calls are also planned to verify that patients are using the solution both safely and efficiently.

Overall, any residual risk is outweighed by the benefit patients are expected to have by using the FeetMe Rehabilitation solution.

#### 4.7 Non-investigational Medical Device

The investigational site will be provided their own FeetMe® Monitor insoles together with the FeetMe® Evaluation application as a back-up (e.g.: for instances when a patient forgets their own device). During the on-site visits the gait assessments might therefore be recorded using these devices. Patients on the CPt arm will be provided the Evaluation application along their insoles in order to download the data during their remote gait monitoring. As these actions are within the intended use the devices, they are not considered as investigational medical devices in the study.

# 5 STUDY OBJECTIVES AND ENDPOINTS

Table 5.1 Study Objectives and Endpoints

| Primary Objective | Primary Endpoints |
|---|---|
| To evaluate the efficacy of FeetMe home-based rehabilitation program compared to conventional physiotherapy at Week 12 in PD patients assessed by gait velocity. | velocity (cm/s) assessed during the 6 Minutes |
| Key Secondary Objective | Key Secondary Endpoint |
| To evaluate the efficacy of FeetMe home-based rehabilitation program compared to conventional physiotherapy at Week 12 in PD patients assessed by stance time variability. | |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the efficacy of FeetMe home-based rehabilitation program compared to conventional physiotherapy at Week 12 in PD patients assessed | results of the falls diary. |
| <ul> <li>by:</li> <li>rate of falls</li> <li>standard gait and balance exercises</li> </ul> | • Change from baseline to Week 12 (Visit 3) in the asymmetry of the swing duration assessed during the 6 Minutes Walk Test (6MWT). |
| <ul><li>MDS-UPDRS Part III</li><li>quality of life</li></ul> | • Change from baseline to Week 12 (Visit 3) in the MiniBESTest. |
| | Change from baseline to Week 12 (Visit 3) in MDS-UPDRS part III sub-score. |
| | Change from baseline to Week 12 (Visit 3) the results of the Parkinson Disease Questionnaire (PDQ-39) |
| Exploratory Objectives | Exploratory Endpoints |

- To explore the long term efficacy of FeetMe home-based rehabilitation program compared to conventional physiotherapy in patients who continue to Week 24
- To explore the maintenance of the effect after 3 months in patients who stop physiotherapy at Week 12.
- To explore the efficacy in patients who switch from one treatment to the other at Week 12.
- Rate of falls at Week 24 based on the results of the falls diary.
- Change from Baseline to Week 24 (Visit 4) and from Week 12 (Visit 3) to Week 24 in:
  - Gait velocity (cm/s) assessed during the 6MWT
  - Stance Time Variability assessed during the 6MWT
  - Asymmetry of the swing duration assessed during 6MWT
  - the Mini-BESTest
  - MDS-UPDRS Part III sub-score
  - the results of the PDQ-39
- Change from Baseline to Week 12 (Visit 3) and to Week 24 (Visit 4) and from Week 12 to Week 24 in the:
  - gait parameters measured by the FeetMe Monitor during the 6MWTs other than ones of the primary and secondary endpoints
  - gait parameters measured by the FeetMe Monitor during remote gait monitoring
  - results of the pain VAS
  - results of the Parkinson Disease Sleep Scale 2 (PDSS2)
  - results of the Clinical and Patient Global Impression of Severity scales (CGI/PGI-
  - results of the Clinical and Patient Global Impression of Improvement scales (CGI/PGI-I)
  - results of the MDS-UPDRS I, II and IV sub scores

acceptability, patient's throughout the study

To explore the compliance with training, Actual versus prescribed time spent on engagement physiotherapy

To explore the satisfaction with the service

Results of the Patient and Investigator satisfaction questionnaire

rehabilitation program.

To evaluate the safety of FeetMe home-based Number of device and clinical investigational plan procedure related adverse events.

#### **5.1** Appropriateness of Measurements

Several studies support the clinical utility of using gait parameters to provide insight into the efficacy of rehabilitation. Gait velocity appears as an outcome measure for therapies such as the LSVT BIG (Millage et al, 2016) or DBS (Roger et al, 2016) and for almost all alternative forms of physical exercises aiming at improving mobility of PD patients. In the European Physiotherapy Guideline for Parkinson's Disease walking speed is graded as a "critical outcome", with an importance score of 8.6 over 10 (Keus et al, 2014). The FeetMe devices provide the opportunity to objectively and reliably measure this important outcome.

During a discussion between the HAS and the Sponsor in February 2021, the agency has supported the proposal of using gait velocity as a primary endpoint for this study. The reason being that gait velocity is shown to correlate with several other aspects of disease, e.g. risk of falls or quality of life.

In one study conducted on individuals aged 70 and older, each 10 cm/s decrease in gait speed was associated with a 7% increased risk for falls (Verghese et al., 2009). Participants with slow gait speed (≤ 70 cm/s) had a 1.5-fold increased risk for falls compared with those with normal speed. Since these falls occur during walking, apart from reduced speed, gait disturbances such as changes in stride time variability, or medio-lateral symmetry are also associated with falls. Therefore, walking speed can be an optimal proxy measure for evaluating fall risk in PD patients (Creaby and Cole, 2018; Paul et al., 2013; Rodríguez-Molinero et al., 2019; Verghese et al., 2009).

For better interpretability of the change in velocity the key secondary outcome measure of stance time variability is introduced. This parameter is described to be related to balance and motor control (Rennie et al, 2020). It is expected that a quantitative change in the gait (i.e.: speed) complemented with the quality of the change (i.e.: stance time variability) will reflect the stability of the walk and will best depict the impact of the rehabilitation therapy.

Additionally, a large pool of gait parameters will be available to further characterise the motor functions of the patients. The standards in clinic tests will be complemented with the special feature of the FeetMe devices which allows the remote continuous gait monitoring within home settings. This will provide a new pool of evidence thanks to the digital technology that can be newly adopted within this population. The non-gait-based endpoints are there to provide a holistic view on the status of the patients as they represent the clinically relevant domains of the non-motor aspects of the disease. They will be looked at independently and in relation to the various gait parameters.

#### **6 INVESTIGATIONAL PLAN**

#### 6.1 Study design and rationale

This is a multicentre, controlled, randomised in two parallel groups, open label study. The study will enroll 150 patients over approximately 18 months and 6 investigational sites.

Having multiple centres enrolling patients will not only maximise the capacity of recruitment but will allow for the evaluation of differences represented by geographical imbalances in the physiotherapy practices across France.

Patients who are found eligible and consent to participate will be randomised either on the conventional physiotherapy or on the FeetMe arm in a 1:1 ratio. Due to the set-up of the FeetMe program (i.e.: personal follow-up of the patients by an APA and the difference in the device needs between the two groups) and the obvious difference in the treatments, a blinded design is not possible. Nevertheless, the objective nature of the primary and main secondary endpoints measured by digital technology and the patient reported nature of most of the remaining outcome measures minimise any potential biassing effect originating from the open label design. Additionally, the final analysis will be performed by a independent blinded statistician.

The equal allocation of patients is maintained during the Primary Intervention Period (from the Baseline Visit till Visit 3) up to the primary endpoint evaluation at Week 12. It is in line with the duration of the FeetMe rehabilitation program. The program is built based on several regulatory recommendation including the HAS and the WHO and expert opinions suggesting that rehabilitation trainings typically show benefit after ten weeks. Additionally, most of the published data supports this duration together with the list of interventions analysed in the European Physiotherapy Guideline for Parkinson's Disease (Keus et al, 2014) where the median duration of the programs is eight weeks. The timing of the primary endpoint at Week 12 is adopted to this standard duration of an intensive rehabilitation therapy off approximately 3 months.

After the Primary Intervention Period patients will be offered to chose how to proceed i.e.: to continue on their original allocation, to switch arms or to stop treatment. In any case the patients will remain in the study until the week 26 EOS visit. The number of patients on the arms at this point will not be controlled and the data gathered will be exploratory in nature. This design is expected to:

- provide the opportunity to those patients on the conventional physiotherapy arm who will not find a therapist during the study to get access to treatment by switching to FeetMe;
- assess the ratio of the willingness to continue on the FeetMe arm in comparison to the conventional arm;
- assess the maintenance of the treatment effect in patients who decide to stop;
- compare efficacy of the two treatment within the same individual who decides to switch;
- compare the long-term efficacy of the two treatments at 6 month in patients who continue on their original allocation.

Based on the emerging data, the Sponsor may decide to open an extension phase, where all participants have the option to take part or prolong their participation in the FeetMe rehabilitation program. Such extension to this study may be offered to all patients, contingent on the Sponsor's decision to implement it and could be described in a separate document.

In case study conduct will be compromised by the COVID-19 pandemic a contingency plan will be provided in a clinical investigational plan addendum.

FeetMe reserves the right to temporarily suspend or prematurely discontinue the study at any time. The study may also be terminated prematurely at any time when agreed by both the Investigators and the Sponsor as being in the best interest of the patients. In terminating the study, FeetMe and the Investigator will ensure that adequate consideration is given to the protection of the patients' interests. If the study is prematurely terminated or suspended, FeetMe will inform the Investigators/institution and the regulatory authorities and IEC in accordance with applicable regulatory requirements. In addition, arrangements will be made for the return of all study material provided by the Sponsor.

Figure 3. Schematic of the study design



#### 6.2 Schedule of Assessments

Table 6.1 Schedule of Assessments

### CONFIDENTIAL May 2023

| | | Primary Intervention Period | | | | Long Term Intervention Period | | | |
|---|---|---|---|---|---|---|---|---|---|
| Visit | Screening <sup>1</sup> | Baseline <sup>2</sup> | Visit 1 | Visit 2 | Visit 3 | Visit 1.2 | Visit 2.2 | Visit 4 | End of Study<br>Visit |
| Timepoint | Day 1 | Day 1 | Week 4 | Week 8 | Week 12 | Week 16 | Week 20 | Week 24 | Week 26 |
| Visit Window | NA | NA | ± 7 days | ± 7 days | ± 7 days | ± 7 days | ± 7 days | ± 7 days | ± 7 days |
| Assessments | In-Clinic +<br>Remote | In-Clinic | Remote | Remote | In-Clinic | Remote | Remote | In-Clinic | Remote |
| | | | | | | patients | who switch | | |
| ICF | • | | | | | | | | |
| Eligibility Check | • | | | | | | | | |
| Modified Hoehn and<br>Yahr staging | • | | | | | | | • | |
| MoCA | • | | | | | | | | |
| Medical History &<br>Demographics | | • | | | | | | | |
| Randomisation | • | | | | | | | | |
| Prior Rehabilitation<br>History | • | | | | | | | | |
| Prior- and Concomitant<br>Medication | • | | | | • | | | | |
| 6MWT <sup>3</sup> | | • | | | • | | | • | |
| Ecological remote gait data collection | | for 2 weeks<br>after BL | | | for 2 weeks<br>after V3 | | | for 2 weeks<br>after V4 | |
| Mini-BESTest | | • | | | • | | | • | |
| MDS-UPDRS | | • | | | • | | | • | |

# CONFIDENTIAL May 2023

| FOG-Q | | • | | | • | | | • |
|---|---|---|---|---|---|---|---|---|
| PDSS-2 | | • | • | • | • | • | • | • |
| Pain VAS | | • | • | • | • | • | • | • |
| PDQ-39 | | • | | | • | | | • |
| PDQ-8 | | | • | • | | • | • | |
| CGI-S / PGI-S | | • | | | | | | |
| CGI-I / PGI-I | | | | | • | | | • |
| Satisfaction Questionnaire | | • | | | • | | | • |
| Falls diary | | | | | | | | |
| Conventional<br>Physiotherapy tracking | From ICF to EOS | | | | | | | |
| AEs | | | | | | | | |
| Adherence | | | | | • | | | • |

ICF: Informed Consent Form; 6MWT: 6 Minutes Walk Test; Mini-BESTest: Mini Balance Evaluation Systems Test; MOCA: Montreal Cognitive Assessment; AEs: Adverse Events; FOG-Q: Freezing of Gait Questionnaire; MDS-UPDRS I, II & III: Unified Parkinson's Disease Rating Scale parts I, II and III; PDQ-39: Parkinson Disease Questionnaire; PDQ-8: Parkinson Disease Questionnaire Short Form; CGI-S/PGI-S: Clinical/Patient Global Impression of Severity; CGI-I/PGI-I: Clinical/Patient Global Impression of Improvement; PDSS-2: Parkinson Disease Sleep Scale 2;

<sup>&</sup>lt;sup>1</sup>A reflection period of fifteen to thirty days must be given to the subject to decide upon their participation.

<sup>&</sup>lt;sup>2</sup> BL assessments will take place right after the Screening Visit.

<sup>&</sup>lt;sup>3</sup> Patients on the FeetMe arm will perform weekly 6MWTs as part of their rehabilitation program using the FeetMe Rehabilitation application. Note: Visit windows are to be calculated compared to the original schedule, not the previous visit

#### 6.3 Study Population

#### 6.3.1 Sample Size

A total of 150 patients will be recruited for this study. A drop-out percentage of 20% was inferred from previous studies using FeetMe Rehabilitation application on a similar population and was considered in the calculation of the sample size.

#### 6.3.2 Inclusion Criteria

All patients must fulfil the following criteria:

- 1. Written informed consent to participate in the study.
- 2. Male or female patients between 40 to 70 years of age, inclusive.
- 3. Body weight range of 40 kg to 120 kg and a body mass index (BMI) of 18 to 34 kg/m2.
- 4. Diagnosis of Idiopathic Parkinson's disease (PD) according to UK Brain Bank Criteria (2/3 symptoms), with Hoehn and Yahr (H&Y) staging level 2, 2.5 or 3.
- 5. Disease onset of at least 3 years prior to enrolment.
- 6. Patients with a history of 50% levodopa responsiveness based on motor signs.
- 7. On stable treatment of PD medication for at least 30 days before screening and with no expected major changes during the first 3 months of the study.
- 8. Prescription for physiotherapy available.
- 9. Ability to walk without aid for at least 6 minutes.
- 10. Shoe size between 35 46 (European Standard).
- 11. Intact skin on feet.
- 12. Adequate visual and auditory acuity to perform the rehabilitation program and the assessments in the Investigator's judgement.
- 13. Comfortable with the use of a smartphone. If assistance is required for the use of FeetMe technology, a caregiver or volunteer is fully available to assist the patient.
- 14. Willingness to be regularly contacted via phone-calls.
- 15. Willingness to suspend conventional physiotherapy treatment and start the FeetMe rehabilitation program, if applicable.
- 16. French speaker.

#### 6.3.3 Exclusion Criteria

Patients must not fulfil the following criteria:

- 1. Medical history indicating a Parkinsonian syndrome other than idiopathic PD.
- 2. Unable to walk without walking aid or presence of an injury preventing the patient to walk.
- 3. Any relevant comorbidity or vestibular/visual dysfunctions limiting locomotion or balance.
- 4. Clinically significant comorbidities which in the judgement of the investigator may preclude the reliable gait assessment of the patient.
- 5. Patients with poor wound healing or broken skin on the feet.
- 6. Patients with foot implants.

- 7. Montreal Cognitive Assessment (MoCA) score  $\leq 24/30$ .
- 8. Patients with dementia.
- 9. Patients with apathy.
- 10. Participation in another clinical trial with an investigational drug/ therapeutic within the three months before screening and during the study, unless agreed by the Sponsor.
- 11. Patients who had Lee Silverman Voice Treatment (LSVT) Big therapy within the past 12 months or have it planned during the course of the study.
- 12. Patients with Deep Brain Stimulation planned during the first 12 weeks of the study.
- 13. Patients with pacemakers.
- 14. Patients performing vigorous exercise > three times a week, 30 mins or more per session

#### 6.3.4 Patient Replacement

Patients will not be replaced in the study.

#### 6.4 Investigational Medical Device

#### 6.4.1 Device Description

FeetMe® Monitor connected insoles is a wearable medical device that measure spatio-temporal gait parameters and plantar pressure to support the mobility assessment of individuals. The hardware product consists of two regular shape insoles and a double-head wireless charger with wall adaptor to charge both insoles simultaneously. The insoles are available in 12 sizes ranging from 35 to 46 (EU standard) or from 4.5 to 13 (US standard for men) or 5.5 to 14 (US standard for women).

An insole includes one Inertial Measurement Unit (IMU) with a 3-D accelerometer and a 3-D gyroscope to capture movement in 6 directions and eighteen capacitive cell pressure sensors, around 15 mm² cell area each. In the insoles heel strike (HS) and toe off (TO) events are detected by the pressure sensors and the related temporal parameters are calculated from HS and TO event timings. HS, TO and stride length are calculated in each insole and are defined as insole-based parameters. For each insole, these parameters are sent to a mobile application via Bluetooth Low Energy. The velocity, stride length, stride duration, stance duration, swing duration, step duration, single support duration and double support durations, cadence, number of steps, distance, duration of walking test are defined as mobile-based parameters and are calculated by a dedicated mobile application. The mobile application allows the real-time recording and/or visualization of the gait parameters. FeetMe® Monitor is marketed, CE-marked class Im medical devices (under rule 1 and under rule 12 of ANNEX IX of Medical Device Directive 93/42/EEC amended by Directive 2007/47/EC) (MDD), and FDA approved (510k exempt)). Insoles are manufactured by FeetMe.

Figure 4. Picture of a FeetMe Insole with charger and related smartphone application





CIP Number 2023-A00150-45 Final version 0.2

The individual chargers are to be connected to a power outlet and positioned on the white round marks of the insoles. The induction chargers will position themselves automatically. LED lights will indicate the charging status of the insoles. It takes approximately 2.5 hours for a complete charge of the insoles.

Detailed user guides will be provided for both the patients and investigators on each device.

For further information please refer to the Investigator's Brochure.

#### 6.4.2 Data collection

Data collected by the insoles are described below.

#### Unipedal parameters collected

- Stride duration (ms)
- Stance duration (ms)
- Swing duration (ms)
- Stride length (m)
- Stride elevation (m)
- Velocity (m/s)
- Swing velocity (m/s)
- Cadence (steps/min)

#### Bipedal parameters collected

- Single support duration (ms)
- Double support duration (ms)
- Step duration (ms)

#### Balance data and pressure data

- Mean CAPA values during stance phase for each sensor
- Extraction of 16 points of the estimated center of pressure (COP) trajectory during stance phase
- antero-posterior & medio-lateral COP trajectories: amplitude of COP
- Center of pressure trajectory
- ground force reaction (heel & toe)

#### **Exercises data**

- percentage of success of exercise
- daily/weekly/monthly practiced time
- practiced time per exercise
- daily/weekly/monthly number of exercises performed

All personal data collected for the patient follow-up (name,phone number, email adress) will be deleted at the end of the study.

#### 6.4.3 Packaging and Labelling

Each pair of insoles will be packed individually along with chargers and will be identified with a unique serial number. The sites will be supplied with multiple pairs in each size. Each patient will receive one pair of insoles and the charger. A mobile device with the FeetMe Rehabilitation application will be provided to the patients in the FeetMe rehabilitation program and patients in the Conventional physiotherapy arm who don't have Android devices. Additionally, each site will receive a mobile device with the FeetMe Evaluation application installed on it to perform on-site gait analysis, in case necessary (e.g.: a patient forgets to bring their device to a visit). No study specific labelling will be used.

#### 6.4.4 Blinding

Blinding is not applicable (see Section 6.1).

#### 6.4.5 Supply and Accountability

The devices (insoles, chargers, mobile devices) will be supplied by FeetMe. It is not allowed to use the devices for other uses than those defined in the clinical investigational plan. Devices must be exclusively used for the identified patients of this study.

The Investigator or designee must confirm the receipt of the devices. Upon receipt of the devices the Investigator or designee will conduct an inventory of supplies, verify and document that the devices are intact and the correct amount have been shipped. The CRA must verify the documentation. Request of new insoles (e.g.: due to higher need of a particular size) or exchange of faulty ones will be ensured by the Sponsor. The site must keep track of the return of any equipment.

At the end of the study all devices will need to be returned to the Sponsor in their original packaging.

Further details are provided in the Study Procedure Manual.
#### 7 STUDY ASSESSMENTS BY VISIT

#### 7.1 Introduction and reflection period

During their routinely scheduled visit at the investigational site patients who express interest in participating in the study will be introduced to the device. Then, patients return to their home and have a reflection period of 15 days to 1 month. If judged to be comfortable with and interested in the technology they will screened for participation. Beforehand the inclusion / exclusion criteria will be assessed at high level without capturing any data to make sure there are no obvious exclusionary factors. The MoCA and no other only protocol mandated assessment will not be performed.

#### 7.2 Screening

#### 7.2.1.1 Screening

If the patients deciced during the reflection period to participate they will return to the site for the Screening Visit.

The following assessments will take place within the Screening Visit done by the investigators (neurologists):

- Verify the informed consent.
- Eligibility criteria evaluation, including the definition of disease stage (H&Y) and cognitive status (MoCA), dementia and apathy.

All inclusion and exclusion criteria will be assessed to confirm the patient's eligibility for the study. Study sites are required to document all screened patients initially considered for inclusion in the study and collect the reason of screening failure. For the evaluation of dementia and apathy there are no protocol mandated assessments, the sites can use their routine diagnostic tools.

• Rehabilitation history

#### 7.2.1.2 Randomisation

Eligible patients will be randomised using an Interactive Voice/Web Response System (IXRS) randomised either on the conventional physiotherapy or on the FeetMe arm in a 1:1 ratio. Randomisation will be stratified by the covariable "already in a rehabilitation program" and by study site. We will use a dynamic randomisation procedure by minimization using the Pocock and Simon method. Randomization will result in the assignement of the unique Patient ID, which will be used on all study-related documents pertaining to the patient. Any identification numbers that are assigned will not be reused even if the patient does not continue in the study.

#### 7.2.2 Re-Screening

Patients who fail screening criteria can be retested once according to the Investigator's judgement. In this case, the same ID previously assigned will be used in the study.

#### 7.2.3 Screen Failure

Patients who do not meet the eligibility criteria will be considered screen failed. The reason for screen failure must as a minimum be documented.

#### 7.3 Baseline Visit

All randomised patients will participate in the Baseline Visit. This visit will be on the same day as the Screening Visit.

Patients will be instructed in the use of the FeetMe Monitor and wear the insoles for the duration of the visit, while performing a series of assessments.

The following assessments will be performed at the Baseline Visit:

- Demographic data collection (month and year of birth; gender, weight, height, leg length, shoe size)
- Recording of relevant medical history, prior medications
- Gait Assessments, which must be performed in ON-phase:
  - 6 Minutes Walk Tests (6MWT)
  - Mini-BESTest

During the 6MWT and the Mini-BEST gait data will be recorded using the FeetMe Rehabilitation or Evaluation application. Specific instructions set out in the Site User Manual must be followed when setting up and executing the assessments.

- Disease specific rating scales:
  - The Movement Disorder Society sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
- Other Assessments:
  - Freezing of Gait Questionnaire (FOG-Q)
  - Parkinson Disease Sleep Scale 2 (PDSS2)
  - Pain VAS
  - Parkinson Disease Questionnaire (PDQ39)
  - Patient Global Impression of Severity (PGI-S)
  - Clinical Global Impression of Severity (CGI-S)

## 7.4 Primary Intervention Period

Following the Baseline Visit, all patients will begin their 12-week physiotherapy (or no-physiotherapy) regimen according to their randomisation.

During this period:

- All patients will participate in the Remote Gait Monitoring 1 and Visits 1-3 (Sections 7.3.1, 7.3.2, 7.3.3).
- Patients on the Conventional Physiotherapy arm, if they have access to it will start or continue their conventional physiotherapy and will keep track of it using the Conventional Physiotherapy Tracking Sheet (Appendix F). Patients who did not have access to CPt at the time of inclusion but manage to arrange one during the Primary Intervention Period will restart their PIP.
- On the other arm patients will start the FeetMe rehabilitation program (Section 4.4, Appendix A and B).
- In addition, all patients will keep a falls diary (Appendix G).

#### 7.4.1 Remote Gait Monitoring 1

At the end of the Baseline Visit, all patients will take the FeetMe Insoles, mobile devices and chargers with them to their homes. A Patient User Guide will be provided.

- All patients will use the insoles remotely while performing their day-to-day activities (including physiotherapy) for two weeks. Data will be recorded in standalone mode (without a phone).
- Patients will download the data from the insoles at the end of each day.

#### 7.4.2 Visits 1 and 2

Four and eight weeks after Baseline Visit, two remote visits (Visit 1 and 2) will take place. Patients will be asked to fill in the following questionnaires:

- PDSS-2
- Pain VAS
- Parkinson Disease Questionnaire, Short Form (PDQ-8).

#### 7.4.3 Visit 3

Twelve weeks after Baseline Visit, that is, at the end of the 12-week Primary Intervention Period, all patients will participate in an in-clinic visit (Visit 3), where they will perform the same series of assessments as in the Baseline Visit. Patients will need to bring their FeetMe devices, their diaries, trackers and filled-in questionnaires to the visit.

The following assessments will be performed at Visit 3:

- Gait Assessments, which must be performed in the ON-phase:
  - 6 Minutes Walk Tests (6MWT)
  - Mini-BESTest.

During the 6MWT and the Mini-BESTest patients must wear the insoles. Specific instructions set out in the Site User Manual must be followed when setting up and executing the assessments.

- Disease specific rating scales:
  - MDS-UPDRS
- Other Assessments:
  - FOG-Q
  - PDSS2
  - Pain VAS
  - PDQ39
  - Clinical Global Impression of Improvement / Patient Global Impression of Improvement (CGI/PGI-I)
- Potential adverse events and change in concomitant medication since the last contact.
- The source documents must be collected from the patients and the diary and tracker transcribed into the database.
- Also, the patients further allocation is to be decided (Section 7.4).
- At the end of the visit the patients will return home with their devices (as applicable based on their new or unchanged treatment) and proceed into the Remote Gait Monitoring 2 (Section 7.4.1).

#### 7.5 Long Term Intervention Period

During Visit 3 patients will be asked whether they want to:

a) continue with their already assigned treatment;

Patients will continue with their respective rehabilitation programs.

b) switch to the other arm;


If patients on the conventional physiotherapy arm would like to start the FeetMe program they will be trained to use the devices and will start their 12 weeks program. Patients of FeetMe group wanting to switch from FeetMe to CPt will need to arrange the care themselves. Patients who switch will have the same visit schedule as during the first three months.

c) discontinue rehabilitation.

If a patient would like to discontinue rehabilitation they will still be asked to remain in the study for further data collection.

## 7.5.1 Remote Gait Monitoring 2

At the end of Visit 3, all patients will perform a second remote gait monitoring period. All patients will use the insoles remotely while performing their day-to-day activities (including physiotherapy) for 2 weeks. Data will be recorded in standalone mode (without a phone).

#### 7.5.2 Visits 1.2 and 2.2

Four and eight weeks after Visit 3, that is at week 16 and week 20 from Baseline Visit patients who decided to switch will take part in a virtual remote visit (Visit 1.2 and Visit 2.2 respectively).

Patients will be asked to fill in the following questionnaires:

- PDSS-2
- Pain VAS
- Parkinson Disease Questionnaire, Short Form (PDQ-8).

#### 7.5.3 Visit 4

Twelve weeks after Visit 3, that is, at the end of the 12-week Long Term Intervention Period, all patients will participate in an in-clinic visit (Visit 4), where they will perform the same series of assessments as in the Baseline Visit and Visit 3. Patients will need to bring their FeetMe devices, their diaries, trackers and filled-in questionnaires to the visit.

The following assessments will be performed at Visit 4:

- Gait Assessments, which must be performed in the ON-phase:
  - 6 Minutes Walk Tests (6MWT)
  - Mini-BESTest.

During the 6MWT and the Mini-BESTest, patients must wear the insoles. Specific instructions set out in the Site User Manual must be followed when setting up and executing the assessments.

- Disease specific rating scales:
  - MDS-UPDRS
- Other Assessments:
  - FOG-O
  - PDSS2
  - Pain VAS
  - PDQ39
  - Clinical Global Impression of Improvement / Patient Global Impression of Improvement (CGI/PGI-I)
- Potential adverse events and change in concomitant medication since the last contact.

- The source documents must be collected from the patients and the diary and tracker transcribed into the database.
- At the end of the visit the patients will return home with their devices and proceed into the Remote Gait Monitoring 3 (Section 7.4.4).

## 7.5.4 Remote Gait Monitoring 3

At the end of Visit 4, all patients will take the FeetMe Insoles with them to their homes. All patients will again use the insoles remotely while performing their day-to-day activities (including physiotherapy) for two weeks. Data will be recorded in standalone mode.

Once the Remote Gait Monitoring 3 period is completed, all patients will return all the FeetMe devices to the site via courier. The site personnel will make sure the data is downloaded as described in the Site User Manual.

## 7.6 End of Study Visit

An End of Study Visit will be scheduled remotely. Patients will receive a phone call from the Investigator who will ask them about:

- Potential adverse events and change in concomitant medication since the last contact.
- Satisfaction with the medical device and smartphone applications (Appendix D).

Once the End of Study Visit is completed, the patient's participation in the study will be considered concluded.

## 7.7 Withdrawal / Early Termination Visit

Patients may withdraw from the study at any time at their request or following a decision of the Investigator or Sponsor. In case of termination due to a patient's decision, every effort should be made to determine the primary reason for withdrawal and to document it in the eCRF.

#### 8 STUDY ASSESSMENTS

## 8.1 Gait Assessments

## 8.1.1 6 Minutes Walk Test (6MWT)

The 6 Minutes Walk Test is a standard performance exercise test designed to assess the functional capacity and walking endurance of a patient in the clinical setting (American Thoracic Society, 2002). The 6MWT consists of a single activity, administered by the Investigator, in a flat indoor corridor at least 30 metres in length, marked every three metres and delimited by cones indicating turnaround points. During the 6MWTs the patients should be in ON state. They will be wearing the insoles. The test will be recorded using a FeetMe application.

The Investigator instructs the patient to walk at a comfortable pace and cover the longest distance possible, then measures the total distance the subject can travel over a six minute period. The total score is the walked distance in metres. This test can be administered by the Investigator or by health care personnel trained in the procedures of the evaluation. The 6MWT takes approximately 10 minutes to complete. The date and time of the assessment are to be recorded in the eCRF.

The standard 6MWT will be performed during the on site visits at BL, Visit 3 and Visit 4. Detailed instructions on how to execute the test are given in the Site User Manual.

## 8.1.2 Remote 6 Minutes Walk Test (6MWT)

The remote version of the 6MWT is a self-administered adaptation of the 6MWT (see paragraph 8.1.1), designed to assess the functional capacity and walking endurance of a patient in a more familiar setting (e.g. home, workplace). This test consists of a single activity, self-administered by the subject in a place of their choosing, preferably featuring a hard, flat surface which presents sufficient space for an adult person to walk safely, without objects or obstacles hindering the subject's performance or putting the subject in danger of falling or hurting themselves. The remote 6MWT shall be performed outdoors to avoid many U-turns. The patient is asked to do the test in ON conditions and at the same time and place every week.

Weekly 6MWT tests are part of the FeetMe rehabilitation program, therefore only patients who are on the FeetMe arm will perform them using the FeetMe Rehabilitation application. The application instructs the patient to walk at pace to cover the longest distance possible, then measures the total distance the subject can travel over a six minute period. The total score is the walked distance in metres. The remote 6MWT takes approximately 10 minutes to complete. The date and time of the assessment will need to be recorded in the eCRF.

## 8.1.3 Mini Balance Evaluation Systems Test (Mini-BESTest (Appendix L))

The Mini Balance Evaluation Systems Test is a standard performance rating scale designed to evaluate a patient's static and dynamic balance (Franchignoni et al., 2010). The assessment, administered by the Investigator, includes fourteen balance-related tasks, each scored on a scale from 0-2 based on the observed patient ability and independence in performing each exercise. The Investigator evaluates the patient's performance and assigns a score to each exercise. The individual scores are subsequently summed to yield a total score ranging from 0 to 28, where higher scores indicate better performance. The Mini-BESTest takes approximately 15 minutes to complete. During the test the patients should be in ON state and will be wearing the insoles. The date and time of the assessment and the sub-scores will be captured in the eCRF.

The MiniBESTest will be performed during the on site visits at BL, Visit 3 and Visit 4. Detailed instructions on how to execute the test are given in the Site User Manual.

#### **8.2** Medical History

A complete past medical history will be collected by the Investigator or appropriate site staff according to standard practice and recorded in the eCRF. This will include a history of all previous diseases and illnesses, those currently being treated until the time of the screening visit, as well as those which have any residual effects on the patient's health. Moreover, surgical history will be collected, including all invasive procedures the patient has undergone until the time of the screening visit. Previous falls should be recorded to the extent possible.

## 8.3 Prior- and Concomitant Medication

Details of all medication taken  $\leq$ 3 months prior to the Screening Visit or during the study until the EOS Visit will be collected by the Investigator or the site staff according to standard practice and recorded in the eCRF.

Patients are eligible if on stable treatment of PD medication for at least 30 days before screening. Major changes in PD treatment during the first 3 months of the study are not allowed. What is considered a major change is up to investigator judgement, nevertheless, in principle anything that would alter the gait of the patient is considered as such. For example, adaptation of the levodopa dose to maintain current level of ambulation is not considered a major change, while changing the posology of the

treatment (e.g.: switching from per os to parenteral), or introducing a new one would classify as one. Ideally no major changes should be issued during the whole duration of the study in other medication that can influence overall data interpretation either (e.g.: antidepressants).

In case major changes in concomitant medication are unuvoidable, either due to the worsening of a disease or a new disorder, it must be recorded in the eCRF specifying the reason (e.g.: worsening of a medical history, adverse event or as a new adverse event) and will be taken into account during analysis.

#### 8.4 Rehabilitation

A history of prior rehabilitation therapy (e.g. physiotherapy, aerobic exercise) will be collected by the investigator or the site staff and recorded in the eCRF. This will include information about the type (e.g. treadmill, nordic walking), frequency (hours/week) and duration of the rehabilitation performed by the patient until the Screening Visit.

In addition, concurrent rehabilitation for the CPt arm will be collected using the Conventional Physiotherapy Tracking Sheet (Appendix F) in an electronic form from the signature of the ICF until EOS, including the type and frequency of the rehabilitation performed.

## 8.5 Device Deficiencies and Complaints

Device deficiency is the inadequacy of a medical device with respect to its identity, quality, durability, reliability, usability, safety or performance. Device deficiencies include malfunctions, use errors, and inadequacy in the information supplied by the manufacturer, including labelling.

All device deficiencies of the investigational device will be documented throughout the study by the Investigator on a dedicated form provided or by the Sponsor directly. The Sponsor is responsible for managing the deficiencies in accordance with written procedures for the control of a non-conforming product and complying with the reporting rules to authorities. The Sponsor will take, where applicable, appropriate corrective and preventive actions to protect the safety of subjects, users, and other persons. The Sponsor will arrange for the safe return of the investigational device that is related to the device deficiency.

Any device deficiencies resulting in a safety event must be recorded as an adverse event indicating the relatedness.

Complaints regarding the usability of the device coming either from the patient or the site staff will be documented on the dedicated form and will be provided to the Sponsor for evaluation on a regular basis.

## 8.6 Clinical Scales

Clinical scales will be either completed during site visits or remotely by the patient in a paper format which will serve as a source document. Sub- and/or final scores will be recorded in the eCRF.

#### 8.6.1 Montreal Cognitive Assessment (MoCA)

The Montreal cognitive assessment is a widely used clinical screening assessment designed to evaluate cognitive impairment (Nasreddine et al., 2005). The MoCA consists of 16 items belonging to multiple cognitive domains (visuo-spatial and executive functions, naming, memory, attention, language, abstraction and orientation). Each element is scored according to its individual procedure to yield a total score ranging from 0 to 30, where lower numbers indicate worse cognitive performance. The neurologist administers the assessment and performs the scoring. The MoCA takes approximately 10 minutes to complete.

The MoCA will be performed at Screening (Appendix K).

## 8.6.2 Modified Hoehn and Yahr staging (mH&Y)

The modified Hoehn and Yahr scale is a standard clinical rating scale, designed to evaluate the progression and level of functional disability associated with Parkinson's disease and Parkinsonism in a clinical setting (Hoehn and Yahr, 1967). The Hoehn and Yahr scale consists of seven stages describing the extent and impact of symptoms (Goetz et al., 2004). The Investigator performs an interview and a medical examination aimed at evaluating the extent of the patient's symptoms and functional disability. The Investigator scores the stage based on the clinical criteria, where a higher stage value indicates more severe symptoms. The Hoehn and Yahr staging takes approximately 15 minutes to complete.

The mH&Y staging will be performed at Screening and at Visit 4 (Appendix N).

# 8.6.3 The Movement Disorder Society sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS)

The Movement Disorder Society sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is a comprehensive assessment of the Non-Motor aspects of Experiences of Daily living (nM-EDL), Activities of Daily Living (ADL), motor symptoms and motor complications of Parkinson's Disease (Goetz et al., 2008). The MDS-UPDRS Part I is a clinician rated (question 1-6) and patient self-reported scale (question 7-13) consisting of 13 questions about Non-Motor aspects of daily living; Part II is a patient self-rated scale consisting of 13 questions about ADLs; Part III is a clinician-rated scale consisting of 18 neurological motor examinations and part IV is a clinician rated scale consisting of 6 motor examinations evaluating dyskinesias and motor fluctuations. All sections are scored on a five point interval scale ranging from 0 (absence of impact) to 4 (most severe impact). Part I is administered partly by the Investigator and partly self-reported by the patient or caregiver; Part II is self-administered by the patient or caregiver and reviewed by the Investigator for consistency; Part III and IV are administered by the Investigator. The MDS-UPDRS takes overall approximately 35 minutes to complete.

The MDS-UPDRS will be performed on site at Baseline Visit, Visit 3 and Visit 4 (Appendix M).

## 8.6.4 Parkinson's Disease Questionnaire (PDQ-39)

The Parkinson's Disease Questionnaire is a reliable patient self-rated scale, designed to evaluate the impact of disease on quality of life in Parkinson's patients (Peto et al., 1995). The PDQ-39 consists of 39 questions divided in eight dimensions corresponding to different aspects of daily life (mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort). The questions are scored on a five point interval scale ranging from 0 (absence of impact) to 4 (most severe impact). The individual scores of each dimension are subsequently summed to yield a total, where higher values indicate a more severe impact on that aspect of the patient's life. This test is self-administered by the patient. The PDQ-39 takes approximately ten minutes to complete.

The PDQ-39 will be performed on site at Baseline Visit, Visit 3 and Visit 4 (Appendix I).

#### 8.6.5 Parkinson's Disease Questionnaire (PDO-8)

The Parkinson's Disease Questionnaire is a short-form patient self-rated scale derived from the PDQ-39, designed to quickly evaluate the impact of disease on quality of life in Parkinson's patients (Jenkinson et al., 1997). The PDQ-8 was created by selecting the one question in each of the eight dimensions of PDQ-39 which had the highest correlation with the final sub score of that dimension (Mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication and bodily discomfort). The PDQ-8 therefore consists of eight questions, each already present in the original PDQ-39 and representing all dimensions. The questions are scored on a five point interval scale ranging from 0 (absence of issue) to 4 (issue always present). The individual scores of each dimension are subsequently summed to yield a total, which is reported as a percentage of the total possible score, where higher percentage values indicate a more severe impact on that aspect of the

patient's life. This test is self-administered by the patient. The PDQ-8 takes approximately five minutes to complete.

The PDQ-8 will be performed remotely at Visit 1, Visit 2, Visit 1.1 and Visit 2.1 (Appendix J).

#### 8.6.6 Clinical Global Impression of Severity (CGI-S)

The Clinical Global Impression of Severity is a standard clinician rating scale commonly used in Parkinsonism clinical trials, designed to assess the severity of symptoms of a patient (Guy, 1976). The CGI-S consists of a single assessment, scored on a scale ranging from 1 (normal/least severe symptoms) to 7 (most severe symptoms). The Investigator performs a medical examination and the scoring. The CGI-S takes around three minutes to complete.

The CGI-S will be performed at the Baseline Visit (Appendix R).

## 8.6.7 Patient Global Impression of Severity (PGI-S)

The Patient Global Impression of Severity is a standard patient self-rated scale, designed to evaluate the severity of symptoms of a patient (Guy, 1976). The PGI-S consists of a single assessment, scored on a scale ranging from 1 (normal/least severe symptoms) to 7 (most severe symptoms). This assessment is self-administered by the patient. The PGI-S takes approximately three minutes to complete.

The PGI-S will be performed at the Baseline Visit (Appendix Q).

## 8.6.8 Clinical Global Impression of Improvement (CGI-I)

The Clinical Global Impression of Improvement is a standard clinician rating scale commonly used in Parkinsonism clinical trials, designed to assess the patient's improvement over a period of time (Guy, 1976). The CGI-I consists of a single assessment, scored on a scale ranging from 1 (very much improved) to 7 (very much worse). The investigator performs a medical examination and the scoring. The CGI-I takes around three minutes to complete.

The CGI-I will be performed at Visit 3 and Visit 4 (Appendix R).

## 8.6.9 Patient Global Impression of Improvement (PGI-I)

The Patient Global Impression of Improvement is a standard patient self-rated scale, designed to evaluate the improvement of the patient's condition over a defined period of time from his/her own perception (Yalcin and Bump, 2003). The PGI-I consists of a single assessment, scored on a scale ranging from 1 (normal/least severe symptoms) to 4 (most severe symptoms). This assessment is self-administered by the patient. The PGI-I takes approximately three minutes to complete.

The PGI-I will be performed at Visit 3 and Visit 4 (Appendix Q).

#### 8.6.10 Parkinson Disease Sleep Scale 2 (PDSS-2)

The Parkinson Disease Sleep Scale 2 is a reliable instrument for quantifying sleep disruption in Parkinson's Disease patients (Chaudhuri, 2002). The PDSS-2 consists of 15 questions, addressing the frequency of sleep-related difficulties and disturbances. The PDSS-2 is scored on a 11-point interval scale ranging from 0 (most frequent presence of sleep disturbances) to 10 (absence of sleep disturbances). The individual scores are subsequently summed to yield a total score ranging from 0 to 150. This test is self-administered by the patient. The PDSS-2 test takes approximately five minutes to complete.

The PDSS-2 will be performed at the site during the Baseline Visit, Visit 3 and Visit 4 and remotely during Visit 1, Visit 2, Visit 1.1 and Visit 2.1 (Appendix P).

## 8.6.11 Pain Visual Analog scale (VAS)

The pain Visual Analog Scale is a standard patient rating scale, commonly used to evaluate the intensity of pain experienced by the patient. The pain VAS consists of a unidimensional graduated segment indicating pain in the form of numbers from 0 (no pain) to 10 (maximum imaginable pain). The pain VAS is therefore scored on a 11-point interval scale ranging from 0 to 10. This test is self administered by the patient. The pain VAS takes approximately 3 minutes to complete.

The Pain VAS will be performed at the site during the Baseline Visit, Visit 3 and Visit 4 and remotely during Visit 1, Visit 2, Visit 1.1 and Visit 2.1 (Appendix H).

## 8.6.12 Freezing of gait questionnaire (FOG-Q)

The Freezing of gait questionnaire is a patient self-rated, investigator administered scale designed to evaluate freezing of gait in patients with Parkinson's disease or Parkinsonism (Giladi et al., 2000). The FOG-Q consists of six questions scored on a five point interval scale ranging from 0 (absence of symptoms) to 4 (most severe symptoms). The individual scores are subsequently summed to yield a total score ranging from 0 to 24, where higher scores indicate a more severe freezing of gait. The FOG-Q test takes approximately five minutes to complete.

The FOG-Q will be performed at Baseline Visit, Visit 3 and Visit 4 (Appendix O).

## 8.7 Falls Diary

Patients have to keep a falls diary throughout their participation in the study by registering falls and near falls, as described in Appendix G. They will need to bring their diaries to the site visits so the data can be registered in the database.

## 8.8 Conventional Physiotherapy tracking

Patients on the conventional physiotherapy arm will need to keep track of the quantity and type of physical rehabilitation they receive, as described in Appendix F. They can request help from their physiotherapist. Patients will need to bring their diaries to the site visits so the data can be registered in the database.

#### 8.9 Safety Assessments

Adverse events of special interest, serious adverse events and all device related non-serious and serious adverse events will be collected from the signature of the ICF until the participation of the patient is completed within the study. Serious Adverse Device Effects will be reported to the authorities.

In case an adverse event is suspected during the regular follow-up calls between the patient and the APA specialist, the APA specialist will contact the Investigator to enquire the investigation of the event and the assessment of severity and causality.

Detailed instructions on recording and reporting of serious safety incidents will be provided in the Study Procedure Manual.

#### 8.9.1 Adverse Events

An Adverse Event (AE) is "any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment". Since no pharmaceutical products will be administered in this study no AEs will be collected other than the AEs of Special Interest (Section 8.7.3).

### 8.9.2 Serious Adverse Events (SAE)

An SAE is an adverse event that could lead to any of the following:

- a) Death
- b) Serious deterioration in the health of the patient, users, or other persons as defined by one or more of the following:
  - 1) a life-threatening illness or injury
  - 2) a permanent impairment of a body structure or a body function including chronic diseases
  - 3) in-patient hospitalisation or prolonged hospitalisation
  - 4) medical or surgical intervention to prevent life-threatening illness or injury, or permanent impairment to a body structure or a body function.
- c) Foetal distress, foetal death, a congenital abnormality, or birth defect including physical or mental impairment.

Serious Adverse Events will be collected and reported as described in the Study Procedure Manual.

## 8.9.3 AEs of Special Interest

Given the objective of the study and the disease assessed, AEs of special interest will be collected irrespective of seriousness and relatedness. These AEs are typically ones concerning the motor functions of the patients and include but are not limited to falls, freezing of gait, rigidity, bradykinesia, dyskinesia, dizziness, stiffness, vertigo and in general the worsening of the disease.

#### 8.9.4 Adverse Device Effect (ADE)

An ADE is an adverse event related to the use of an investigational medical device. This definition includes adverse events resulting from; insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device. It also covers any event resulting from use error or from intentional misuse of the investigational medical device.

## 8.9.5 Serious Adverse Device Effect (SADE)

A serious adverse device effect is an adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event (8.7.2). If a serious safety incident occurs related to a device or study procedure, the incident will be recorded in the eCRF and reported to the Ethics Committee as required. Instructions on recording and reporting of serious safety incidents will be provided in the Study Procedure Manual.

#### 8.9.6 Assessment Definitions

## Assessment of Intensity

The investigator must assess the intensity of the safety event using the following definitions:

- Mild the event causes minimal discomfort and does not interfere in a significant manner with the patient's normal activities.
- Moderate the event is sufficiently uncomfortable to produce some impairment of the patient's normal activities.
- Severe the event is incapacitating, preventing the patient from participating in the patient's normal activities.

## Assessment of Causal Relationship

The investigator must assess the causal relationship between the adverse event and the Investigational Medicinal Product (IMP) using the following definitions:

- Probable – the event has a strong temporal relationship to the IMP or recurs on rechallenge, and another aetiology is unlikely or significantly less likely.

- Possible the event has a suggestive temporal relationship to the IMP, and an alternative actiology is equally or less likely.
- Not related the event has no temporal relationship to the IMP or is due to an underlying/concurrent disorder or effect of another drug (that is, there is no causal relationship between the IMP and the adverse event).

An event is considered causally related to the use of the IMP when the causality assessment is probable or possible.

#### Assessment of Outcome

The investigator must assess the outcome of an event using the following definitions:

- Recovered the patient has recovered completely, and no symptoms remain.
- Recovering the patient's condition is improving, but symptoms remain.
- Recovered with sequelae the patient has recovered, but some symptoms remain (for example, the patient had a stroke and is functioning normally, but has some motor impairment).
- Not recovered the patient's condition has not improved, and the symptoms are unchanged
- Death

#### 9 STATISTICAL METHODS AND CONSIDERATIONS

The SAP will provide full details of the analyses, data displays, and algorithms to be used for data derivations. It will be written before the first patient is enrolled in the study. All statistical analyses will be conducted by a blinded independent statistician.

## 9.1 Analysis sets

The Screened set includes all subjects for whom informed consent to participate in the study was obtained and have a subject identification number.

The Full Analysis Set (FAS) includes all subjects randomised to one of the pre-defined treatment arms and who had a baseline gait measurement.

No Per Protocol Set (PPS) is planned to be defined for this study.

The Safety Set (SAF) includes all subjects who were randomised, removing only patients who do not start their assigned therapy.

## 9.1.1 Usage of the analysis sets

The efficacy analysis will be performed on the FAS. The safety analysis will be performed on the SAF.

Table 9.1 outlines the randomised treatment groups and the analysis sets, for each of efficacy and safety.

Table 9.1 Combination of patient cohorts, patient treatment groups and analysis sets

| Randomised treatment group | Efficacy | Safety |
|----------------------------------------------|----------|--------|
| Patient group A (conventional physiotherapy) | FAS | SAF |
| Patient group B (FeetMe Rehabilitation) | FAS | SAF |

## 9.1.2 Short description of endpoints and time periods

The primary and all secondary endpoints are limited to the primary intervention period. The majority of the exploratory endpoints, in line with the exploratory objectives, are related to both the primary and long-term intervention periods.

#### 9.2 Description of statistical analysis

The following sections describe the estimands for the primary and key secondary objectives / endpoints, the overall testing strategies and the overall analysis methods.

#### 9.2.1 Estimands for primary and key secondary objectives

The main treatment policy estimands for the primary and key secondary objectives of this study, are defined in <u>Table 9.2</u> below. This table describes the four attributes of target population, endpoint, strategy for addressing intercurrent events, and population-level summary for the endpoints (ICH E9 (R1)).

Table 9.2 Treatment policy estimands for the primary and key secondary objectives

| Target population | Endpoint | Strategy for addressing intercurrent events | Population-level summary |
|---|---|---|---|
| Primary object | Primary objective in line with H0_1_Primary | | |
| Idiopathic Parkinson's Disease (PD) patients on Conventional Physiotherapy (CPt). | Change from<br>baseline to<br>Week 12 in gait<br>velocity (cm/s)<br>assessed during<br>the 6MWT | All available data to be included. This is in alignment with the FAS definition. If a patient has a fall up to week 12 and has available week 12 gait data, then the week 12 data will be used and the fall ignored. If the week 12 measurement is not available, whatever the reason (death or injury) the baseline data are used (the patient is not excluded). | In Idiopathic PD patients on CPt, what is the change in gait velocity 12 weeks after randomisation, assessed during the 6MWT, between Conventional Physiotherapy and FeetMe Rehabilitation and whilst the patient is on treatment? |
| Key secondary | objective in line w | ith H0_2_KeySecondary | |
| Idiopathic<br>Parkinson's<br>Disease (PD)<br>patients on<br>Conventional<br>Physiotherapy<br>(CPt) | Change from baseline to Week 12 in stance time variability (ms) assessed during the 6MWT. | All available data to be included. This is in alignment with the FAS definition. If a patient has a fall up to week 12 and has available week 12 gait data, then the week 12 data will be used and the fall ignored. If the week 12 measurement is not available, whatever the reason (death or injury) the baseline data are used (the patient is not excluded). | In Idiopathic PD patients on CPt what is the change in stance time variability 12 weeks after randomisation, assessed during the 6MWT, between Conventional Physiotherapy and FeetMe Rehabilitation and whilst the patient is on treatment? |

## 9.2.2 Overall testing strategy

In line with the primary and key secondary objectives of the statistical analysis (see <u>Table 9.2</u>), a confirmatory hierarchical testing procedure will be applied. As a first step, the null hypothesis 'H0\_1\_Primary' will be tested at the 2-sided alpha level of 0.05. If this null hypothesis is rejected, the key secondary endpoint hypothesis 'H0\_2\_KeySecondary' will then be tested in a second step, again using a 2-sided alpha of 0.05.

<u>H0\_1 Primary</u>: The null hypothesis to be tested for the primary endpoint is that the change in week 12 gait velocity from baseline in FeetMe Rehabilitation arm is equal to that in the conventional physiotherapy arm. The alternative is that they are not equal. Superiority will be declared if the difference (FeetMe Rehabilitation vs Conventional Physiotherapy) is significantly greater than 0 at the two-sided type I error level alpha=0.05.

<u>H0\_2 KeySecondary</u>: The null hypothesis to be tested for the key secondary endpoint is that the change in week 12 stance time variability from baseline in FeetMe Rehabilitation arm is equal to that in the conventional physiotherapy arm. The alternative is that they are not equal. Superiority will be declared if the difference (FeetMe Rehabilitation vs Conventional Physiotherapy) is significantly greater than 0 at the two-sided type I error level alpha=0.05.

## 9.2.3 Analysis of the primary efficacy outcome

The primary analysis of the primary endpoint will be performed in line with the primary objective and the treatment policy estimand as outlined in Table 9.2. We will use the constrained longitudinal data analysis (cLDA) model which allows to analyse all available data.

As secondary analysis of the primary end point a sensitivity analysis will be performed excluding patients from the FAS population who have a change in levodopa medication during the first 3 months.

All basic data will be described.

## 9.2.4 Analysis of the key secondary efficacy outcome

The primary analysis of the key secondary endpoint will be performed in line with the key secondary objective and the treatment policy estimand. It will be analysed using the same methods as the primary endpoint.

## 9.2.5 Analysis of other secondary efficacy outcomes

Other secondary efficacy endpoints, all continuous in nature, will be analysed in a similar manner to the primary endpoint. Handling of intercurrent events will be in line with the treatment policy estimands as outlined in Table 9.2.

## 9.2.6 Analysis of exploratory efficacy outcomes

Descriptive methods will be used to summarise the exploratory endpoints. Those continuous in nature will be described using means and standard deviations, medians and their interquartile ranges, including full ranges. Binary endpoints will be presented with their frequencies.

## 9.2.7 Analysis of safety outcomes

The SAF will be used to perform all safety analyses.

If not otherwise stated, only device-related safety data will be considered in tables and figures. All safety data will be included in listings, with flags for safety data not considered to be treatment emergent.

Device-related AEs and SAEs will be tabulated by patient cohorts, SOC, and preferred terms. The events will also be summarized by maximum intensity, relationship to study treatment and outcome (premature discontinuation from treatment).

#### 9.3 Interim analysis

No interim analysis is planned for this study.

## 9.4 Determination of sample size

Sample size calculations have been performed using the software PASS 12.

The main objective of the RE-CONNECT study is to demonstrate the efficacy of FeetMe home-based rehabilitation program compared to conventional physiotherapy at Week 12 in PD patients. The primary endpoint is the change from baseline to Week 12 in gait velocity (cm/s) assessed during the 6 Minutes Walk-Test (6MWT).

The sample size computation is based on the study of Chris J Hass et al (Hass et al, 2014). aiming to determine the Minimal Clinically Important Difference (MCID) for the gait velocity in patients with idiopathic Parkinson's disease. In this study including 324 patients, MCID for gait velocity was classified as small, moderate and large with values of 6 cm/s, of 14 cm/s and 22 cm/s respectively (using a distribution-based analysis and the categorization defined by Cohen (Cohen et al, 1988.)). We aim to show that the Feetme rehabilitation procedure will allow to improve the change in gait speed at least in a moderate range in comparison with that in standard rehabilitation group and we set the difference to

be detected at 14 cm/s. In the Chris J Hass et al, the standard deviation of gait velocity was estimated at 27cm/s.

To detect a difference of 14cm/s between the two groups for the change in velocity with a standard deviation of 27cm/s for the change from baseline to Week 12 in gait speed (assuming a conservative correlation coefficient of 0.5 between the measures at baseline and at week 12), 60 patients per group are needed (two-sided Student's test, type I error of 0.05 and a power of 80%). To take into account a 20% rate of drop out for the measurement of the gait velocity at week 12 (based on previous studies using FeetMe Rehabilitation application on a similar population, 15% of lost to follow up and 5% of deaths or injuries), we plan to recruit 75 patients per group (a total of 150 patients).

## 9.5 Statistical analysis

Baseline characteristics will be described according treatment groups. Quantitative variables will be expressed as mean (standard deviation) or median (interquartile range) for non-Gaussian distribution. Categorical variables will be expressed as frequencies and percentages. Normality of distribution will be assessed graphically and using the Shapiro-Wilk test. The number of missing data will be also reported. No formal statistical comparisons will be done; clinical importance of any imbalance will be noted.

## 9.5.1 Analysis for the primary endpoint

The primary outcome (the change in the gait velocity between baseline and week 12, assessed during the 6 Minutes Walk-Test) will be estimated and compared between Feetme rehabilitation and conventional physiotherapy groups using the constrained longitudinal data analysis (cLDA) model proposed by Liang and Zeger including centre as random effect and adjusted for the covariable "already in a rehabilitation program" considered as stratification factor in the randomisation. We chose to use cLDA model in view of its potential advantages compared to the conventional ANCOVA model. First, the cLDA model provides more flexibility in handling missing data by including all observed data, which, in general, results in more power when testing treatment differences compared with the longitudinal ANCOVA model. Second, compared with the ANCOVA model, the cLDA model provides more appropriate confidence interval estimates, especially in the context of randomised clinical trials where proper randomisation ensures baseline balance. In the cLDA model, both the baseline and postbaseline values are modelled as dependent variables using a linear mixed model (using an unstructured covariance pattern model), and the true baseline means are constrained to be the same for the 2 treatment groups. The between-group mean differences in 12-week change in gait velocity will be estimated by the time-by-arm interaction as treatment effect size. The assumptions of the cLDA model will be checked. We will use the analysis of cDLA model residuals by examining graphically the normality of residuals (histogram and Quantile-quantile plot) and by using the Shapiro Wilk test. In case of strong departure from the normality assumptions (even after applying a logarithmic transformation), nonparametric analysis will be used as recommended by Vickers et al. (reference: 1) Andrew J Vickers. Parametric versus non-parametric statistics in the analysis of randomised trials with non-normally distributed data. BMC Medical Research Methodology 2005, 5:35 2) Conover WJ, Iman RL: Analysis of covariance using the rank transformation. Biometrics 1982, 38:715-724.); absolute changes between baseline and 12-week will be calculated and compared between the 2 treatments groups using nonparametric analysis of covariance adjusted for baseline values. The effect size will be assessed by Hedges's g (standardized differences) computed on rank transformed data with its 95% confidence interval (using the method based on noncentral Student distribution which is a corrected version of Cohen's d taking into account the sample size). A sensitivity analysis will be performed excluding from the FAS population patients who have a change in levodopa medication during the first 3 months. For this sensitivity analysis, we will use the same methodology as that described for the primary analysis.

## 9.5.2 Analysis for the secondary endpoints

The statistical method described for the primary objective will be used for the analysis of the following secondary endpoints:

- Change from baseline to Week 12 (Visit 3) in Stance Time Variability assessed during the 6 Minutes Walk Test (6MWT).
- Change from baseline to Week 12 (Visit 3) in the asymmetry of the swing duration assessed during the 6 Minutes Walk Test (6MWT).
- Change from baseline to Week 12 (Visit 3) in the MiniBESTest.
- Change from baseline to Week 12 (Visit 3) in MDS-UPDRS part III sub-score.
- Change from baseline to Week 12 (Visit 3) the results of the Parkinson Disease Questionnaire (PDQ-39)

The rate of falls during the primary intervention period will be compared between the 2 groups using a generalized linear model (GLM with log link function and negative binomial distribution) with the logarithm of duration of patient's follow up (censored at week 12) as offset variable. Effect size will be estimated by the relative risk ((Feetme rehabilitation versus conventional rehabilitation) and it's 95% confidence interval from the using GLM model.

## 9.5.3 Exploratory analysis

Inferential analysis will not be performed if the smallest group involving in the comparison has a size smaller than 10.

To explore the long term efficacy of FeetMe home-based rehabilitation program compared to conventional physiotherapy in patients who continue to Week 24, the following will be applied:

The change in gait velocity and Stance Time Variability from baseline to week 24 will be compared between the Feetme group and the conventional rehabilitation group using the constrained longitudinal data analysis (cLDA) model or a non-parametric analysis of covariance in case of violation of the assumption of cLDA model, as indicated for the primary objective. The change in these 2 parameters from week 12 to week 24 will be compared using the linear mixed model with an adjustment on the value at week 12 and on the covariable used in the stratified randomisation "conventional physiotherapy in progress". In this model, the centre will be included as a random effect. The rate of falls assessed within 24 weeks will be compared between the two groups using the generalized linear model (GLM with log link function and negative binomial distribution) with the logarithm of duration of patient's follow up (censored at week 24) as offset variable.

All other endpoints will be analysed using descriptive statistics:

- To explore the maintenance of the effect after 3 months in patients who stop physiotherapy at Week 12, the method described previously will be employed for the analysis of the first exploratory objective, namely inferential analysis for the three parameters gait velocity, stance time variability and rate of falls and descriptive analyses for the other endpoints.
- To explore the efficacy in patients who switch from one treatment to the other at Week 12, descriptive analyses will be performed.

#### 10 DATA HANDLING

#### 10.1 Data Monitoring Committee

No Data Monitoring Committee is planned for this study.

#### 10.2 Gait Data Collection and Management

Gait Data are collected and processed internally by FeetMe according to Standard Operating Procedures on data management.

## 10.3 Clinical Data Collection and Monitoring

Clinical data – other than gait data – will be entered by the site into an electronic data capture system (EDC) by completing the eCRF via a secure internet connection. Data entered into the eCRF must be verifiable against the source documents at the study centre. Any changes to the data entered in the EDC will have an audit trail. Missing or inconsistent data will be queried via the system to the Investigator for clarification. Subsequent modifications to the database will be documented.

Monitoring of this study is the responsibility of the Sponsor and may be delegated to a CRO or a contract monitor. It is understood that the study Sponsor and/or its appointee will regularly contact the Investigator and conduct onsite visits at the study site with the purpose of maintaining compliance with this clinical investigational plan, GCP and all relevant regulatory requirements.

The Investigator agrees that the Sponsor and/or Sponsor-authorised personnel will be allowed to inspect all records pertinent with the study and to have direct access to patient files (provided that subject confidentiality is maintained, in accordance with local laws and regulations) with the aim of verifying eCRF entries, their completeness and clinical investigational plan compliance.

The Investigator also agrees to cooperate with the monitor's activities when requested and to coordinate with the monitor to ensure that any issue uncovered in the course of such visits are analysed and solved.

The Investigator agrees to supply the Sponsor with relevant original data from the clinical records or study documentation, especially in case doubts about data transcription should arise. Complete access to the study records is as well required in case of audit inspections and inquiries from competent national or local authorities, provided that confidentiality of the study patients is protected.

A clinical site monitoring plan, including all details about the monitoring strategy will be provided to the Investigator.

#### 10.4 Record Retention

The Investigators will retain all study records for a minimum of 15 years after the conclusion of the study, or, alternatively, for a period of time meeting the local, regional, or national standards; whichever is greater. The Investigator will be responsible for maintaining adequate and accurate electronic or hard copy source documents of all observations and data generated during this trial including any data clarification forms received from the Sponsor. Such documentation is subject to inspection by the Sponsor and relevant regulatory authorities.

Before proceeding with the destruction of the study records or any study-related document, the Investigator must contact the Sponsor and receive explicit authorisation from the Sponsor to destroy such records. This notification must happen even if retention requirements have been met. A notification must be provided to the Sponsor prior to the transferring of any study records to another party or moving them to a new location.

Should the Investigator leave the clinical site of this study, a notification must be provided to the Sponsor in a timely manner, allowing for suitable arrangements to be made, aimed at ensuring the retainment of all study records and maintaining continuing access to the study records for the Sponsor and Regulatory authorities. Notice of such transfer will be given to the Sponsor in writing.

## 10.5 Reporting and Publication

The Sponsor will register this study and its results on a public online repository (e.g. Clinicaltrials.gov) regardless of the outcome, in accordance with the applicable laws.

All type(s) of publication (including presentations at scientific meetings) of any results derived from this study is only permitted if the publication is approved by the Sponsor. Published data must not compromise the objectives of the study. If the publication is initiated by the Investigator, s/he agrees to provide relative abstracts and manuscripts to the Sponsor prior to any submission activity. This has the purpose of protecting possible Sponsor's confidential or proprietary information and/or to allow the Sponsor to share information from other clinical studies which may be unknown to the Investigator. Investigators who do not qualify for authorship may be acknowledged in publications resulting from the trial. By agreeing to participate in the trial, Investigators consent to such acknowledgement in any publications resulting from its conduct.

All type(s) of publication of any results derived from this study is only permitted if the publication is approved by the Sponsor. Published data must not compromise the objectives of the study.

All information concerning this study which was not previously published is to be considered confidential property of the Sponsor and must not be disclosed without express consent.

The Sponsor is responsible for producing the clinical study report in compliance with ICH E3.

## 11 QUALITY ASSURANCE AND QUALITY CONTROL

Measures to ensure quality and completeness of the data will be implemented by the Sponsor, in order to assure that all data are reliable and have been correctly processed. The Sponsor, CRO and data management vendor will be responsible for the management of data for this study. The Investigator will be responsible for the correct recording of study data in the eCRF using the EDC system and for approving all eCRF data before final database lock.

Over the course of the study, as well as after completion, quality assurance officers appointed by the Sponsor or pertinent authorities may perform inspections and audits. The Investigator has the responsibility of cooperating and facilitating such inspections as well as to provide relevant documents if requested. In the event of discrepancies in data, the study site will be queried in order to resolve them through the EDC system.

## 12 ETHICS

## 12.1 Independent Ethics Committee or Institutional Review Board

The Sponsor must obtain approval of this clinical investigational plan and any relevant study material (e.g., ICF) from the Independent Ethics Committee before starting the study. Approval from the committee must be documented in writing, in the form of a letter to the study Sponsor before the study can start, specifying the date of approval.

Any modification to this clinical investigational plan or relevant study material after EC approval must be re-submitted by the Sponsor to the committee in accordance with local or national regulatory requirements.

## 12.2 Regulatory Authorities

Notifications and submissions to the appropriate regulatory Authorities will be executed as prescribed by national or local legislation in the country where this study is taking place.

## 12.3 Ethical Conduct of the Study

This study will comply and will be conducted in full conformance with the ICH E6 guideline for Good Clinical Practice, with the principles stated in the World Medical Association's Declaration of Helsinki, MDR 2017/745 and MPDG, ISO 14155, 2020 and all applicable local, regional, and national laws or regulations of the country in which the research is conducted.

#### 12.4 Informed Consent

Prior to any data collection for this study, each subject will be informed in detail about the study device and the nature of the clinical investigation, with particular care given to any potential risks or discomforts to be expected by the subjects.

The Sponsor's Informed Consent Form (ICF) will be provided to the study site. The ICF will be provided in a certified translation of the local language.

It is the responsibility of the Investigator to obtain written subject informed consent from any subject considering participation in this study by using the approved ICF. The consent forms must be signed and dated by the subject before any study procedure is initiated.

The Investigator must also explain to any potential subject candidate that they are completely free to refuse to enter the study, or to withdraw at any time without having to give any explanation. The Investigator must further explain to any potential subject candidate that, should they refuse to enter the

study or withdraw from it, their standard of care will not be subject to any change. Patients who decline to participate will not provide any signature.

Each patient will receive a copy of their signed and dated ICF, while the original will be kept with the study records. If applicable, the Investigator or other authorised staff must document the date of informed consent of each subject in the eCRF. Confirmation of informed consent must also be documented in the medical record of the subject.

The ICF should be revised whenever there are changes to the study procedures, in case new safety information changes significantly the risk/benefit assessment or when there is the possibility that such changes may affect the disposition of the subject towards participation in the study. In any of such cases, the ICF should be reviewed, updated, and approved by the EC. To ensure its continued participation to the study, the subject must re-consent to the most updated approved version of the ICF.

#### 12.5 Patient Confidentiality

The Sponsor of this study will maintain the highest confidentiality standards, ensuring patient's anonymity and protecting their identities from unauthorised parties. Through this study, each patient will be identified through the assignment of a unique identification number (i.e. Patient ID) on all study documents and electronic databases. All study-related documents will be securely stored and accessible only by the Investigator, the study staff, and authorised personnel. No personal detail will be included in any data transmitted to the Sponsor.

Any medical information pertaining to the patients is considered confidential and may be only disclosed to third parties as permitted by the ICF, once dated, and signed by the patient.

#### 12.6 Data Protection

Before any data can be collected in the context of this trial, all patients must provide all pertinent authorisations, as per local or national law. Additionally, each patient will be informed about their rights regarding access, objection and correction to any of their data recorded during the course of the study. Every database is GDPR compliant.

#### 12.7 Financing and Insurance

The Sponsor is financially responsible for the conduct of the study.

The Sponsor has an insurance policy for the duration of the study, covering subjects and Investigators in respect to the risks involved in conducting this study according to this clinical investigational plan. The insurance policy can be made available to the Investigator and the EC upon request.

## 13 STUDY PERSONNEL AND ADMINISTRATIVE STRUCTURE

The Sponsor of this trial is FeetMe. Six study centres will participate in this study to recruit approximately 150 patients. The Sponsor will be responsible for data management, statistical analysis and medical oversight.

A contract research organisation (CRO) will be contracted and will be responsible for the administrative aspects of the study. This includes but is not limited to: initiation of the study, management and monitoring of the study and data monitoring.

#### 14 APPENDICES

#### 14.1 Appendix A – Rehabilitation Exercises

During the static exercises the phone should be positioned at eye level and an object to provide the patient with support should be placed nearby (e.g.: a chair to hold on to). For the dynamic exercises the patient should keep the phone in their pocket.

#### 14.1.1 Static Exercises

#### 14.1.1.1 Balance

#### **Support Transfer**

The objective of this exercise is to improve multi directional support transfer. The task is to catch the targets appearing on the screen by moving the centre of gravity without moving the feet on the ground. The patient should reach the highest number of targets during the allocated time. The exercise has six difficulty levels across which the amplitude of the movement required to reach a target increases and the directions of the transfer support needed become more complex. The biofeedback given includes the total number of targets reached and the percentage of success.

#### **Stabilization**

The objective of this exercise is to reinforce balance by working on stabilising the body. The task is to catch the targets appearing on the screen by moving the centre of gravity without moving the feet on the ground and then to maintain the position for 5 to 7s until the object disappears and repeat this as many times as possible during the allocated time. The exercise has six difficulty levels across which the amplitude of the movement required to reach a target increases and the directions of the transfer support needed become more complex. The biofeedback given includes the total number of targets on which the patient stabilized and the percentage of success.

## Balance and speed

The objective of this exercise is to improve the speed of transfer support to facilitate daily activities. The task is to catch the targets appearing on the screen as quick as possible by moving the centre of gravity without moving the feet on the ground. Targets that are not reached within 5 seconds will automatically disappear and will be regenerated somewhere else. The patient should reach the highest number of targets during the allocated time. The exercise has six difficulty levels across which the amplitude of the movement required to reach a target increases and the directions of the transfer support needed become more complex. The biofeedback given includes the total number of targets reached and the percentage of success.

## 14.1.1.2 Muscle strengthening

#### **Plantar flexion**

The objective of this exercise is to reinforce the lower limbs to facilitate balance and walking. The task is to move the centre of gravity forward towards the toes from a position of having both feet flat on the ground to lifting the heels off. A gauge is displayed on the screen during the exercise and the patient should fill the gauge as much as possible. Each time the patient puts more than 85% of their weight on the front sensors of the insoles the plantar flexion is indicated as done. The biofeedback given includes the total number of movements completed and the percentage of success.

#### Sit to Stand

The objective of this exercise is to reinforce muscle strength and improve postural symmetry. The task is to stand up from sitting position and sit back down completely with equally distributed body weight on both feet. The patient should complete as many sit to stand rounds as possible during the time allocated. The biofeedback given includes the total number of rounds correctly performed and the distribution of the pressure on each leg.

#### 14.1.2 Dynamic Exercises

#### 14.1.2.1 Gait Quality

#### **Big Step**

The objective of this exercise is to improve balance and walking. The task is to walk with the longest possible stride length. Prior to the task the patient needs to perform a thirty second comfortable walk to set the baseline for the evaluation of success and to serve as a basis for recalibrating the difficulty level by assessing their natural stride length. A stride is considered successful if it is at least fifteen percent longer than the average natural step. As the patient improves their gait quality throughout the program they will need to keep doing better compared to their actual status. The biofeedback given includes the percentage of success that is calculated in comparison to the patient's regular stride length using a specific formula.

## **Step Sequence**

The objective of this exercise is to improve gait quality. The task is to preform steps which follow the sequence of heel-strike – full contact with the ground – toe-off (propulsion). If any of the components of the sequence is missing it will not be counted. The biofeedback given is the percentage of success for the left and right foot separately.

#### 14.1.2.2 Endurance

#### **Rhythmic Stimulation**

The objective of this exercise is to improve the velocity and to regulate cadence. The task is to follow the pace of a metronome. Prior to the task the patient needs to perform a thirty second comfortable walk to set the baseline for the evaluation of success and to serve as a basis for recalibrating the difficulty level by assessing the natural cadence. The metronome is set to a pace ten percent higher than assessed during this regular walk. The biofeedback given includes the percentage of success and the reached cadence versus the target one.

#### **Heel Strike**

The objective of this exercise is to improve gait quality and endurance. The task is the same as during the Step Sequence (walk at a normal pace starting each step with a heel strike and finishing with toe-off), only for a longer duration. Therefor, an additional objective of this task is to assess whether gait quality decreases over time.

#### Free Walking

The objective of this exercise is to improve endurance and to assess gait evolution by all the spatiotemporal and pressure parameters. The patient will need to perform comfortable pace walking for the duration defined in their allocated program (e.g.: sixty minutes per week). Patients can distribute the total time to be completed at their convenience.

## 14.2 Appendix B – Rehabilitation Program

## 14.2.1 Decision Tree for Initial Program



## 14.2.2 Program Adaptation Principles



## 14.2.3 Program A

| Periods | Nb<br>sessions | Duration of sessions | Free<br>walking<br>/ week | Total<br>weekly<br>time | |
|---|---|---|---|---|---|
| W1-W3 | 4x/week | 30min | 60min | =3h | |
| W4-W6 | 4x/week | 45min | 60min | =4h | |
| W7-W9 | 4x/week | 60min | 60min | =5h | |
| W10-W12 | 4x/week | 60min | 60min | =5h | Intensity<br>level |
| W12-W24<br>(if the patient pursues) | 4x/week | 60min | 60min | =5h | |

## 14.2.4 Program B

| Periods | Nb<br>sessions | Duration of<br>sessions | Free<br>walking<br>/ week | Total<br>weekly<br>time |
|---|---|---|---|---|
| W1-W3 | 3x/week | 30 <i>min</i> | 60min | =2h3o |
| W4-W6 | 4x/week | 30min | 60min | =3h |
| W7-W9 | 4x/week | 45min | 60min | =4h |
| W10-W12 | 4x/week | 60min | 60min | =5h |
| W12-W24<br>(if the patient pursues) | 4x/week | 60min | 60 <i>min</i> | =5h |

## 14.2.5 Program C

| Periods | Nb<br>sessions | Duration of sessions | Free<br>walking<br>/ week | Total<br>weekly<br>time | |
|---|---|---|---|---|---|
| W1-W3 | 3x/week | 30 <i>min</i> | 30min | =2h | |
| W4-W6 | 4x/week | 30min | 30min | =2h3o | |
| W7-W9 | 4x/week | 45 <i>min</i> | 30min | <b>=</b> 3 <i>h</i> 3 <i>o</i> | |
| W10-W12 | 4x/week | 60min | 30min | =4h3o | Intensity<br>level |
| W12-W24<br>(if the patient pursues) | 4x/week | 60min | 30min | <del>-</del> 4h3o | |

## 14.3 Appendix C – FeetMe Satisfaction Questionnaire for Initial Patient Training

A compléter après la formation initiale.

| 1) | Le temps | de | formation | était-il | suffisant | ? |
|----|----------|----|-----------|----------|-----------|---|
|----|----------|----|-----------|----------|-----------|---|

- o Oui complètement
- o Plutôt oui
- Je ne sais pas
- o Plutôt non
- o Non pas du tout

| 2) | Suite à | la f | ormation | initiale, | vous | êtes- | vous | senti | en | confiance | conc | ernant | l'utilisation | du | disposi | tif |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ? | | | | | | | | | | | | | | | | |

- o Oui complètement
- o Plutôt oui
- o Je ne sais pas
- o Plutôt non
- Non pas du tout
- 3) Le format par visio-conférence de la formation était-il satisfaisant ?
  - o Oui complètement
  - o Plutôt oui
  - o Je ne sais pas
  - o Plutôt non
  - o Non pas du tout
- 4) Les informations communiquées lors de la formation initiale ont-elles été claires ?
  - o Oui complètement
  - o Plutôt oui
  - o Je ne sais pas
  - o Plutôt non
  - Non pas du tout
- 5) Sur une échelle de 0 à 10, quelle note donneriez-vous à cette formation initiale ?
- 6) Selon vous, comment pourrions-nous améliorer cette formation initiale?

## 14.4 Appendix D – FeetMe Satisfaction Questionnaire – Patient Version

A compléter à Visite 3 et à Visite 4, si applicable.

#### Questions spécifiques au programme

- 1) Les objectifs du programme sont-ils en accord avec mes objectifs personnels (ex: sortir en autonomie pour faire des courses ou bien se promener) ?
  - o Tout à fait d'accord
  - o D'accord
  - o Pas d'avis
  - o Pas d'accord
  - o Pas du tout d'accord
- 2) Quelle est pour vous la valeur ajoutée de FeetMe Rehabilitation dans votre vie quotidienne ? (plusieurs réponses possibles)
  - o Exercices personnalisés
  - o Je peux pratiquer quand et où je veux
  - o Un suivi téléphonique régulier personnalisé
  - o Éviter les déplacements
  - o Me permet de pratiquer davantage
  - o Me motive
  - o Non applicable
  - o Autre:
- 3) Lorsque vous utilisez FeetMe Rehabilitation, vous sentez-vous en sécurité lors de la réalisation des exercices ?
  - o Tout à fait d'accord
  - o D'accord
  - o Pas d'avis
  - o Pas d'accord
  - o Pas du tout d'accord
- 4) Quel est votre niveau de satisfaction en ce qui concerne le suivi?
  - o Très satisfait
  - Plutôt satisfait
  - o Ni satisfait, ni insatisfait
  - o Plutôt insatisfait
  - o Insatisfait
- 5) Si vous deviez changer quoi que ce soit concernant le suivi, qu'est ce que ce serait ? (ex: la fréquence, la durée, le contenu..)
- 6) Quel est votre niveau de satisfaction concernant votre relation avec l'APA en charge de votre suivi
  - Très satisfait
  - o Plutôt satisfait
  - o Ni satisfait, ni insatisfait
  - o Plutôt insatisfait
  - Insatisfait

- 7) Parmi les propositions suivantes, quel moyen de rééducation préférez-vous ?
  - o Rééducation à domicile
  - o Rééducation chez le kinésithérapeute
  - Une combinaison des deux
  - Non applicable
- 8)Recommanderiez-vous la solution à quelqu'un qui se trouve dans la même situation que vous ?
  - Très probablement
  - Probablement
  - Je ne sais pas
  - o Probablement pas
  - Très probablement pas

## Questions spécifiques au matériel

- 1) Quel est votre niveau de satisfaction en ce qui concerne l'utilisation de la solution FeetMe Rehabiltation ? (semelles, application, chargeur)
  - Très satisfait
  - Plutôt satisfait.
  - O Ni satisfait, ni insatisfait
  - o Plutôt insatisfait
  - o Insatisfait
- 2) Quel est votre niveau de satisfaction en ce qui concerne l'utilisation des semelles FeetMe (confort, utilisation...)
  - o Très satisfait
  - Plutôt satisfait
  - O Ni satisfait, ni insatisfait
  - o Plutôt insatisfait
  - Insatisfait
- 3) Si vous pouviez changer quoi que ce soit sur les semelles FeetMe Monitor, qu'est ce que ce serait ? (ex: matériau, couleur, forme, chargeur, etc)?
- 4) Si vous pouviez changer quoi que ce soit concernant l'application FeetMe rehabilitation, qu'est ce que ce serait ? (ex: interface, retour en temps réel, menu, etc...) ?
- 5) Avez-vous rencontré des difficultés lors de l'utilisation ? Si oui, lesquelles ?
- 6) Quel est votre niveau de satisfaction concernant l'assistance technique ?
  - o Très satisfait
  - o Plutôt satisfait
  - o Ni satisfait, ni insatisfait
  - Plutôt insatisfait
  - o Insatisfait

## 14.5 Appendix E – Satisfaction Questionnaire – Investigator Version

A compléter à la fin de l'étude.

| 14.5 | 5.1 Application FeetMe Evaluation application et semelles FeetMe Monitor |
|---|---|
| | <ol> <li>Comment trouvez-vous l'utilisation de la solution ?</li> <li>Très simple d'utilisation</li> </ol> |
| 0 | Plutôt facile d'utilisation Ni facile ni difficile d'utilisation |
| | Plutôt difficile d'utilisation |
| | Très difficile à utiliser |
| | 2. A quelle fréquence intégrez-vous l'utilisation de la solution dans votre pratique quotidienne ? |
| | Très souvent<br>Souvent |
| | Neutre |
| | Pas souvent |
| | Rarement |
| | 3. Pour quelle raison implémentiez-vous cette solution ? |
| | Expliquer certaines choses et faire des retours aux patients |
| | Suivre l'évolution de l'avancée de la maladie<br>Guider la rééducation ou le traitement |
| | Autre : |
| | NA |
| | 4. De 0 à 10, dans quelle mesure êtes-vous susceptible de recommander la solution FeetMe Evaluation à vos collègues ? (0: je ne recommande pas FeetMe, 10: je recommande absolument) |
| | 5 Oud est victue divisor de estisfection concernant le mulité des compiles FeetMe Meniter 0 |
| | <ol> <li>Quel est votre niveau de satisfaction concernant la qualité des semelles FeetMe Monitor?</li> <li>Très satisfait</li> </ol> |
| | Plutôt satisfait |
| | Ni satisfait, ni insatisfait Plutôt insatisfait |
| | Insatisfait |
| | 6. Quel est votre niveau de satisfaction concernant la qualité des de l'application FeetMe |
| _ | Evaluation ? Très satisfait |
| _ | Plutôt satisfait |
| | Ni satisfait, ni insatisfait |
| | Plutôt insatisfait<br>Insatisfait |
| _ | |
| | 7. Si vous pouviez changer quelque chose sur l'application FeetMe Evaluation, qu'est-ce que ce<br>serait ? (ex : interface, menu, etc)? |
| | 8. Si vous pouviez changer quelque chose sur les semelles FeetMe Minitor, qu'est-ce que ce serait (ex.: matière, couleur, forme, mode de chargement, etc)? |
| | (ex.: mattere, content, forme, mode de chargement, etc): |
| | 9. Avez-vous rencontré des difficultés ? Si oui précisez lesquelles |

□ Insatisfait

| 0 0 | 10. Quel est votre niveau de satisfaction concernant le support technique ? Très satisfait Plutôt satisfait Ni satisfait, ni insatisfait Plutôt insatisfait Insatisfait |
|---|---|
| Fe | etMe Rehabilitation |
| | 1. Quel a été le niveau de satisfaction de vos patients le programme FeetMe Rehabilitation ? |
| 0 | Très satisfait Plutôt satisfait Ni satisfait, ni insatisfait Plutôt insatisfait Insatisfait |
| | <ol> <li>Avez-vous observé une amélioration globale des patients grâce à FeetMe Rehabilitation?<br/>(Oui/Non)</li> </ol> |
| 2.<br>gro | Comment les patients dans le groupe FeetMe Rehabilitation se comparent-ils aux patients dans le<br>oupe kinésithérapie conventionnelle en termes de progression ? |
| 0 | Beaucoup plus de progrès<br>Plus de progrès |
| | Identique<br>Moins de progrès<br>Beaucoup moins de progrès |
| Ve | uillez expliquer pourquoi selon vous : |
| | <ol> <li>De 0 à 10, dans quelle mesure êtes-vous susceptible de recommander la solution FeetMe<br/>Rehabilitation à vos collègues ? (0: je ne recommande pas FeetMe, 10: je recommande<br/>absolument)</li> </ol> |
| 4. | Si la solution était remboursée, quelle serait la probabilité que vous la proposeriez à vos patients ? |
| | Très souvent<br>Souvent |
| | Neutre |
| | Pas souvent<br>Rarement |
| 6.<br>en | Quel est votre niveau de satisfaction concernant la solution Rehabilitation ? (ex: interface, retour temps réel, programme, plateforme web, etc)? |
| | Très satisfait |
| | Plutôt satisfait<br>Ni satisfait, ni insatisfait |
| | Plutôt insatisfait |

| | Si vous pouviez changer quelque chose sur la solution FeetMe Rehabilitation, qu'est-ce qu'ex: composition des exercices, l'interface, les retours en temps réel, le menu, etc?) | e ce |
|---|---|---|
| 8.<br>des séa | Si vous pouviez changer quelque chose sur les programmes, qu'est-ce que ce serait (ex : fréquences, les règles d'adaptation, la fréquence des suivis, etc) | ence |

## 14.6 Appendix F – Conventional Physiotherapy Tracking Sheet

A remplir tout au long de la durée de l'étude.

## Fiche de suivi kinésithérapie

| ID Patient: | | |
|---|---|---|
| Date de la séance<br>(DD/MM/YY) | Durée de la séance<br>(heure) | Type d'exercice de rééducation réalisé |
| // | | |
| // | | |
| / | | |
| // | | |
| / | | |
| // | | |
| // | | |

## Instructions pour compléter le formulaire

Vous devez remplir ce formulaire car vous suivez une rééducation conventionnelle chez un kinésithérapeute. Nous vous demandons de garder une trace de votre traitement en l'enregistrant selon les instructions ci-dessous durant toute la durée de l'étude. Vous pouvez demander à votre kinésithérapeute de remplir le formulaire pour vous ou de vérifier les informations que vous avez renseignées. Si vous n'avez plus de place, veuillez en informer votre site pour vous fournir un nouveau formulaire.

Nous vous demandons de bien vouloir :

- mettre votre identifiant patient en haut du formulaire.
- mettre la date de votre séance de kinésithérapie dans la première colonne. Seules les séances qui ont un impact sur vos mouvements sont à renseigner. Si vous recevez un autre traitement (ex : orthophonie), il n'est pas nécessaire de remplir ce formulaire.
- mettre la durée de la séance dans la deuxième colonne.
- décrire les exercices que vous réalisez au cours de la séance.

Merci de rapporter ce formulaire lors de vos visites en centre et de le donner à votre évaluateur.

#### Exemple:

| Date de la séance<br>(DD/MM/YY) | Durée de la séance<br>(heure) | Type d'exercice de rééducation réalisé |
|---|---|---|
| 14/04/2023 | 1.5 | Exercices d'équilibre<br>Entrainement endurance |
| 21/04/2023 | 1 | Vélo d'intérieur, étirements |

## 14.7 Appendix G – Falls Diary

A compléter tout au long de la durée de l'étude.

## Carnet de chute du patient

| Identifiant / ID Patient: | | | | | | | |
|---|---|---|---|---|---|---|---|
| Date de l'évènement<br>(DD/MM/YY) | Nombre<br>de chutes | Nombre de chutes de type | | | | Nombre de | Nombre de |
| | | A | В | С | D | « presque<br>chutes » | Déséquilibre rattrapé<br>par l'aidant |
| / | | | | | | | |
| // | | | | | | | |
## Guide de remplissage du carnet de chutes

Vous devez remplir ce carnet de chutes au cours de l'étude.

#### L'identification du carnet doit comporter :

- Le numéro de patient qui vous aura été attribué
- La date à laquelle la « chute » / « presque chute » / « déséquilibre rattrapé par l'aidant » est survenue.

#### Les informations attendues le jour où l'évènement est survenu sont:

- Le nombre de types de « chute » / « presque chute » / « déséquilibre rattrapé par l'aidant »
- Le nombre de chutes par gravité => seules les « chutes » sont concernées, identifier pour chacune par leur gravité : A, B, C ou D

#### Définition des chutes :

La chute est définie comme le fait de se retrouver involontairement sur le sol ou dans une position de niveau inférieur par rapport à sa position de départ.

La presque chute est définie comme le fait de se rattraper à un objet pour éviter de tomber ou de se rattraper spontanément sans objet.

Le Déséquilibre rattrapé par l'aidant est définie comme le fait que l'aidant intercepte le patient avant qu'il ne tombe.

#### Les différentes gravités de chutes sont les suivantes :

- A Blessure sérieuse : fractures enregistrées médicalement, blessure interne ou blessure de la tête nécessitant un passage aux urgences ou une hospitalisation.
- **B Blessure modérée** : Contusion, entorse, coupure, nécessitant une consultation par un professionnel médical ou de santé, examen tel que examen clinique, radiographies, sutures.
- C Blessure mineure : Contusion ou écorchure ne requérant pas l'assistance d'un professionnel, diminution des fonctions physiques (due à la douleur ou à la peur de chuter) pendant au moins trois jours.
- D Pas de blessure : Aucune blessure physique détectée.

#### Par exemple:

| Date de l'évènement | Nombre | Nombre de chutes de type | | | | Nombre de | Déséquilibre |
|---|---|---|---|---|---|---|---|
| (DD/MM/YY) | de chutes | A | В | С | D | « presque<br>chutes » | rattrapé par<br>1'aidant |
| 05/03/23 | 1 | | | 1 | | | |
| 23/05/23 | | | | | | 2 | |

### 14.8 Appendix H – Visual analog scale

A remplir à chaque visite : Baseline, Visite 1, Visite 2, Visite 3 et Visite 1.2, Visite 2.2, Visite 4 si applicable.

Cette échelle est la plus utilisée des méthodes d'évaluation de la douleur. Elle se présente le plus souvent sous forme d'une réglette comportant deux faces :

- Une face que l'on présente au patient ou se trouve un trait horizontal de 10 cm avec à chaque extrémité un qualificatif, à gauche "pas de douleur", à droite "douleur maximale imaginable",
- Une face évaluateur, gradué de 0 à 10 cm ou de 0 à 100mm

### Mode d'emploi :

On demande au patient de déplacer le curseur figurant sur la réglette et le soignant relève le chiffre correspondant à l'endroit où le patient a placé ce curseur.



#### Interprétation :

Le patient nécessite une prise en charge de la douleur si EVA  $\geq$  4/10 (échelle de 0 à 10 en cm) ou EVA  $\geq$  40/100 (échelle de 0 à 100 en mm).

### 14.9 Appendix I – Parkinson disease questionnaire-39

A compléter à Baseline, Visite 3 et Visite 4, si applicable.

Au cours de la dernière semaine,

#### 1. Avez-vous eu des difficultés dans la pratique de vos loisirs ?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 2. Avez-vous eu des difficultés à vous occuper de votre maison : ménage, cuisine, bricolage, ...

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- O Toujours, ou ne peut jamais faire (4)

#### 3. Avez-vous eu des difficultés à porter des sacs de provisions ?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 4. Avez-vous eu des problèmes pour faire 1 km à pied ?

- o Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 5. Avez-vous eu des problèmes pour faire 100 m à pied ?

- o Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

# 6. Avez-vous eu des problèmes à vous déplacer chez vous, aussi aisément que vous l'auriez souhaité ?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 7. Avez-vous eu des problèmes à vous déplacer dans les lieux publics ?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 8. Avez-vous eu besoin de quelqu'un pour vous accompagner quand vous sortez?

- 1. Jamais (0)
- 2. Rarement (1)
- 3. Parfois (2)
- 4. Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 9. Avez-vous eu peur ou avez-vous été inquiet à l'idée de tomber en public ?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 10. Avez-vous été confiné(e) chez vous plus que vous ne l'auriez souhaité ?

- o Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 11. Avez-vous eu des difficultés pour vous laver ?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 12. Avez-vous eu des difficultés pour vous habiller?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 13. Avez-vous eu des difficultés pour boutonner vos vêtements ou pour lacer vos chaussures ?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 14. Avez-vous eu des difficultés pour écrire lisiblement ?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- O Toujours, ou ne peut jamais faire (4)

#### 15. Avez-vous eu des difficultés pour couper la nourriture ?

- o Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 16. Avez-vous eu des difficultés pour tenir un verre sans le renverser ?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 17. Vous êtes-vous senti(e) déprimé(e) ?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 18. Vous êtes-vous senti(e) isolé(e) et seul(e)?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 19. Vous êtes-vous senti(e) au bord des larmes ou avez-vous pleuré?

- o Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 20. Avez-vous ressenti de la colère ou de l'amertume ?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 21. Vous êtes vous-senti(e) anxieux(se)?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 22. Vous êtes-vous senti(e) inquiet(e) pour votre avenir?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- O Toujours, ou ne peut jamais faire (4)

### 23. Avez-vous ressenti le besoin de dissimuler aux autres votre maladie de Parkinson?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

## 24. Avez-vous évité des situations où vous deviez manger ou boire en public ? $\circ$ Jamais (0) o Rarement (1) o Parfois (2) o Souvent (3) o Toujours, ou ne peut jamais faire (4) 25. Vous êtes-vous senti(e) gêné(e) en public à cause de votre maladie de Parkinson ? $\circ$ Jamais (0) o Rarement (1)

- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 26. Vous êtes vous-senti(e) inquiet(e) des réactions des autres à votre égard ?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 27. Avez-vous eu des problèmes dans vos relations avec vos proches?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 28. Avez-vous manqué du soutien dont vous aviez besoin, de la part de votre époux(se) ou conjoint(e)?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 29. Avez-vous manqué du soutien dont vous aviez besoin, de la part de votre famille ou de vos ami(e)s proches?

- o Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 30. Vous êtes-vous endormi(e) dans la journée d'une façon inattendue ?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

# 31. Avez-vous eu des problèmes de concentration, par exemple en lisant ou en regardant la télévision ?

- o Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 32. Avez-vous senti que votre mémoire était mauvaise?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 33. Avez-vous fait de mauvais rêves ou eu des hallucinations?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- O Toujours, ou ne peut jamais faire (4)

### 34. Avez-vous des difficultés pour parler?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 35. Vous êtes-vous senti(e) incapable de communiquer normalement avec les autres ?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 36. Vous êtes-vous senti(e) ignoré(e) par les autres ?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

#### 37. Avez-vous eu des crampes ou spasmes musculaires douloureux ?

- o Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

#### 38. Avez-vous eu mal ou avez-vous eu des douleurs dans les articulations ou dans le corps?

- o Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- O Toujours, ou ne peut jamais faire (4)

## 39. Avez-vous eu la sensation désagréable de chaud ou de froid ?

- o Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 14.10 Appendix J – Parkinson disease questionnaire 8

A compléter à Visite 1, Visite 2, Visite 1.2 et Visite 2.2 si applicable.

Au cours de la dernière semaine,

#### 1. Avez-vous eu des problèmes à vous déplacer dans les lieux publics ?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 2. Avez-vous eu des difficultés pour vous habiller ?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

#### 3. Vous êtes-vous senti(e) déprimé(e) ?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 4. Vous êtes-vous senti(e) gêné(e) en public à cause de votre maladie de Parkinson ?

- o Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

#### 5. Avez-vous eu des problèmes dans vos relations avec vos proches?

- o Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

# 6. Avez-vous eu des problèmes de concentration, par exemple en lisant ou en regardant la télévision ?

- $\circ$  Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 7. Vous êtes-vous senti(e) incapable de communiquer normalement avec les autres ?

- o Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

## 8. Avez-vous eu des crampes ou spasmes musculaires douloureux ?

- o Jamais (0)
- o Rarement (1)
- o Parfois (2)
- o Souvent (3)
- o Toujours, ou ne peut jamais faire (4)

### 14.11 Appendix K – MOCA

A compléter lors du screening.



### 14.12 Appendix L – MiniBEST

A compléter à Baseline, Visite 3 et Visite 4.



Horak FB, Wrisley DM & Frank J (2009), The Balance Evaluation Systems Test (BESTest) to differentiate balance deficits. Phys Ther 89, 484-98. Oregon Health & Science University http://www.bestest.us/kes\_copies

| | Version franiaise du Mini Balance Evaluation Systems Test (Mini-BESTest')<br>Jean-François Lemay phit, PhD Audrey Roy pht, MSc Dany H. Gagnon pht, PhD | Patient ID:<br>Date: | RE-<br>Visite Baseline / Visite 3 | CONN<br>/ Visit | |
|---|---|---|---|---|---|
| | 7. DEBOUT (PIEDS JOINTS): YEUX OUVERTS, SURFACE FERME | | | | |
| Ш | Placez les mains sur les hanches. Placez vos pieds ensembles jusqu'à ce qu'ils soient | Temps en | Normal : 30 secondes. | 2 | |
| ᆸ | presque en contact. Regardez droit devant. | secondes : | Modéré : < 30 secondes. | 1 | 1 1 |
| ~ | Demeurez aussi stable et immobile que possible, jusqu'à ce que je vous dise d'arrêter. | | Sévère : Incapable. | 0 | 1 1 |
| S | 8. DEBOUT (PIEDS JOINTS): YEUX FERMÉS, SURFACE EN MOUSSE | | | | |
| | Montez sur la surface en mousse. Placez les mains sur les hanches. Placez vos pieds ensembles | Temps en | Normal: 30 secondes. | 2 | |
| S | jusqu'à ce qu'ils soient presque en contact. Demeurez aussi stable et immobile que possible, jusqu'à ce que je vous dise d'arrêter. Je vais commencer à chronométrer quand vous allez fermer les yeux. | secondes : | Modéré : < 30 secondes. | 1 | 1 1 |
| 6 | ce que je vous dise d'arreter. Je vais commencer à chronometrer quand vous allez termer les yeux. | | Sévère : Incapable. | 0 | 1 |
| Ē | 9. PLAN INCLINÉ- YEUX FERMÉS | | | | |
| ORIENTATION SENSORIELL | Montez sur le plan incliné, les orteils pointant vers le haut de la pente. Placez vos pieds à la largeur des épaules, les bras le long du corps. | Temps en secondes : | Normal : Se tient debout de façon indépendante durant 30 secondes et s'aligne avec la gravité. | 2 | |
| ₹ | Je vais commencer à chronométrer quand vous allez fermer les yeux. | | Modéré : Se tient debout de façon indépendante < 30 secondes OU s'aligne avec la surface. | 1 | 1 |
| 0 | | | Sévère : Incapable. | 0 | 1 1 |
| | | | TOTAL ORIENTATION SENSORIE | ELLE | /6 |
| | 10. CHANGEMENT DE VITESSE DE MARCHE | | | | |
| | Commencez à marcher à votre vitesse normale. Quand je dirai "vite", marchez le plus vite possible.<br>Quand je dirai "lent", marchez très lentement. | | significativement de vitesse de marche sans déséquilibre. | 2 | |
| | Quanti je dirar tent , marchez trestentement. | | ble de changer de vitesse de marche ou signes de déséquilibre. | 1 | |
| | | Sévère : Incapat | ole de changer significativement de vitesse de marche ET signes de déséquilibre. | 0 | |
| | 11. MARCHER EN TOURNANT LA TÊTE – À L'HORIZONTALE | 1 | la tête sans changer la vitesse de marche et en gardant un bon équilibre. | | |
| | Commencez à marcher à votre vitesse normale. Quand je dirai "droite", tournez la tête<br>pour regarder à droite. Quand je dirai "gauche", tournez la tête pour regarder à gauche. | | 2 | | |
| | Essayez de marcher en ligne droite. | | la vitesse de marche en tournant la tête. | 1 | |
| Щ | | Sévère : Présenc | e de déséquilibres en tournant la tête. | 0 | |
| DYNAMIQUE | 12. MARCHER ET PIVOTER | | | | |
| ₹ | Commencez à marcher à votre vitesse normale. Quand je dirai "tournez et arrêtez", faites demi-tour aussi vite que possible et arrêtez. Après le demi-tour. | | avec les pieds rapprochés RAPIDEMENT (≤ 3 pas) et avec un bon équilibre. | 2 | |
| Ž | vos pieds devraient être rapprochés." | | avec les pieds rapprochés LENTEMENT (≥ 4 pas) et avec un bon équilibre. | 1 | |
| | 42 ENLANDED UN ODETACLE | Sévère : Ne peut | tourner avec les pieds rapprochés sans déséquilibre, peu importe la vitesse. | 0 | |
| MARCHE | 13. ENJAMBER UN OBSTACLE | N 1.0 | | | |
| 호 | Commencez à marcher à votre vitesse normale. Quand vous arriverez à la boîte, passez par-dessus,<br>et non autour, et continuez à marcher. | | njamber la boîte en changeant minimalement sa vitesse de marche avec un bon équilibre. | 2 | |
| ¥ | | | e la boîte mais lui touche OU démontre un comportement prudent en ralentissant sa marche. | 0 | |
| Σ | 44 TIMED UP 9 CO AVEC DOUBLE TÂCHE ( | Severe : Incapab | le d'enjamber boîte OU contourne la boîte. | U | |
| | 14. TIMED UP & GO AVEC DOUBLE TÂCHE (marche sur 3 mètres) TUG: Quand je dirai "go", levez-vous de la chaise, marchez à votre vitesse normale, franchissez la | TUG: | TUG avec une double tâche : | | |
| | marque au sol, puis faites demi-tour et revenez vous asseoir sur la chaise. | | changement notable en position assise, debout ou en marchant lorsque le sujet compte à | (temps e | en secondes) |
| | TUG AVEC DOUBLE TÂCHE: "Comptez à rebours à voix haute par bonds de 3 à partir de :<br>Quand je dirai "go" levez-vous de la chaise, marchez à votre vitesse normale, franchissez la marque | | nparaison avec le TUG sans double tâche. | | |
| | au sol, puis faites demi-tour et revenez vous asseoir sur la chaise. Continuez à compter à rebours<br>pendant tout ce temps." Pour attribuer un score à l'épreuve 14, si la vitesse de marche du sujet ralentit | | | | |
| | de plus de 10% entre le TUG sans et avec la double tâche, le score devrait être diminué d'un point. | Sévère : Arrête d | de compter en marchant OU arrête de marcher en comptant. | 0 | |
| | | | TOTAL MARCHE DYNAMI | QUE | /10 |

<sup>&#</sup>x27;Horak FB, Wrisley DM & Frank J (2009), The Balance Evaluation Systems Test (BESTest) to differentiate balance deficits. Phys Ther 89, 484-98. Oregon Health & Science University http://www.bestest.us/test\_copies

RE-CONNECT

Version franiaise du Mini Balance Evaluation Systems Test (Mini-BESTest') Jean-François Lemay pht, PhD | Audrey Roy pht, MSc | Dany H. Gagnon pht, PhD

Patient ID: Visite Baseline / Visite 3 / Visit 4 Date:

#### Directives pour le Mini-BESTest

Directives pour le Mini-BES lest
Préparation du sujet : Le sujet devrait être évalué avec des souliers à talons plats OU sans souliers ni chaussette.
Équipement: Une surface en mousse Temper® (aussi appelé T-foamT)l de 10cm (4") d'épaisseur, de densité moyenne T41), une chaise sans accoudoir ni roulette, un plan incliné (10", au moins 60x60 cm (2"x2")), un chronomètre, une boite (23 cm (9") de haut) et une distance de 3 mètres mesurée à partir de la chaise et indiquée au plancher par des marques.
Attribution des soores : Le soore maximal pour ce test est de 28 points. Chacune des 61 4é preuves est notée de 0 à 2.
"0" représente le plus bas niveau fonctionnel et "2" le plus haut niveau fonctionnel.
Si un sujet oit utilister une adde technique pour une épreuve, diminuez le soore d'une catégorie.
Si un sujet oit utilister une adde technique pour une épreuve, diminuez le soore d'une catégorie.
Pour l'épreuve 3 (5 tenirs ur une jambe) et l'épreuve (5 (Stratégie de pas compensatoire: LATÉRAL), utilisez le soore d'un seul côté (le moins bon).
Pour l'èpreuve 3 (5 tenirs ur une jambe), sélectionnez le meilleur temps des deux essais (pour un côté donné) pour attribuer le soore de ce côté.
Pour l'èpreuve 14 (Timed up 8 go avec double tâche), si la vitesse de marche du sujet ralentit de plus de 10% entre le TUG sans et avec la double tâche, le score devrait être diminué d'un point.

| 1. ASSIS À DEBOUT | Observez l'initiation du mouvement ainsi que le recours aux mains sur le siège ou sur les cuisses de même que la projection des bras vers l'avant. |
|---|---|
| 2. MONTER SUR LA<br>POINTEDES PIEDS | Accordez deux essais au sujet. Attribuez un score au meilleur essai. (Si vous soupçonnez que le sujet ne monte pas à la hauteur maximale, demandez-lui de remonter en tenant les mains de l'évaluateur). Assurez-vous que le sujet regarde une cible fixe située devant lui à une distance de 1,25 à 3,7 m (4 à 12°). |
| 3. SE TENIR SUR UNE<br>JAMBE | Accordez deux essais au sujet et notez le temps en seconde que le sujet peut tenír jusqu'à un maximum de 20 secondes. Arrêtez de chronométrer si le sujet enlève les mains de ses hanches ou qu'il pose son pried au sol. Assurez-vous que le sujet regarde une cible fixe située devant lui à une distance de 1,25 à 3,7 m (4 à 12'). Répétez pour l'autre côté. |
| 4. STRATÉGIE DE<br>PAS<br>COMPENSATOIRE:<br>ANTÉRIEUR | Tenez-vous devant le sujet avec une main sur chacune de ses épaules. Demandez-lui de se pencher vers l'avant (assurez-vous qu'il y a assez d'espace pour qu'il puisse faire un pas vers l'avant). Demandez au sujet de se pencher jusqu'à ce que ses épaules et ses hanches soient devant ses orteils. Lorsque vous sentez que le poids du sujet repose dans vos mains, retirez très subitement votre support. Le test doit provoquer un pas. REMARQUE: Soyez prêt à attraper le sujet en cas d'une perte d'équilibre. |
| 5. STRATÉGIE DE<br>PAS<br>COMPENSATOIRE:<br>POSTÉRIEUR | Tenez-vous derrière le sujet avec une main sur chacune de ses omoplates. Demandez-lui de se pencher vers l'arrière. (Assurez-vous qu'il y a assez d'espace pour qu'il puisse faire un pas vers l'arrière). Demandez au sujet de se pencher jusqu'à ce que ses épaules et ses hanches soient derrière ses taions. Lorsque vous sentez que le poids du sujet repose dans vos mains, retirez très subitement votre support. Le test doit provoquer un pas. REMARQUE: Soyez prêt à attraper le sujet en cas d'une perte d'équilibre. |
| 6. STRATÉGIE DE PAS<br>COMPENSATOIRE:<br>LATÉRAL | Tenez-vous à côté du sujet et placez une main sur le côté du bassin. Demandez-lui d'appuyer tout son corps dans votre main. Demandez au sujet de se pencher jusqu'à ce que le centre de son bassin soit au-dessus du pied droit (ou gauche) puis retirez subitement votre support. REMARQUE: Soyez prêt à attraper le sujet en cas d'une perte d'équilibre. |
| 7. DEBOUT (PIEDS<br>JOINTS): YEUX OUVERTS,<br>SURFACE FERME | Notez le temps que le sujet peut tenir debout pieds joints jusqu'à un maximum de 30 secondes. Assurez-vous que le sujet regarde une cible fixe située devant lui à une distance de 1,25 à 3,7 m (4 à 12'). |
| 8. DEBOUT (PIEDS<br>JOINTS): YEUX FERMÉS,<br>SURFACE ENMOUSSE | Utilisez une surface en mousse de densité moyenne Temper® de 10 cm (4") d'épaisseur. Aidez le sujet à monter sur le coussin. Notez le temps que le sujet peut tenir débout jusqu'à un maximum de 30 secondes. Demandez au sujet de descendre du coussin entre les essais. Retournez le coussin entre chaque essai pour s'assurer qu'il ait conservé sa forme. |
| 9. PLAN INCLINÉ-<br>YEUXFERMÉS | Aidez le sujet à monter sur le plan incliné. Commencez à chronométrer une fois les yeux du sujet fermés et notez le temps. Notez la présence d'oscillations posturales excessives. |
| 10. CHANGEMENT<br>DEVITESSE DE<br>MARCHE | Laissez le sujet faire de 3 à 5 pas à vitesse normale, puis dites : "vite". Après 3 à 5 pas rapides, dites : "lent". Laissez le sujet faire 3 à 5 pas lents avant qu'il arrête de marcher. |
| 11. MARCHER EN<br>TOURNANTLA TÊTE – À<br>L'HORIZONTALE | Laissez le sujet atteindre sa vitesse normale puis dites "droite, gauche" à tous les 3 à 5 pas. Notez si vous voyez un problème dans l'une ou l'autre des directions.<br>Si le sujet a des restrictions cervicales sevères, permettez un mouvement combiné de la tête et du tronc |
| 12. MARCHER ET PIVOTER | Faites la démonstration du pivot. Une fois que le sujet marche à vitesse normale, dites "tournez et arrêtez". Comptez le nombre de pas à partir de la commande "tournez" jusqu'à ce que le sujet soit stable. Les déséquilibres peuvent se manifester par une position élargie des pieds, des pas supplémentaires ou des mouvements du tronc. |
| 13. ENJAMBER UN<br>OBSTACLE | Placez une boîte (23 cm (9") de haut) à 3 m (10') de l'endroit où le sujet commencera à marcher. Deux boîtes de souliers superposées peuvent être utilisées pour confectionner cet équipement. |

Horak FB, Wrisley DM & Frank J (2009), The Balance Evaluation Systems Test (BESTest) to differentiate balance deficits. Phys Ther 89, 484-98. Oregon Health & Science University http://www.bestest.us/test\_copies

Version franiaise du Mini Balance Evaluation Systems Test (Mini-BESTest') Jean-François Lemay pht, PhD | Audrey Roy pht, MSc | Dany H. Gagnon pht, PhD

Patient ID: Date:

RE-CONNECT Visite Baseline / Visite 3 / Visit 4

14. TIMED UP & GO AVECDOUBLE TÂCHE

Utilisez le temps du TUG pour déterminer les effets de la double tâche. Le sujet devrait parcourir une distance de 3 mètres. others e temps ou to pool uctermine reservets our a double talors. Es sujet cert and particul if un expected of since the Since test in the Since the Since test is a common to the Since test in the Since test is a common test of the Since test in the Since test is a common test of the Since test is a since test in the Since test in the Since test is a since test in the Since test in the signes de déséquilibre.

### 14.13 Appendix M – MDS-UPDRS

A compléter à Baseline, Visite 3 et Visite 4.

### MDS UPDRS I-IV

Source principale d'information :

- patient
- □ aidant
- patient et aidant en proportion égale

Partie I : expérience non motrice de la vie quotidienne

#### 1.1 Altération cognitive

Prendre en compte tous types de niveau d'altération des fonctions cognitives, y compris le ralentissement cognitif, l'altération du raisonnement, la perte de mémoire, les déficits de l'attention et de l'orientation. Evaluer leur impact sur les activités de la vie quotidienne telles qu'elles sont perçues par le patient et/ou l'aidant.

(au cours de la semaine précédente, avez-vous eu des problèmes pour vous rappeler des choses ; pour suivre des conversations, pour fixer votre attention, pour avoir des pensées claires ou pour trouver votre chemin dans la maison ? si oui, l'examinateur demande au patient ou à l'aidant de donner des détails et des approfondissements pour information)

0 = normal : pas d'altération cognitive

1 = minime : altération appréciée par le patient ou l'aidant sans interférence concrète avec

l'aptitude du patient à mener des activités et des interactions sociales

2 = léger : dysfonctionnement cognitif cliniquement évident, mais avec seulement des

interférences minimes avec l'aptitude du patient à mener des activités et des

interactions sociales normales.

3 = modéré : les déficits cognitifs interfèrent mais n'empêchent pas l'aptitude du patient à mener des

activités et des interactions sociales normales.

4 = sévère : le dysfonctionnement cognitif empêche l'aptitude du patient à mener des activités et

des interactions sociales normales.

### 1.2 Hallucinations et psychose

Considérer à la fois les illusions (interprétations erronées de stimuli réels) et les hallucinations (fausses sensations spontanées). Considérez tous les principaux domaines sensoriels (visuel, auditif, olfactif, gustatif). Déterminez la présence de sensations non formées, aussi bien que des sensations formées. Evaluez la capacité du patient à critiquer ses hallucinations et identifiez l'existence d'illusions et des pensées psychotiques.

(au cours de la semaine précédente, avez-vous vu, entendu, senti ou ressenti des choses qui n'existaient pas réellement)

0 = normal : pas d'hallucinations, ni de comportement psychotique

1 = minime : illusions ou hallucinations non formées, mais le patient les reconnaît et les critique
 2 = léger : hallucinations structurées indépendantes des stimuli environnementaux, pas de perte

de sens critique à leur égard

3 = modéré : hallucinations structurées non critiquées par le patient 4 = sévère : le patient a des idées délirantes ou paranoïaques

#### 1.3 Humeur dépressive

Considérez la baisse de l'humeur, la tristesse, la désespérance, les sentiments de vide ou la perte de plaisir. Déterminez leur présence et leur durée pendant la période de la semaine précédente et évaluez leur interférence avec l'aptitude du malade à mener sa routine quotidienne et à participer à des interactions sociales.

(au cours de la semaine précédente, vous êtes-vous sentie sans ressort, triste, désespéré(e) ou incapable d'apprécier les choses ? si oui ce sentiment durait-il plus d'un jour à la fois ?rendait-il difficile pour vous le fait de mener vos activités et d'être avec les autres ?)

pas d'humeur dépressive normal

minime épisodes d'humeur dépressive ne durant pas plus d'un jour à la fois. Pas

d'interférence avec l'aptitude du patient à mener des activités et des interactions

humeur dépressive durant plusieurs jours, mais sans interférence avec des activités et léger

des interactions sociales normales

modéré humeur dépressive interférant avec l'aptitude du patient à mener des activités et

des interactions sociales normales

sévère humeur dépressive empêchant l'aptitude du patient à mener des activités et

des interactions sociales normales

#### 1.4 Etat anxieux

Déterminez les sensations de nervosité, de tension, d'inquiétude ou d'anxiété (incluant les attaques de panique) au cours de la semaine précédente et évaluez leur durée et les interférences avec l'aptitude du patient à mener des activités journalières et à participer à des interactions sociales.

(au cours de la semaine précédente, vous êtes-vous senti(e), nerveux, inquiet(e), tendu(e) ? si oui, ce sentiment durait- il plus d'1 jour à la fois. Est-ce que cela a constitué pour vous une difficulté pour suivre vos activités habituelles ou peut-être avec d'autres personnes)

pas de sentiment d'anxiété

sentiments anxieux présents, mais ne durant pas plus d'un jour à la fois. Pas minime

d'interférence avec l'aptitude du patient à mener des activités et des interactions

sociales normales.

léger sentiments anxieux persistant plus d'un jour à la fois, mais sans interférence

avec l'aptitude du patient à mener des activités et des interactions sociales

sentiments anxieux interférant avec, mais n'empêchant pas l'aptitude du patient à modéré

mener des activités et des interactions sociales normales

sévère sentiments anxieux empêchant l'aptitude du patient à mener des activités et

des interactions sociales normales

#### 1.5 Apathie

Déterminez le niveau d'activité spontanée, d'assurance, de motivation et d'initiative, et évaluez l'impact d'une réduction de performance sur les activités quotidiennes routinières et les interactions sociales

(au cours de la semaine précédente, vous êtes-vous senti(e) indifférent à faire des activités ou à être avec des gens ?)

normal pas d'apathie

l'apathie est percue par le patient et/ou aidant, mais sans interférence avec les activités minime

quotidiennes ni les interactions sociales

l'apathie interfère avec des activités et des interactions sociales isolées = léger 3 modéré l'apathie interfère avec la plupart des activités et des interactions sociales

sévère attitude passive et retirée, avec perte totale d'initiative

#### 1.6 Signes de syndrome de dysrégulation dopaminergique

Déterminez la participation du malade à diverses activités par ex une passion atypique ou excessive du jeu, des pulsions ou des intérêts sexuels atypiques ou excessifs, ainsi qu'à d'autres activités répétitives, ou à la prise des médicaments non prescrits sans raison clinique. Evaluez l'impact de telles activités ou comportements anormaux sur la vie personnelle du patient et sur celle de sa famille et de ses relations sociales (emprunter de l'argent, conflits familiaux majeurs, perte d'une partie du temps de travail, sauter des repas ou manquer de sommeil en raison de ces activités.

(au cours de la semaine précédente, avez-vous ressenti(e) des fortes pulsions inhabituelles que vous avez eues du mal à contrôler ? vous êtes-vous poussé(e)) faire ou penser des choses et éprouvez-vous de la difficulté à les arrêter ?)

0 = normal ; pas de problème présent

= minime : des problèmes existent mais n'entraînent habituellement pas de difficulté pour le patient

ou la famille/l'aidant

2 = léger : des problèmes existent et entraînent habituellement quelques difficultés dans la

vie personnelle du patient et sa vie de famille

3 = modéré : des problèmes existent et entraînent habituellement beaucoup de difficultés dans la

vie personnelle du patient et sa vie de famille

4 = sévère : des problèmes existent et empêchent l'aptitude du patient à mener des activités et

de interactions sociales normales, ou de maintenir les standards antérieurs de sa

vie personnelle et familiale

#### 1.7 Problèmes de sommeil

Au cours de la semaine précédente, avez-vous rencontré des problèmes pour vous endormir la nuit ou pour rester endormi pendant la nuit ?prenez en compte la façon dont vous vous êtes senti(e)reposé(e) après vous être réveillé(e) le matin

0 = normal ; pas de problème

1 = minime : des problèmes de sommeil sont présents mais n'entraînent pas habituellement

de difficultés à avoir une nuit complète de sommeil

2 = léger : des problèmes de sommeil entraînent habituellement quelques difficultés à avoir une nuit

complète de sommeil

3 = modéré : des problèmes de sommeil entraînent beaucoup de difficultés à avoir une nuit

complète de sommeil, mais je dors encore habituellement plus de la moitié de la nuit

4 = sévère : je ne dors habituellement pas la plus grande partie de la nuit

#### 1.8 Somnolence diurne

Au cours de la semaine précédente, avez-vous rencontré des problèmes pour rester éveillé(e)pendant la journée ?

0 = normal : pas de somnolence diurne

1 = minime : une somnolence diume apparaît mais je peux résister et rester éveillé(e)

2 = léger : je m'endors parfois quand je suis seul et au repos. Par exemple, pendant que je lis ou

en regardant la télévision

3 = modéré : je m'endors parfois alors que je ne devrais pas. Par exemple, en mangeant ou en parlant

à d'autres personnes

4 = sévère : je m'endors souvent alors que je ne devrais pas. Par exemple, en mangeant ou

en parlant à d'autres personnes

#### 1.9 Douleurs et autres sensations

Au cours de la semaine précédente, avez-vous eu des sensations inconfortables dans votre corps telles que douleur, courbatures, fourmillements ou crampes ?

0 = normal ; pas de sensations inconfortables

1 = minime : je ressens ces sensations. Cependant, je peux faire les choses et être avec

d'autres personnes sans difficulté

2 = léger : ces sensations me procurent quelques problèmes quand je fais des choses et quand je

suis avec d'autres personnes

3 = modéré : ces sensations me procurent beaucoup de problèmes, mais ne m'empêchent

pas d'effectuer des choses ou d'être avec d'autres personnes

4 = sévère : ces sensations m'empêchent de faire des choses et d'être avec d'autres

#### 1.10 Problèmes urinaires

Au cours de la semaine précédente, avez-vous eu des difficultés à contrôler vos urines ? par exemple, besoin urgent d'uriner, besoin d'uriner trop souvent ou accidents urinaires

0 = normal ; pas de problème urinaire

1 = minime : j'ai besoin d'uriner souvent ou urgemment. Cependant, ces problèmes ne causent pas

de difficultés dans mes activités quotidiennes

2 = Jéger : les problèmes urinaires causent quelques difficultés dans mes activités quotidiennes.

Cependant je n'ai pas d'accidents urinaires

3 = modéré : les problèmes urinaires causent beaucoup de difficultés dans ma vie

quotidienne, incluant des accidents urinaires

4 = sévère : je ne peux pas contrôler mes urines, et utilise une garniture de protection ou une

sonde urinaire

#### 1.11 Problèmes de constipation

Au cours de la semaine précédente, avez-vous eu des problèmes de constipation entraînant des difficultés à aller la selle ?

0 = normal ; pas de constipation

1 = minime : j'ai été constipé(e). Je fais des efforts supplémentaires pour aller à la selle. Cependant

ce problème ne perturbe pas mes activités ou mon confort

2 = léger : la constipation me pose quelques difficultés à faire des choses ou à me sentir confortable

3 = modéré : la constipation me pose beaucoup de problème à faire les choses ou à me

sentir confortable. Cependant, elle ne m'empêche pas de faire quoi que ce soit

4 = sévère : j'ai habituellement besoin de l'aide physique d'un tiers pour aller à la selle

### 1.12 Sensation de tête vide au lever

Au cours de la semaine précédente, avez-vous eu une sensation d'évanouissement, de vertige, de brouillard lorsque vous vous levez d'une position assise ou couchée ?

0 = normal : pas de sensation de vertige ou de brouillard

1 = minime : des sensations de vertige ou de brouillard surviennent. Cependant elles ne me

causent pas de problèmes à faire les choses

2 = léger : des sensations de vertige ou de brouillard m'obligent à me tenir à quelque chose, mais

je n'ai pas besoin de m'asseoir ou de me recoucher

3 = modéré : des sensations de vertige ou de brouillard m'obligent à m'asseoir ou à me coucher

pour éviter de m'évanouir ou de tomber

4 = sévère : des sensations de vertige ou de brouillard me conduisent à tomber ou à m'évanouir

### 1.13 Fatigue

Au cours de la semaine précédente, vous êtes-vous senti(e) habituellement fatigué(e) ? ce sentiment ne fait pas partie du fait d'avoir sommeil ou d'être triste

0 = normal 1 = minime

: pas de fatigue : la fatigue la fatigue se présente. Cependant, elle ne me cause pas de problème à faire les choses

ou à être avec les gens

2 = léger la fatigue me cause quelques problèmes à faire les choses ou à être avec les gens 3 = modéré la fatigue me cause beaucoup de problèmes à faire les choses ou être avec les

gens. Cependant, elle ne m'empêche pas à faire quoi que ce soit 4 = sévère la fatigue m'empêche de faire des choses ou d'être avec des gens

repos

#### Partie III: examen moteur en ON

| | | ∟e patient<br>inson ? | reçoit- | il des médicaments pour traiter les symptômes de la maladie de |
|---|---|---|---|---|
| | 0 | UI | | |
| | ) N | ON | | |
| | | | | it des médications pour traiter les symptômes de la maladie de<br>at clinique du patient en utilisant les définitions suivantes : |
| | | N. ON corr<br>nt une bonr | | d à l'état fonctionnel type quand les patients reçoivent leur(s) médication(s) et<br>onse. |
| | | | | nd à l'état fonctionnel type quand les patients ont une mauvaise réponse<br>prennent des médications. |
| 3 | ic : L | e patient | est-il s | ous lévodopa ? |
| | 0 | UI : | 3.C1 S | i oui, minutes écoulées depuis la dernière dose de lévodopa : |
| | ) No | ON | | |
| 3 | 3.1 | Parole | | ON _ |
| 0<br>1<br>2<br>3 | mme<br>arté,<br>nt les | ent il s'est<br>incluant l'a<br>s syllabes e<br>normal<br>minime<br>léger<br>modéré<br>sévère | rendu :<br>rticulat<br>ensemb<br>:<br>: | pas de problème de parole perte de modulation, de diction ou de volume, mais tous les mots sont encore faciles à comprendre. perte de modulation, de diction ou de volume avec quelques mots peu clairs mais la majorité des phrases sont faciles à suivre. le discours est difficile à comprendre à tel point que quelques phrases, mais pas la plupa sont mal comprises. la plupart du discours est difficile à comprendre ou inintelligible. |
| 3 | 3.2 | Expressi | ion fac | ciale ON _ |
| pa<br>fac<br>0<br>1 | rle. (<br>ciale, | Observez la<br>, le sourire<br>normal<br>minime | a fréqu | s, au repos pendant 10 secondes, sans qu'il parle et aussi pendant qu'il ence du clignement de l'œil, faciès en masque ou la perte d'expression iné et l'intervalle entre les lèvres. expression faciale normale. faciès en masque minime, seulement manifestés par une diminution de la fréquence du clignement des paupières. en plus de la diminution de la fréquence du clignement, le faciès en masque est présent dans la partie inférieure du visage, à savoir rareté des mouvements autour de la bouche, tel qu'un amoindrissement du sourire spontané, mais les lèvres ne sont pas |
| 3 | = | modéré | : | séparées.<br>faciès en masque avec quelquefois les lèvres séparées quand la bouche est au repos. |
| 4 | = | sévère | : | faciès en masque avec lèvres séparées la plupart du temps quand la bouche est au |

| INITIALES PATIENT : _ / _ N | I° D'INCLUSION : _ _ |
|-----------------------------------|--------------------------|
|-----------------------------------|--------------------------|

#### 3.3 Rigidité

La rigidité est jugée sur des mouvements lents et passifs des principales articulations, quand le patient est en position relâchée et que l'investigateur lui manipule les membres et le cou. En premier, testez sans manœuvre d'activation. Testez et évaluez le cou et chaque membre séparément. Pour les bras, testez les articulations du poignet et du coude simultanément. Pour les jambes, testez les articulations de la hanche et du genou simultanément. Si aucune rigidité n'est détectée, utilisez une manœuvre d'activation (de sensibilisation) tel que tapotement des doigts, ouverture et fermeture du poing, ou taper du talon, sur un membre n'étant pas testé. Expliquez au patient d'être aussi relâché que possible puisque vous testez la rigidité.

| | | | | | ON |
|---|---|---|---|---|---|
| 0 | = | normal | : | pas de rigidité. | cou _ |
| 1 | = | minime | : | rigidité seulement détectée avec la manœuvre d'activation. | |
| 2 | = | léger | : | rigidité détectée sans manœuvre d'activation, mais | MSD _ |
| | | | | l'amplitude complète de mobilisation est facilement<br>effectuée. | MSG _ |
| 3 | = | modéré | : | rigidité détectée sans manœuvre d'activation ; l'amplitude complète de mobilisation est effectuée avec effort. | |
| 4 | = | sévère | : | rigidité détectée sans manœuvre d'activation et l'amplitude complète | MID _ |
| | | | | de mobilisation n'est pas réalisée. | MIG I I |

#### 3.4 Tapotement de doigt

Chaque main est testée séparément. Faites la démonstration de la tâche, mais ne continuez pas à effectuer la tâche pendant que le patient est testé. Donnez au patient l'instruction de tapoter l'index sur le pouce 10 fois aussi rapidement et amplement que possible. Evaluer chaque côté séparément en évaluant la vitesse, l'amplitude, les hésitations, les haltes et la diminution de l'amplitude.

| 0 | = | normal | aucun problème. | |
|---|---|---|---|---|
| 1 | = | minime | n'importe laquelle des situations suivantes : a) le rythme régulier Of est cassé par une ou deux interruptions ou hésitations du | N |
| | | | mouvement de tapotement ; b) raientissement minime ; c) MD l'amplitude diminue près de la fin des 10 tapotements. | _ |
| 2 | = | léger | n'importe laquelle des situations suivantes : a) 3 à 5 interruptions pendant le tapotement ; b) léger ralentissement ; c) l'amplitude diminue à la moitié de la séquence des 10 tapotements. | _ |
| 3 | = | modéré | n'importe laquelle des situations suivantes : a) plus de 5 interruptions pendant le tapotement ou au moins un arrêt prolongé dans le mouvement en cours ; b) ralentissement modéré ; c) l'amplitude diminue commençant dès le premier tapotement. | |
| 4 | = | sévère | ne peut pas ou peut seulement à peine effectuer la tâche à cause du ralentissement, des interruptions ou des diminutions d'amplitude. | |

#### 3.5 Mouvements de la main

Testez chaque main séparément. Faites la démonstration de la tâche mais ne continuez pas à effectuer la tâche pendant que le patient est testé. Donnez au patient l'instruction de fermer le poing, coude plié, de telle sorte que la paume soit face à l'investigateur. Demandez au patient d'ouvrir la main 10 fois aussi amplement et aussi rapidement que possible. Si le patient ne réussit pas à avoir le poing serré ou à ouvrir la main en grand, rappelez-lui de le faire. Evaluez chaque côté séparément, en évaluant la vitesse, l'amplitude, les hésitations, les haltes et la diminution de l'amplitude.

| | | | | ON |
|---|---|---|---|---|
| 1 | = | normal<br>minime | aucun problème. n'importe laquelle des situations suivantes : a) le rythme régulier est cassé par une ou deux interruptions ou hésitations du mouvement ; b) ralentissement minime ; c) l'amplitude diminue près de la fin de la tâche. | MD _ |
| 2 | = | léger | n'importe laquelle des situations suivantes : a) 3 à 5 interruptions<br>pendant les mouvements ; b) léger ralentissement ; c) l'amplitude<br>diminue à la moitié de la tâche. | MG _ |
| 3 | = | modéré | n'importe laquelle des situations suivantes : a) plus de 5 interruptions<br>pendant le mouvement ou au moins un arrêt prolongé (blocage) dans le<br>mouvement en cours ; b) ralentissement modéré ; c) l'amplitude diminue<br>dès la première séquence d'ouverture et de fermeture. | |
| 4 | = | sévère | ne peut pas ou peut seulement à peine effectuer la tâche à cause<br>du ralentissement, des interruptions ou des diminutions | |

### 3.6 Mouvements pronation et supination des mains

Testez chaque main séparément. Faites la démonstration de la tâche, mais ne continuez pas à effectuer la tâche pendant que le patient est testé. Donnez au patient l'instruction d'étendre le bras devant son corps, paume vers le bas, puis de tourner les paumes de haut en bas, alternativement 10 fois aussi rapidement et amplement que possible. Evaluez chaque côté séparément en évaluant la vitesse, l'amplitude, les hésitations, les haltes et la diminution de l'amplitude.

| 0 | = | normal | | aucun problème. | ON |
|---|---|---|---|---|---|
| 1 | = | minime | | n'importe laquelle des situations suivantes : a) le rythme régulier est cassé par une ou deux interruptions ou hésitations du | MD _ |
| | | | | mouvement ; b) ralentissement minime ; c) l'amplitude diminue près de la fin de la séquence. | MG _ |
| 2 | = | léger | : | n'importe laquelle des situations suivantes : a) 3 à 5 interruptions<br>pendant les mouvements ; b) léger ralentissement ; c) l'amplitude<br>diminue à la moitié de la séquence. | |
| 3 | = | modéré | : | n'importe laquelle des situations suivantes : a) plus de 5 interruptions pendant le mouvement ou au moins un arrêt prolongé (blocage) dans le mouvement en cours ; b) ralentissement modéré ; c) l'amplitude diminue commençant dès la première séquence de prono- supination. | |
| 4 | = | sévère | : | ne peut pas ou peut seulement à peine effectuer la tâche à cause<br>du ralentissement, des interruptions ou des diminutions | |

ON

#### 3.7 Tapotement de l'orteil

Installez le patient assis dans un fauteuil à dossier droit et accoudoirs, les deux pieds au sol. Testez chaque pied séparément. Faites la démonstration de la tâche, mais ne continuez pas à effectuer la tâche pendant que le patient est testé. Donnez au patient, l'instruction de mettre le talon au sol dans une position confortable, puis de taper les orteils 10 fois aussi amplement et rapidement que possible. Evaluez chaque côté séparément en évaluant la vitesse, l'amplitude, les hésitations, les haltes et la diminution de l'amplitude.

normal 0 aucun problème. MD |\_| minime n'importe laquelle des situations suivantes : a) le rythme régulier est cassé par une ou deux interruptions ou hésitations du mouvement de tapotement ; b) ralentissement minime ; c) l'amplitude diminue près de la fin des 10 tapotements. n'importe laquelle des situations suivantes : a) 3 à 5 interruptions léger MG |\_| pendant les mouvements de tapotement ; b) léger ralentissement ; c) l'amplitude diminue à la moitié de la tâche. n'importe laquelle des situations suivantes : a) plus de 5 = modéré interruptions pendant les mouvements de tapotement ou au moins

interruptions pendant les mouvements de tapotement ou au moins un arrêt prolongé (blocage) dans le mouvement en cours ; b) ralentissement modéré ; c) l'amplitude diminue après le premier tapotement.

4 = sévère : ne peut pas ou peut seulement à peine effectuer la tâche à cause du ralentissement, des interruptions ou des diminutions d'amplitude.

#### 3.8 Agilité de la jambe

Installez le patient assis dans un fauteuil à dossier droit et accoudoirs. Le patient doit avoir les deux pieds confortablement au sol. Testez chaque jambe séparément. Faites la démonstration de la tâche, mais ne continuez pas à effectuer la tâche pendant que le patient est testé. Donnez au patient, l'instruction de mettre le pied au sol dans une position confortable et puis de lever et de taper le pied au sol 10 fois aussi haut et rapidement que possible. Evaluez chaque côté séparément en évaluant la vitesse, l'amplitude, les hésitations, les haltes et la diminution de l'amplitude.

ON : aucun problème. 0 normal minime n'importe laquelle des situations suivantes : a) le rythme régulier MD |\_| est cassé par une ou deux interruptions ou hésitations du mouvement. b) ralentissement minime; c) l'amplitude diminue vers la fin de la : n'importe laquelle des situations suivantes : a) 3 à 5 interruptions léger MG |\_ | pendant les mouvements ; b) léger ralentissement ; c) l'amplitude diminue à la moitié de la tâche. modéré : n'importe laquelle des situations suivantes : a) plus de 5 interruptions pendant le mouvement ou au moins un arrêt prolongé (blocage) dans le mouvement en cours ; b) ralentissement modéré de la vitesse ; c) l'amplitude diminue après le premier tapotement. sévère : ne peut pas ou peut seulement à peine effectuer la tâche à cause du ralentissement, des interruptions ou des diminutions d'amplitude.

Installez le patient assis dans un fauteuil à dossier droit et accoudoirs, les deux pieds au sol et bien enfoncé dans la chaise (si le patient n'est pas trop petit). Demandez au patient de croiser les bras sur la poitrine et puis de se lever. Si le patient ne réussit pas, répétez cet essai jusqu'à un maximum de 2 fois plus. S'il ne réussit toujours pas, autorisez le patient à s'avancer au bord de la chaise pour se lever les bras croisés sur la poitrine. Autorisez seulement un essai dans cette position. S'il ne réussit pas, autorisez le patient à se soulever en s'aidant de ses mains sur les accoudoirs de la chaise. Autorisez un maximum de 3 essais de poussées. S'il ne réussit toujours pas aidez le patient à se lever. Après que le patient soit debout, observez la posture pour l'item 3 13

0 = normal ; aucun problème ; capable de se lever rapidement sans hésitation.

= minime : le lever est plus lent que la normale ; ou peut avoir nécessité plus d'un essai ; ou peut

avoir besoin de s'avancer au bord du fauteuil pour se lever. Pas besoin d'utiliser les

accoudoirs du fauteuil.

2 = léger : se lève en s'aidant des accoudoirs du fauteuil sans difficulté.

3 = modéré : a besoin de s'aider pour se lever, mais a tendance à tomber en arrière ; ou peut devoir

essayer plus d'une fois en utilisant les accoudoirs du fauteuil, mais peut se lever sans

4 = sévère : incapable de se lever sans aide.

### 3.10 Marche ON |

On évalue la marche de la meilleure façon en faisant que le patient marche en s'éloignant et puis revienne vers l'investigateur de façon à ce que les deux côtés, droit et gauche du corps, puissent être facilement observés et simultanément. Le patient devra marcher au moins 10 m puis tourner et revenir vers l'investigateur. Cet item mesure des comportements multiples : l'amplitude de la foulée, la vitesse de la foulée, la hauteur à laquelle le pied est soulevé, la frappe du talon pendant la marche, la façon de pivoter, et le ballant des bras, mais non le blocage de la marche (freezing). Evaluez aussi pour « blocage de la marche » (freezing) (item suivant 3.11) pendant que le patient marche. Observez la posture pour l'item 3.13.

0 = normal ; aucun problème.

1 = minime : déambulation autonome avec altération minime de la marche.

2 = léger : déambulation autonome mais avec une altération substantielle de la marche.
3 = modéré : nécessite un dispositif d'assistance pour une marche sûre (canne, déambulateur).

mais pas d'aide humaine.

4 = sévère : ne peut pas marcher du tout ou seulement avec l'aide d'une autre personne.

#### 3.11 Blocage de la marche (freezing)

Pendant l'évaluation de la marche, évaluez aussi la présence d'épisodes de blocage de marche (freezing). Observez l'hésitation au démarrage et les mouvements de piétinements particulièrement au demi-tour et en atteignant la fin de la tâche. Dans la mesure autorisée par leur sécurité, les patients ne peuvent pas utiliser des astuces sensorielles pendant l'évaluation.

0 = normal ; pas de blocage.

1 = minime : se bloque au démarrage, au demi-tour ou en passant le seuil d'une porte avec un seul

arrêt durant n'importe lequel de ces événements, mais ensuite continue de façon unie

sans blocage pendant la marche en ligne droite.

2 = léger : se bloque au démarrage, au demi-tour ou en passant le seuil d'une porte avec plus d'un

seul arrêt durant n'importe laquelle de ces activités, mais continue de façon unie sans

blocage pendant la marche en ligne droite.

3 = modéré : se bloque une fois pendant la marche en ligne droite. 4 = sévère : se bloque plusieurs fois pendant la marche en ligne droite.

### 3.12 Stabilité posturale

ON |

Le test examine la réaction à un déplacement soudain du corps produit par une poussée rapide et énergique sur les épaules, tandis que le patient est debout, les yeux ouverts, les pieds confortablement séparés et parallèles. Test de rétropulsion. Tenez-vous derrière le patient et indiquez lui ce qu'il va se passer. Expliquez lui, qu'il ou elle, est autorisé(e) à faire un pas en arrière pour éviter de tomber. Il devrait y avoir un mur solide derrière l'examinateur, à au moins 1 ou 2 m de distance pour permettre l'observation du nombre de pas rétropulsifs. La première poussée est une démonstration instructionnelle et est intentionnellement plus légère et non évaluée. La deuxième fois, les épaules sont tirés brusquement et énergiquement vers l'investigateur avec assez de force pour déplacer le centre de gravité de telle sorte que le patient DOIT faire un pas en arrière. L'investigateur a besoin d'être près pour rattraper le patient mais doit se tenir suffisamment en arrière de façon à laisser assez de place pour que le patient puisse faire plusieurs pas et retrouver son équilibre. N'autorisez pas le patient à fléchir le corps anormalement en avant pour anticiper l'impact. Observez le nombre de pas vers l'arrière ou la chute. On considère le test comme normal tant que le malade ne fait pas plus de 2 pas (2 pas y compris) en arrière pour retrouver son équilibre, de telle sorte que les évaluations anormales commencent à partir de 3 pas. Si le patient ne comprend pas le test, l'investigateur peut le répéter de façon à ce que son évaluation corresponde à une estimation qu'il considère reflétant les limites du patient, plutôt que son incompréhension du test ou son manque de préparation. Observez la posture debout pour l'item 3.13.

0 = normal : aucun problème : retrouve son équilibre avec 1 ou 2 pas.
1 = minime : 3 à 5 pas, mais le sujet retrouve son équilibre sans aide.
2 = léger : plus de 5 pas, mais le sujet retrouve son équilibre sans aide.

3 = modéré : tient l'équilibre debout en sécurité, mais avec absence de réponse posturale ;

chute s'il n'est pas rattrapé par l'examinateur.

4 = sévère : très instable, tend à perdre l'équilibre spontanément ou juste avec une légère

poussée sur les épaules.

3.13 Posture ON | \_ |

La posture est évaluée alors que le patient se tient debout après s'être levé d'une chaise, pendant la marche, et pendant l'examen des réflexes posturaux. Si vous remarquez une mauvaise posture, dites au patient de se tenir droit et voyez si la posture s'améliore (voir option 2 ci-dessous). Evaluez la plus mauvaise posture observée dans ces 3 points. Observez la flexion et la tendance à pencher sur les côtés.

0 = normal ; aucun problème.

= minime : ne se tient pas tout à fait droit, mais la posture pourrait être considérée comme

normale pour une personne plus âgée.

2 = léger : flexion indiscutable, scoliose ou latéro-déviation, mais le patient peut corriger la

posture vers une posture normale quand on lui demande de le faire.

3 = modéré : posture fléchie, scoliose ou latéro-déviation qui ne peut être corrigée volontairement

vers une posture normale par le patient.

4 = sévère : flexion, scoliose ou attitude penchée avec une posture extrêmement anormale.

ON |

ON

#### 3.14 Spontanéité globale du mouvement (bradykinésie corporelle)

Cette évaluation globale combine toutes les observations sur la lenteur, les hésitations, l'amplitude réduite et la rareté du mouvement en général, incluant une réduction des gestes et du croisement des jambes. Cette observation est fondée sur l'impression globale de l'investigateur après avoir observé des gestes spontanés en position assise, et la nature du lever et de la marche.

0 = normal ; aucun problème.

1 = mínime : lenteur globale et pauvreté des mouvements spontanés minimes.
 2 = léger : lenteur globale et pauvreté des mouvements spontanés légères.
 3 = modéré : lenteur globale et pauvreté des mouvements spontanés modérées.
 4 = sévère : lenteur globale et pauvreté des mouvements spontanés sévères.

#### 3.15 Tremblement postural des mains

Tout tremblement incluant la réémergence du tremblement de repos présent dans cette posture, doit être inclus dans cette évaluation. Cotez chaque main séparément. Cotez la plus grande amplitude observée. Donnez l'instruction au patient d'étendre les bras devant son corps, paumes vers le bas. Le poignet doit être droit et les doigts confortablement séparés de sorte qu'ils ne se touchent pas. Observez cette posture pendant 10 secondes.

0 = normal ; pas de tremblement.

1 = minime : le tremblement est présent mais a moins d'1

cm d'amplitude.

MD | \_ |

2 = léger : le tremblement a au moins 1 mais pas plus de 3

cm d'amplitude.

3 = modéré : le tremblement a au moins 3 mais pas plus de 10 MG | \_ |

cm d'amplitude.

4 = sévère : le tremblement a au moins 10 cm d'amplitude.

#### 3.16 Tremblement d'action des mains

Ce test est fondé sur la manœuvre du doigt - nez. Le bras commençant avec la position tendue, faites que le patient exécute au moins 3 manœuvres de doigt - nez avec chaque main, atteignant aussi loin que possible le doigt de l'investigateur. La manœuvre du doigt - nez devra être effectuée assez lentement pour ne cacher aucun tremblement pouvant survenir avec des mouvements de bras très rapide. Répétez avec l'autre main, en évaluant chaque main séparément. Le tremblement peut être présent à travers le mouvement ou alors qu'il a atteint l'une ou l'autre cible (nez ou doigt). Evaluez la plus grande amplitude observée.

ON

0 = normal ; pas de tremblement.

1 = minime : le tremblement est présent mais inférieur à 1 MD | \_ |

cm d'amplitude.

2 = léger : le tremblement a au moins 1 mais pas plus de 3 MG | \_ |

cm d'amplitude.

3 = modéré : le tremblement a au moins 3 mais pas plus de 10

cm d'amplitude.

4 = sévère : le tremblement a au moins 10 cm d'amplitude.

#### 3.17 Amplitude du tremblement de repos

Cet item et le suivant ont été mis intentionnellement à la fin de l'examen afin de permettre à l'évaluateur de rassembler des observations sur le tremblement de repos pouvant apparaître à n'importe quel moment de l'examen, incluant l'attitude tranquillement assise du patient, la marche et toutes les activités pendant lesquelles certaines parties du corps sont en mouvement, mais d'autres sont au repos. Cotez

ON

### INITIALES PATIENT : | \_ | / | N° D'INCLUSION : | \_ | |

l'amplitude maximum observée à n'importe quel moment en tant que score final. Cotez seulement l'amplitude et non la persistance ou l'intermittence du tremblement. Dans le cadre de cette évaluation, le patient devra être tranquillement assis dans un fauteuil, les mains sur les accoudoirs (et non sur les genoux), et les pieds confortablement posés au sol pendant 10 secondes sans aucune autre directive. Le tremblement de repos est évalué séparément pour les 4 membres et aussi pour l'ensemble lèvre / mâchoire. Evaluez seulement l'amplitude maximum observée à n'importe quel moment en tant qu'évaluation finale.

Evaluation des extrémités :

sévère

0 = normal : pas de tremblement.

1 = minime : < 1 cm en amplitude maximale.

2 = léger : > à 1 cm mais < à 3 cm en amplitude

MSG |\_ |

MSG |\_ |

MSG |\_ |

MSG |\_ |

MIG |\_ |

Evaluation pour la lèvre/la mâchoire :

n = normal . pas de tremblement.

1 = minime : < 1 cm en amplitude maximale. ON

2 = léger : > à 1 cm mais < à 2 cm en amplitude maximale. Lèvre, mâchoire | \_ |

3 = modéré ; > à 2 cm mais < à 3 cm en amplitude maximale.

> à 10 cm en amplitude maximale.

4 = sévère ; > à 3 cm en amplitude maximale.

### 3.18 Constance du tremblement de repos ON | \_ |

Cet item reçoit une seule évaluation pour tout le tremblement de repos et se focalise sur la constance du tremblement de repos pendant la période de l'examen quand les différentes parties du corps sont au repos. Il est coté délibérément à la fin de l'examen de telle sorte que plusieurs minutes d'information peuvent être regroupées dans la cotation.

o = normal : pas de tremblement.

1 = minime : le tremblement de repos est présent, inférieur à 25 % de la période entière de

l'examen.

2 = léger : le tremblement de repos est présent, entre 26-50% de la période entière de l'examen.

3 = modéré : le tremblement de repos est présent, entre 51 à 75 % de la période entière de

l'examen.

4 = sévère : le tremblement de repos est présent, plus de 75 % de la période entière de l'examen.

| | INITIAL | ES PATIENT : _ / _ | N° D'INCLUSION : _ _ |
|---|---|---|---|
| | RETENT | TISSEMENT DES DYSKINESIES SUR | R LES EVALUATIONS DE LA PARTIE III |
| A | Des dyskiné | sies (chorée ou dystonie) étaient-elle | es présentes pendant l'examen ? |
| | OUI | one (energe ou ayereme) etaiem em | oo procentee pendant revamen r |
| | NON | | |
| B. | Si oui, ces m | ouvements ont-ils interférés avec ve | os évaluations ? |
| | OUI | | |
| | NON | | |
| Pa | artie IV : | complications motrices | |
| | DV0KW50 | | |
| A | . DYSKINES | ES (à l'exclusion de la période OFF | <u>de</u> |
| | dvstonie) | | |
| _ | | | |
| | | assé avec des dyskinésies | más at puis les hourse de dyskinésies. Calcular |
| Déte<br>e p<br>com<br>d'év<br>nou | erminez les he<br>ourcentage. S<br>ime référence<br>valuer. Vous<br>uvements dysl<br>uvements dysl | ures habituelles d'éveil pendant la jou<br>si le patient a des dyskinésies durar<br>pour vous assurer que les patients et<br>pouvez aussi utiliser vos propres cor<br>kinétiques que vous avez vu précéd<br>kinétiques types vus sur d'autres pa | nt la consultation, vous pouvez les lui signaler<br>t les aidants comprennent ce qu'ils sont en train<br>mpétences d'interprétation pour représenter les<br>demment chez le patient, ou leur montrer des |
| Déte<br>e p<br>com<br>d'év<br>nou<br>nou<br>doul | erminez les he<br>ourcentage. S<br>ame référence<br>valuer. Vous<br>uvements dysi<br>uvements dysi<br>loureuse du m | ures habituelles d'éveil pendant la jou<br>si le patient a des dyskinésies durar<br>pour vous assurer que les patients et<br>pouvez aussi utiliser vos propres co<br>kinétiques que vous avez vu précéd<br>kinétiques types vus sur d'autres pa<br>atin et de la nuit. | nt la consultation, vous pouvez les lui signaler<br>t les aidants comprennent ce qu'ils sont en train<br>mpétences d'interprétation pour représenter les<br>demment chez le patient, ou leur montrer des<br>atients. Excluez de cette question la dystonie |
| Déte<br>e p<br>com<br>d'év<br>mou<br>mou<br>doul | erminez les he<br>lourcentage. Some référence<br>valuer. Vous<br>uvements dysi<br>uvements dysi<br>loureuse du m<br>cours de la s | sures habituelles d'éveil pendant la jou<br>si le patient a des dyskinésies durar<br>pour vous assurer que les patients et<br>pouvez aussi utiliser vos propres coi<br>kinétiques que vous avez vu précéd<br>kinétiques types vus sur d'autres pa<br>atin et de la nuit.<br>semaine précédente, combien d'heur | umée et puis les heures de dyskinésies. Calculez nt la consultation, vous pouvez les lui signaler t les aidants comprennent ce qu'ils sont en train mpétences d'interprétation pour représenter les demment chez le patient, ou leur montrer des atients. Excluez de cette question la dystonie pres dormez-vous habituellement sur une base a sieste diurne ? D'accord, si vous dormez heures vous êtes |
| Déte<br>e p<br>com<br>l'év<br>nou<br>nou<br>loul<br>Au | erminez les he<br>ourcentage. S<br>ime référence<br>valuer. Vous<br>uvements dysi<br>uvements dysi<br>loureuse du m<br>cours de la s<br>tidienne, en i | ures habituelles d'éveil pendant la jou<br>si le patient a des dyskinésies durar<br>pour vous assurer que les patients et<br>pouvez aussi utiliser vos propres cor<br>kinétiques que vous avez vu précéd<br>kinétiques types vus sur d'autres pa<br>atin et de la nuit.<br>semaine précédente, combien d'heur<br>ncluant le sommeil nocturne et la | nt la consultation, vous pouvez les lui signaler<br>t les aidants comprennent ce qu'ils sont en train<br>mpétences d'interprétation pour représenter les<br>demment chez le patient, ou leur montrer des<br>atients. Excluez de cette question la dystonie<br>tres dormez-vous habituellement sur une base<br>a sieste diurne ? D'accord, si vous dormez<br>heures, vous êtes |
| Déte<br>e p<br>com<br>l'év<br>mou<br>mou<br>loul<br>Au<br>mou<br>évei<br>mou | erminez les he courcentage. Somme référence valuer. Vous sivements dysluvements dysluvements du m cours de la stidienne, en i illé(e) heures. | ures habituelles d'éveil pendant la jou<br>si le patient a des dyskinésies durar<br>pour vous assurer que les patients et<br>pouvez aussi utiliser vos propres cor<br>kinétiques que vous avez vu précéd<br>kinétiques types vus sur d'autres pa<br>atin et de la nuit.<br>semaine précédente, combien d'heur<br>incluant le sommeil nocturne et la<br>Durant ces heures d'éveil, combien d'<br>cadiques ou avec secousses ? Ne | nt la consultation, vous pouvez les lui signaler t les aidants comprennent ce qu'ils sont en train mpétences d'interprétation pour représenter les demment chez le patient, ou leur montrer des atients. Excluez de cette question la dystonie ures dormez-vous habituellement sur une base a sieste diurne ? D'accord, si vous dormez heures, vous êtes "heures au total avez-vous de dandinement, de comptez pas les périodes où vous avez des |
| Déte<br>e p<br>com<br>d'év<br>mou<br>doul<br>Au<br>doul<br>doul<br>doul<br>doul<br>doul<br>doul<br>doul<br>dou | erminez les he<br>ourcentage. Se<br>me référence<br>valuer. Vous<br>svements dyst<br>loureuse du m<br>cours de la stidienne, en i<br>illé(e) heures.<br>svements sacinblements, qui | vures habituelles d'éveil pendant la jour si le patient a des dyskinésies durar pour vous assurer que les patients et pouvez aussi utiliser vos propres corkinétiques que vous avez vu précéd kinétiques types vus sur d'autres paratin et de la nuit. semaine précédente, combien d'heur ncluant le sommeil nocturne et la Durant ces heures d'éveil, combien d'cadiques ou avec secousses ? Ne set une secousse régulière d'arrière et | nt la consultation, vous pouvez les lui signaler tes aidants comprennent ce qu'ils sont en train mpétences d'interprétation pour représenter les demment chez le patient, ou leur montrer des atients. Excluez de cette question la dystonie ures dormez-vous habituellement sur une base a sieste diurne ? D'accord, si vous dormez heures, vous êtes l'heures au total avez-vous de dandinement, de comptez pas les périodes où vous avez des en avant, ou les périodes vous avez des crampes |
| Déte<br>e p<br>com<br>d'év<br>mou<br>doul<br>Au<br>quot<br>évei<br>mou<br>frem<br>doul | erminez les he<br>ourcentage. S<br>imme référence. S<br>invements dysl<br>oureuse du m<br>cours de la s<br>tidienne, en i<br>illé(e) heures.<br>illé(e) heures.<br>ourements sacinblements, qui<br>loureuses au judientes sacinblements, qui<br>loureuses au judientes sacinblements, qui<br>loureuses au judientes sacinblements, qui<br>loureuses au judientes sacinblements, qui<br>loureuses au judientes sacinblements, qui loureuses au judientes sacinblements sacinblements qui loureuses au judiente sacinblements qui loureuses au judiente sacinblements qui loureuses au judiente sacinblements qui loureuses au judiente sacinblemente saci | vures habituelles d'éveil pendant la jours le patient a des dyskinésies durar pour vous assurer que les patients et pouvez aussi utiliser vos propres coixinétiques que vous avez vu précéd kinétiques types vus sur d'autres pa atin et de la nuit. semaine précédente, combien d'heur ncluant le sommeil nocturne et la Durant ces heures d'éveil, combien d'cadiques ou avec secousses ? Ne est une secousse régulière d'arrière e pied ou des spasmes tôt le matin, o | nt la consultation, vous pouvez les lui signaler t les aidants comprennent ce qu'ils sont en train mpétences d'interprétation pour représenter les demment chez le patient, ou leur montrer des atients. Excluez de cette question la dystonie ures dormez-vous habituellement sur une base a sieste diurne ? D'accord, si vous dormez heures, vous êtes l'heures au total avez-vous de dandinement, de comptez pas les périodes où vous avez des en avant, ou les périodes vous avez des crampes ou pendant la nuit. Je vous demanderai de m'en |
| Déte<br>e p<br>com<br>d'év<br>mou<br>doul<br>doul<br>doul<br>évei<br>mou<br>rem<br>doul<br>parke | erminez les he<br>ourcentage. S<br>imme référence<br>valuer. Vous<br>syements dysl<br>syements dysl<br>loureuse du m<br>cours de la stidienne, en i<br>illé(e) heures.<br>syements sacconblements, qui<br>loureuses au<br>jer plus tard. | vures habituelles d'éveil pendant la jour si le patient a des dyskinésies durar pour vous assurer que les patients et pouvez aussi utiliser vos propres cokinétiques que vous avez vu précéd kinétiques types vus sur d'autres paratin et de la nuit. semaine précédente, combien d'heur ncluant le sommeil nocturne et la Durant ces heures d'éveil, combien d'acidiques ou avec secousses ? Ne est une secousse régulière d'arrière e poied ou des spasmes tôt le matin, o Concentrez-vous seulement sur ce | nt la consultation, vous pouvez les lui signaler tiles aidants comprennent ce qu'ils sont en train mpétences d'interprétation pour représenter les demment chez le patient, ou leur montrer des atients. Excluez de cette question la dystonie tres dormez-vous habituellement sur une base a sieste diurne ? D'accord, si vous dormez heures, vous êtes l'heures au total avez-vous de dandinement, de comptez pas les périodes où vous avez des propendant la nuit. Je vous demanderai de m'en es types de dandinement, de mouvements |
| Déte<br>peom<br>d'éver<br>mou<br>doul<br>doul<br>dever<br>éver<br>mou<br>rem<br>doul<br>doul<br>dever<br>ever<br>mou<br>rem<br>doul<br>doul<br>doul<br>doul<br>doul<br>doul<br>dever<br>mou<br>dever<br>dev | erminez les he<br>ourcentage. S<br>me référence<br>raluer. Vous<br>svements dys<br>loureuse du m<br>cours de la s<br>tidienne, en i<br>illé(e) heures.<br>illé(e) heures sacun<br>holements, qui<br>loureuses au<br>er plus tard.<br>cadiques ou a | ures habituelles d'éveil pendant la jou si le patient a des dyskinésies durar pour vous assurer que les patients et pouvez aussi utiliser vos propres cokinétiques que vous avez vu précéd kinétiques types vus sur d'autres paratin et de la nuit. Semaine précédente, combien d'heur ncluant le sommeil nocturne et la Durant ces heures d'éveil, combien d'actiques ou avec secousses ? Ne est une secousse régulière d'arrière e pied ou des spasmes tôt le matin, o Concentrez-vous seulement sur ce vec secousses. Additionnez toutes le | nt la consultation, vous pouvez les lui signaler t les aidants comprennent ce qu'ils sont en train mpétences d'interprétation pour représenter les demment chez le patient, ou leur montrer des atients. Excluez de cette question la dystonie ures dormez-vous habituellement sur une base a sieste diurne ? D'accord, si vous dormez heures, vous êtes l'heures au total avez-vous de dandinement, de comptez pas les périodes où vous avez des en avant, ou les périodes vous avez des crampes ou pendant la nuit. Je vous demanderai de m'en |
| Déte<br>e p<br>com<br>l'éven<br>mou<br>doul<br>devei<br>mou<br>rem<br>doul<br>park<br>sacces q | erminez les he pourcentage. Some référence valuer. Vous avements dyslavements dyslavements de la stidienne, en i illé(e) heures avements sacrablements, qui loureuses au juer plus tard, cadiques ou a juelles ceux-ci | ures habituelles d'éveil pendant la jou si le patient a des dyskinésies durar pour vous assurer que les patients et pouvez aussi utiliser vos propres corkinétiques que vous avez vu précéd kinétiques types vus sur d'autres patient de la nuit. semaine précédente, combien d'heur incluant le sommeil nocturne et la Durant ces heures d'éveil, combien d'adiques ou avec secousses ? Ne est une secousse régulière d'arrière e pied ou des spasmes tôt le matin, ou concentrez-vous seulement sur ce vec secousses. Additionnez toutes le surviennent habituellement. Combien | nt la consultation, vous pouvez les lui signaler tiles aidants comprennent ce qu'ils sont en train mpétences d'interprétation pour représenter les demment chez le patient, ou leur montrer des atients. Excluez de cette question la dystonie tres dormez-vous habituellement sur une base a sieste diurne ? D'accord, si vous dormez heures, vous êtes l'heures au total avez-vous de dandinement, de comptez pas les périodes où vous avez des en avant, ou les périodes vous avez des pu pendant la puit. Je vous demanderai de m'en les types de dandinement, de mouvements es heures éveillées pendant la journée durant |
| Déte<br>peom<br>d'éver<br>mou<br>doul<br>doul<br>dever<br>éver<br>mou<br>rem<br>doul<br>doul<br>dever<br>ever<br>mou<br>rem<br>doul<br>doul<br>doul<br>doul<br>doul<br>doul<br>dever<br>mou<br>dever<br>dev | erminez les he courcentage. S me référence valuer. Vous vements dysi vements dysi loureuse du m cours de la s tidienne, en i illé(e) heures. vements sacu holements, qui loureuses au j er plus tard. er diques ou a quelles ceux-ci = normal | ures habituelles d'éveil pendant la jou si le patient a des dyskinésies durar pour vous assurer que les patients et pouvez aussi utiliser vos propres corkinétiques que vous avez vu précéd kinétiques types vus sur d'autres pa atin et de la nuit. semaine précédente, combien d'heur incluant le sommeil nocturne et la Durant ces heures d'éveil, combien d'cadiques ou avec secousses ? Ne est une secousse régulière d'arrière e pied ou des spasmes tôt le matin, or Concentrez-vous seulement sur ce surviennent habituellement. Combien : pas de dyskinésies. | nt la consultation, vous pouvez les lui signaler tes aidants comprennent ce qu'ils sont en train mpétences d'interprétation pour représenter les demment chez le patient, ou leur montrer des atients. Excluez de cette question la dystonie tres dormez-vous habituellement sur une base a sieste diurne ? D'accord, si vous dormez heures, vous êtes heures au total avez-vous de dandinement, de comptez pas les périodes où vous avez des en avant, ou les périodes vous avez des crampes ou pendant la nuit. Je vous demanderai de m'en es types de dandinement, de mouvements sheures éveillées pendant la journée durant d'heures (utilisez ce nombre pour votre calcul). |
| Déte<br>e p<br>com<br>nou<br>nou<br>loul<br>doul<br>évei<br>mou<br>rem<br>doul<br>sacce<br>esq | erminez les he pourcentage. Some référence valuer. Vous avements dyslavements dyslavements de la stidienne, en i illé(e) heures avements sacrablements, qui loureuses au juer plus tard, cadiques ou a juelles ceux-ci | ures habituelles d'éveil pendant la jou si le patient a des dyskinésies durar pour vous assurer que les patients et pouvez aussi utiliser vos propres corkinétiques que vous avez vu précéd kinétiques types vus sur d'autres patient de la nuit. semaine précédente, combien d'heur incluant le sommeil nocturne et la Durant ces heures d'éveil, combien d'adiques ou avec secousses ? Ne est une secousse régulière d'arrière e pied ou des spasmes tôt le matin, ou concentrez-vous seulement sur ce vec secousses. Additionnez toutes le surviennent habituellement. Combien | nt la consultation, vous pouvez les lui signaler tes aidants comprennent ce qu'ils sont en train mpétences d'interprétation pour représenter les demment chez le patient, ou leur montrer des atients. Excluez de cette question la dystonie tres dormez-vous habituellement sur une base a sieste diurne ? D'accord, si vous dormez heures, vous êtes heures au total avez-vous de dandinement, de comptez pas les périodes où vous avez des en avant, ou les périodes vous avez des crampes ou pendant la nuit. Je vous demanderai de m'en es types de dandinement, de mouvements sheures éveillées pendant la journée durant d'heures (utilisez ce nombre pour votre calcul). |
| Déte promoud'éver moudoul d'éver moudoul de la control de | erminez les he courcentage. Some référence valuer. Vous sivements dysl sivements dysl sourceuse du m cours de la si tidienne, en i illé(e) heures. sivements saci nblements, qui loureuses au j er plus tard. a quelles ceux-ci = normal = minime | vures habituelles d'éveil pendant la jours le patient a des dyskinésies durar pour vous assurer que les patients et pouvez aussi utiliser vos propres con kinétiques que vous avez vu précéd kinétiques types vus sur d'autres paratin et de la nuit. Semaine précédente, combien d'heur ncluant le sommeil nocturne et la contrait ces heures d'éveil, combien d'adiques ou avec secousses ? Ne est une secousse régulière d'arrière en pied ou des spasmes tôt le matin, on Concentrez-vous seulement sur ce vec secousses. Additionnez toutes le surviennent habituellement. Combien pas de dyskinésies. | nt la consultation, vous pouvez les lui signaler tes aidants comprennent ce qu'ils sont en train mpétences d'interprétation pour représenter les demment chez le patient, ou leur montrer des atients. Excluez de cette question la dystonie tres dormez-vous habituellement sur une base a sieste diurne ? D'accord, si vous dormez heures, vous êtes heures au total avez-vous de dandinement, de comptez pas les périodes où vous avez des en avant, ou les périodes vous avez des crampes ou pendant la nuit. Je vous demanderai de m'en es types de dandinement, de mouvements sheures éveillées pendant la journée durant d'heures (utilisez ce nombre pour votre calcul). |

2 - total des heures avec dyskinésies\_\_\_\_\_\_ 3 - % de dyskinésies = ((2/1) x100)

1 - total des heures éveillées \_\_\_

#### 4.2 Retentissement fonctionnel des dyskinésies

Déterminez le degré de retentissement que les dyskinésies ont sur la fonction quotidienne du patient en termes d'activités et d'interactions sociales. Utilisez la réponse du patient et de l'aidant à vos questions et vos propres observations pendant la visite en consultation pour arriver à la meilleure réponse. Au cours de la semaine précédente, avez-vous eu des problèmes en faisant des choses ou en étant avec des gens lorsque ces mouvements saccadés apparaissaient ?vous ont-ils empêché de faire des choses ou d'être avec des gens ?

0 = normal : pas de dyskinésies ou pas de retentissement des dyskinésies sur les activités et les

interactions sociales.

1 = minime : les dyskinésies retentissent sur quelques activités, mais le patient effectue habituellement

toutes les activités et participe à toutes les interactions de la vie sociale pendant les

périodes dyskinétiques.

2 = léger : les dyskinésies retentissent sur beaucoup d'activités, mais le patient effectue

habituellement toutes les activités et participe à toutes les interactions de la vie

sociale pendant les périodes dyskinétiques.

3 = modéré : les dyskinésies retentissent sur les activités, au point que le patient ne peut effectuer

certaines activités et ou ne peut pas participer à certaines activités sociales pendant

les épisodes dyskinétiques.

4 = sévère : les dyskinésies retentissent sur la fonction au point que le patient ne peut effectuer

la plupart des activités et ou participer à la plupart des interactions sociales pendant

les épisodes dyskinétiques.

#### **B. FLUCTUATIONS MOTRICES**

#### 4.3 Durée des périodes ON

Utilisez le nombre d'heures éveillées provenant de 4.1 et déterminez les heures passées en condition OFF. Calculez le pourcentage. Si le patient a un épisode OFF durant la consultation, vous pouvez vous appuyer sur cet état comme référence. Vous pouvez aussi utiliser votre connaissance du patient pour décrire une période OFF typique. De plus, vous pouvez aussi utiliser vos propres compétences d'interprétation pour représenter une période OFF déjà vue auparavant chez le patient, ou leur montrer la fonction OFF typique d'autres patients. Notez le nombre type d'heures OFF, car vous aurez besoin de ce nombre pour compléter le 4.6.

Certains patients atteints de la maladie de Parkinson retirent un bon effet de leurs médications pendant les heures éveillées et nous appelons cela la période ON. D'autres patients prennent leurs médications mais ont encore quelques heures de baisse de régime, de période mauvaise, ralentie ou période de tremblement. Les médecins appellent ces mauvaises périodes, période OFF. Au cours de la semaine précédente, vous m'avez dit auparavant que vous êtes généralement éveilléheures par jour. Durant ces heures éveillées, combien d'heures au total avez-vous habituellement ce type de baisse régime ou épisode OFF (utilisez ce nombre pour vos calculs).

0 = normal : pas de période OFF.

1 = minime : < 25% du temps éveillé dans la journée.
2 = léger : de 26% à 50% du temps éveillé dans la journée.
3 = modéré : de 51% à 75% du temps éveillé dans la journée.

4 = sévère : > 75% du temps éveillé dans la journée.

| 1 - total des heures éveillées |
|--------------------------------|
| 2 - total des heures OFF |
| 3 - % OFF = ((2/1) x100) |

#### 4.4 Retentissement fonctionnel des fluctuations

Déterminez le degré de retentissement que les fluctuations motrices ont sur le fonctionnement quotidien du patient en termes d'activités et d'interactions sociales. Cette question se concentre sur la différence entre l'état OP et l'état OFF. Si le patient n'a pas de période OFF, l'évaluation doit être 0, mais il es patients ont de très légères fluctuations, il est encore possible de coter 0 sur cet item s'il n'y a pas de retentissement sur leurs activités. Utilisez la réponse du patient et de l'aidant à votre question et votre propre observation pendant la visite en consultation pour arriver à la meilleure réponse.

Réfléchissez à quel moment ces baisses de régime ou périodes OFF sont survenues au cours de la semaine précédente. Avez-vous habituellement plus de problème à faire les choses ou à être avec des gens par rapport au reste de la journée lorsque vous sentez que vos médicaments marchent bien ? Y-a-t-il certaines choses que vous faites habituellement pendant une bonne période, qui vous posent des problèmes ou que vous arrêtez de faire pendant une période de baisse de régime ?

0 = normal : pas de fluctuation ou pas de retentissement des fluctuations sur l'accomplissement

des

minime

: les fluctuations retentissent sur quelques activités, mais pendant la période OFF, le

patient accomplit habituellement toutes les activités et participe à toutes les interactions sociales qui surviennent typiquement pendant la période ON.

2 = léger : les fluctuations retentissent sur beaucoup d'activités, mais pendant la période OFF, le patient le accomplit encore habituellement toutes les activités et participe à toutes

le patient le accomplit encore habituellement toutes les activités et participe à toutes les interactions sociales qui surviennent typiquement pendant la période ON.

= modéré : les fluctuations retentissent sur la réalisation des activités pendant la période OFF au point que le patient n'accomplit habituellement pas certaines activités et ou ne

participe pas à certaines interactions sociales qui sont effectuées durant les périodes

ON..

4 = sévère : les fluctuations retentissent sur le fonctionnement au point que durant la période OFF

le patient n'accomplit pas la plupart des activités, ni ne participe à la plupart des

interactions sociales qui sont effectuées pendant les périodes ON.

#### 4.5 Complexité des fluctuations

Déterminez la prévisibilité habituelle des épisodes OFF, qu'ils soient dus à la dose, au moment de la journée, à la prise de nourriture ou à d'autres facteurs. Utilisez l'information fournie par le patient et les aidants et complétez avec vos propres observations. Vous demanderez si le patient peut s'attendre à ce qu'elles arrivent toujours à une période précise, survenant la plupart du temps à un moment particulier (dans ce cas- là, vous évaluerez d'avantage pour séparer minime de léger), ou à ce qu'elles arrivent quelquefois à un moment précis ou si elles sont totalement imprévisibles ? En réduisant le pourcentage, vous obtiendrez la réponse correcte.

Pour certains patients, les périodes mauvaises ou OFF arrivent à certains moments de la journée ou quand ils sont engagés dans des activités comme manger ou faire de l'exercice. Au cours de la semaine précédente, savez-vous habituellement quand vos périodes mauvaises vont survenir ? En d'autres mots, est-ce que vos baisses de régime apparaissent toujours à un moment donné ? Apparaissent-elles le plus souvent à un moment donné ? Apparaissent-elles seulement quelquefois à un moment donné ? Vos baisses de régime sont-elles totalement imprévisibles ?

0 = normal ; pas de fluctuation motrice.

1 = minime : les périodes OFF sont prévisibles tout ou presque tout le temps (> 75%).

2 = léger : les périodes OFF sont prévisibles la plupart du temps (51-75%). 3 = modéré : les périodes OFF sont prévisibles quelquefois (26-50%).

4 = sévère : les périodes OFF sont previsibles quelquefois (26-50 les périodes OFF sont rarement prévisibles (<25%).

#### C. DYSTONIE ON

#### 4.6 Dystonie douloureuse en état ON

Pour les patients qui ont des fluctuations motrices, déterminez dans quelle proportion des épisodes OFF comprennent habituellement une dystonie douloureuse ? Vous avez déjà déterminé le nombre d'heures en période OFF (4.3). Parmi ces heures, déterminez combien d'entre-elles sont associées à une dystonie et calculez le pourcentage. S'il n'y a pas de période OFF, notez 0. Dans une question que je vous ai posé(e)précédemment, vous dites avoir généralement d'heures de période mauvaise ou de temps « OFF » quand votre maladie de Parkinson est mal contrôlée. Pendant ces périodes mauvaises ou OFF, avez-vous habituellement des crampes ou des spasmes douloureux ? Sur un total de heures de cette période mauvaise, si vous ajoutez tous les moments de la journée durant lesquels ces crampes douloureuses apparaissent, combien d'heures cela

0 = normal : pas de dystonie ou pas de période OFF.
1 = minime : < 25% du temps en état OFF.
2 = léger : de 26% à 50% du temps en état OFF.
3 = modéré : de 51% à 75% du temps en état OFF. 4 = sévère > 75% du temps en état OFF.

2 - total des heures OFF avec dystonie

3 - % de dystonie OFF = ((2/1) x100) \_\_\_\_

1 - total des heures OFF \_

## 14.14 Appendix N – Hoehn and Yahr stage

A compléter lors du screening et Visite 4.

## **STADE HOEHN & YAHR**

| Stade 0 : pas de signe de la maladie. |
|---|
| Stade 1 : maladie unilatérale. |
| Stade 1,5 : maladie unilatérale, plus atteinte axiale. |
| Stade 2 : maladie bilatérale sans trouble de l'équilibre. |
| <b>Stade 2,5 :</b> maladie bilatérale légère avec rétablissement lors du test de la poussée. |
| Stade 3 : maladie bilatérale légère à modérée : une certaine instabilité posturale, |
| physiquement autonome. |
| Stade 4 : handicap sévère : toujours capable de marcher ou de se tenir debout sans |
| aide. |
| Stade 5 : malade en chaise roulante ou alité sauf s'il est aidé. |

### 14.15 Appendix O – Freezing of gait questionnaire.

A compléter à chaque visite : Baseline, Visite 3, et Visite 4.

#### **Evaluation Freezing – Kinésithérapie**

| ID Patient: | Date: | Visite: | |
|-------------|-------|---------|---|
| | | | İ |

Instructions pour l'administrateur :

Veuillez administrer le questionnaire suivant au patient, en notant sa réponse à chaque question posée avec le numéro correspondant. Le questionnaire doit être réalisé lorsque le patient est en condition "on". Les réponses doivent refléter l'expérience du patient au cours de la dernière semaine.

### 1. Lorsque vous êtes au plus mal, vous marchez :

- 0 Normalement
- 1 presque normalement parfois lentement
- 2 Lentement mais toujours sans aide
- 3 Avec une personne ou une aide technique
- 4 Marche impossible

### 2. Vos difficultés de marche affectent-elles vos activités quotidiennes ou votre indépendance ?

- 0 Pas du tout
- 1 Peu
- 2 Modérément
- 3 Enormément
- 4 Marche impossible

# 3. Ressentez-vous vos pieds « collés » au sol lors de la marche, lors des demi-tours ou lors de l'initiation de la marche ?

- 0 Jamais
- 1 Très rarement une fois par mois
- 2 Rarement une fois par semaine
- 3 Souvent au moins une fois par jour
- 4 Toujours a chaque fois que vous marchez

### 4. Quelle durée peuvent avoir vos épisodes de Freezing ?

- 0 Jamais arrivé
- 1.1 2.s
- 23 10 s
- 311 30 s
- 4 Impossible de marcher plus de 30 s

### 5. Quelle est la durée de votre épisode de freezing lors de l'initiation du premier pas ?

- 0 Aucune
- 1 Environ 1 s pour initier le pas
- 2 Environ 3 s pour initier le pas
- 3 Environ 10 s pour initier le pas
- 4 Environ 30 s pour initier le pas

#### 6. Quelle est la durée de votre épisode de freezing lors des demi-tours?

- 0 Aucune
- 1 Demi-tour en 1-2 s
- 2 Demi-tour en 3 10 s
- 3 Demi-tour en 11 30 s


4 Demi-tour en + de 30 s ou impossible

### 14.16 Appendix P – PDSS 2

A remplir à chaque visite : Baseline, Visite 1, Visite 2, Visite 3 et Visite 1.2, Visite 2.2, Visite 4 si applicable.

#### Questionnaire sur le sommeil Maladie de Parkinson (PDSS)

Comment mesureriez-vous les éléments suivants d'après ce que vous avez vécu au cours des 7 derniers jours ? (Mettez une croix sur la ligne de la page de droite, à l'endroit correspondant à votre situation)



#### Numéro de / ID Patient:

Date de l'évaluation:..../.....
ECHELLE VISUELLE ANALOGIQUE pour PDSS

| 1. | |
|---|---|
| 2. | TRES MAJVAISE DECEMBER DECEMBER |
| | TCWOURS JAMAS: 0 1 2 3 4 5 6 7 8 9 10 |
| 3. | TOUJOURS JAMAS: |
| 4. | 0 1 2 3 4 5 6 7 8 9 11<br>TOUJOURS |
| 5. | 0 1 2 3 4 5 6 7 8 9 10<br>TOWOURS |
| 6. | |
| 7. | TOURDORS JAMA: http://doi.org/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.100/10.1000/10.1000/10.1000/10.1000/10.1000/10.1000/10.1000/10.1000 |
| | TOWOURS JAMAS: 0 1 2 3 4 5 6 7 8 9 10 |
| 8. | TOUJOURS JAMAS: |
| 9. | JAMA: |
| 10. | 0 1 2 3 4 5 6 7 8 9 11<br>TOUJOURS |
| 11. | 0 1 2 3 4 5 6 7 8 9 10<br>TOWOURS |
| 12. | |
| 13. | TOURDURS |
| | TOWOURS JAMAS: |
| 14. | JAMA: |
| 15. | 0 1 2 3 4 5 6 7 8 9 10<br>FREQUEMMENT JAMAS |

# 14.17 Appendix Q – Patient global impression of severity (PGI-S) and improvement (PGI-I)

### 14.17.1 PGI-S: patient global impression of severity

A compléter à la visite Baseline

Veuillez mettre une croix en face de la réponse qui décrit le mieux votre état de santé actuel :

- o Pas de symptôme
- o Très peu de symptômes
- o Peu de symptôme
- o Symptômes modérés
- o Symptômes légèrement sévères
- o Symptômes sévères
- Symptômes très sévères

### 14.17.2 PGI-I: patient global impression of improvement

A compléter à Visite 3 et Visite 4 si applicable.

Veuillez mettre une croix en face de la réponse qui décrit le mieux l'évolution de votre état de santé depuis votre dernière visite :

- o Beaucoup mieux
- o Mieux
- o Pas de changement
- o Un peu moins bien
- o Moins bien
- o Beaucoup moins bien

# 14.18 Appendix R – Clinical global impression of severity (CGI-S) and improvement (CGI-I)

### 14.18.1 Clinical global impression of severity

A compléter à la visite Baseline

Veuillez mettre une croix en face de la réponse qui décrit le mieux l'état de santé actuel du patient

- o Pas de symptôme
- o Très peu de symptômes
- o Peu de symptôme
- o Symptômes modérés
- o Symptômes légèrement sévères
- o Symptômes sévères
- Symptômes très sévères

### 14.18.2 Clinical global impression of improvement

A compléter à Visite 3 et Visite 4 si applicable.

Veuillez mettre une croix en face de la réponse qui décrit le mieux l'évolution de l'état de santé du patient depuis sa dernière visite :

- o Beaucoup mieux
- o Mieux
- o Pas de changement
- o Un peu moins bien
- o Moins bien
- o Beaucoup moins bien

### 14.19 Appendix S – User guides

14.19.1 User guide for patient in the conventional physiotherapy arm





### 14.19.2 User guide for patient in the FeetMe Rehabilitation arm







#### 15 REFERENCES

- Abbruzzese, G., Marchese, R., Avanzino, L., Pelosin, E., 2016. Rehabilitation for Parkinson's disease: Current outlook and future challenges. Parkinsonism Relat Disord 22 Suppl 1, S60-64. https://doi.org/10.1016/j.parkreldis.2015.09.005
- Allen, N.E., Schwarzel, A.K., Canning, C.G., 2013. Recurrent Falls in Parkinson's Disease: A Systematic Review. Parkinson's Disease 2013, 1–16. https://doi.org/10.1155/2013/906274
- American Thoracic Society, 2002. ATS Statement Guidelines for the Six-Minute Walk Test. Am J Respir Crit Care Med 166, 111–117. https://doi.org/10.1164/ajrccm.166.1.at1102
- Ashburn, A., Stack, E., Ballinger, C., Fazakarley, L., Fitton, C., 2008. The circumstances of falls among people with Parkinson's disease and the use of Falls Diaries to facilitate reporting. Disability and Rehabilitation 30, 1205–1212. https://doi.org/10.1080/09638280701828930
- Barbour, P.J., Arroyo, J., High, S., Fichera, L.B., Staska-Pier, M.M., McMahon, M.K., 2016. Telehealth for patients with Parkinson's disease: delivering efficient and sustainable long-term care. Hospital Practice 44, 92–97. https://doi.org/10.1080/21548331.2016.1166922
- Benayoun, Y., Éric Molière, Caroline Moriceau, Nicolas Ponchaut, 2019. LES MASSEURS-KINÉSITHÉRAPEUTES EN ÎLE-DE-FRANCE AUJOURD'HUI ET DEMAIN.
- Bettger, J.P., Thoumi, A., Marquevich, V., Groote, W.D., Battistella, L.R., Imamura, M., Ramos, V.D., Wang, N., Dreinhoefer, K.E., Mangar, A., Ghandi, D.B.C., Ng, Y.S., Lee, K.H., Ming, J.T.W., Pua, Y.H., Inzitari, M., Mmbaga, B.T., Shayo, M.J., Brown, D.A., Carvalho, M., Oh-Park, M., Stein, J., 2020. COVID-19: maintaining essential rehabilitation services across the care continuum. BMJ Global Health 5, e002670. https://doi.org/10.1136/bmjgh-2020-002670
- Braun, T., Weidmann, R., Möller, J.C., Ammann, A., Marks, D., 2021. The impact of a coronavirus disease 2019 pandemic-related interruption of regular physical rehabilitation on functional abilities in a patient with two chronic neurological diseases: a case report. Journal of Medical Case Reports 15, 503. https://doi.org/10.1186/s13256-021-03119-3
- Caglar, A.T., Gurses, H.N., Mutluay, F.K., Kiziltan, G., 2005. Effects of home exercises on motor performance in patients with Parkinson's disease. Clin Rehabil 19, 870–877. https://doi.org/10.1191/0269215505cr924oa
- Cavallieri, F., Sireci, F., Fioravanti, V., Toschi, G., Rispoli, V., Antonelli, F., Costantini, M., Ghirotto, L., Valzania, F., 2021. Parkinson's disease patients' needs during the COVID-19 pandemic in a red zone: A framework analysis of open-ended survey questions. European Journal of Neurology 28, 3254–3262. https://doi.org/10.1111/ene.14745
- Chaudhuri, K.R., 2002. The Parkinson's disease sleep scale: a new instrument for assessing sleep and nocturnal disability in Parkinson's disease. Journal of Neurology, Neurosurgery & Psychiatry 73, 629–635. https://doi.org/10.1136/jnnp.73.6.629
- Chaudhuri, K.R., Schapira, A.H., 2009. Non-motor symptoms of Parkinson's disease: dopaminergic pathophysiology and treatment. The Lancet Neurology 8, 464–474. https://doi.org/10.1016/S1474-4422(09)70068-7
- Cohen J. Statistical Power Analysis for the Behavioral Sciences. 2nd ed. Hillsdale, NJ: Lawrence Earlbaum Associates; 1988.
- Creaby, M.W., Cole, M.H., 2018. Gait characteristics and falls in Parkinson's disease: A systematic review and meta-analysis. Parkinsonism & Related Disorders 57, 1–8. https://doi.org/10.1016/j.parkreldis.2018.07.008
- David, R., Billot, M., Delaire, L., Roulaud, M., Lorgeoux, B., Foucault, P., Louis, F., Duprey, E., Lapoulvereyrie, R., Meklat, H., Visentin, C., Cognon, L., Germaneau, A., Vendeuvre, T., Rigoard, P., 2019. Use of FeetMe monitor® connected soles for real-time measurement of spatial and temporal walking parameters: an illustrative case from the REWALK pilot study highlighting the objectivity of a spastic hemiparetic patient assessment. Computer Methods in Biomechanics and Biomedical Engineering 22, S257–S259. https://doi.org/10.1080/10255842.2020.1714264
- Deane, K.H.O., Ellis-Hill, C., Jones, D., Whurr, R., Ben-Shlomo, Y., Playford, E.D., Clarke, C.E., 2002. Systematic review of paramedical therapies for Parkinson's disease. Movement Disorders 17, 984–991. https://doi.org/10.1002/mds.10197

- Domínguez, A.G., Hochsprung, A., Duarte, S.P., Camino, C.P., Rodríguez, A.A., Durán, C., Navarro, G., Venegas, A., Moreno, M.J., Hernández, B., Izquierdo, G., 2020. Study for the Validation of the FeetMe® Integrated Sensor Insole System Compared to GAITRite® System to Assess the Characteristics of the Gait in Patients with Multiple Sclerosis (4038). Neurology 94.
- Ellis, T., de Goede, C.J., Feldman, R.G., Wolters, E.C., Kwakkel, G., Wagenaar, R.C., 2005. Efficacy of a physical therapy program in patients with Parkinson's disease: a randomised controlled trial. Arch Phys Med Rehabil 86, 626–632. https://doi.org/10.1016/j.apmr.2004.08.008
- Farid, L., Jacobs, D., Do Santos, J., Simon, O., Gracies, J.-M., Hutin, E., 2021. FeetMe® Monitor-connected insoles are a valid and reliable alternative for the evaluation of gait speed after stroke. Topics in Stroke Rehabilitation 28, 127–134. https://doi.org/10.1080/10749357.2020.1792717
- Fasano, A., Canning, C.G., Hausdorff, J.M., Lord, S., Rochester, L., 2017. Falls in Parkinson's disease: A complex and evolving picture: Falls and PD. Mov Disord. 32, 1524–1536. https://doi.org/10.1002/mds.27195
- Franchignoni, F., Horak, F., Godi, M., Nardone, A., Giordano, A., 2010. Using psychometric techniques to improve the Balance Evaluation Systems Test: the mini-BESTest. J Rehabil Med 42, 323–331. https://doi.org/10.2340/16501977-0537
- Giladi, N., Shabtai, H., Simon, E.S., Biran, S., Tal, J., Korczyn, A.D., 2000. Construction of freezing of gait questionnaire for patients with Parkinsonism. Parkinsonism & Related Disorders 6, 165–170. https://doi.org/10.1016/S1353-8020(99)00062-0
- Goetz, C.G., Poewe, W., Rascol, O., Sampaio, C., Stebbins, G.T., Counsell, C., Giladi, N., Holloway, R.G., Moore, C.G., Wenning, G.K., Yahr, M.D., Seidl, L., 2004. *Movement Disorder Society Task Force report on the Hoehn and Yahr staging scale: Status and recommendations The Movement Disorder Society Task Force on rating scales for Parkinson's disease. Mov Disord.* 19, 1020–1028. https://doi.org/10.1002/mds.20213
- Goetz, C.G., Tilley, B.C., Shaftman, S.R., Stebbins, G.T., Fahn, S., Martinez-Martin, P., Poewe, W., Sampaio, C., Stern, M.B., Dodel, R., Dubois, B., Holloway, R., Jankovic, J., Kulisevsky, J., Lang, A.E., Lees, A., Leurgans, S., LeWitt, P.A., Nyenhuis, D., Olanow, C.W., Rascol, O., Schrag, A., Teresi, J.A., van Hilten, J.J., LaPelle, N., 2008. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): Scale presentation and clinimetric testing results: MDS-UPDRS: Clinimetric Assessment. Mov. Disord. 23, 2129–2170. https://doi.org/10.1002/mds.22340
- Granja, Hochsprung, Palao, Páramo, Alemán, Durán, Navarro, Hernández, Romero, Venegas, Izquierdo, 2019. Study for the Validation of the FeetMe® Integrated Sensor Insole System Compared to GAITRite® System to Assess the Characteristics of the Gait in Patients with Multiple Sclerosis: Results of the Interim Analysis. Presented at the 35th Congress of the European Committee for Treatment and Research in Multiple Sclerosis and 24th Annual Conference of Rehabilitation in Multiple Sclerosis, Stockholm, Sweden.
- Guy, W., 1976. ECDEU assessment manual for psychopharmacology. U.S. Department of Health, Education, and Welfare, Public Health Service, Alcohol, Drug Abuse, and Mental Health Administration, National Institute of Mental Health, Psychopharmacology Research Branch, Division of Extramural Research Programs.
- Hass, C., Bishop, M., Moscovich, M., Stegemöller, E.L., Skinner, J., Malaty, I.A., Shukla, A.W., McFarland, N., Okun, M.S. 2014. Defining the Clinically Meaningful Difference in Gait Speed in Persons With Parkinson Disease. J Neurol Phys Ther 2014;38(4):233-8.
- Haute Autorité de Santé, 2016. Guide du parcours de soins Maladie de Parkinson.
- Hirsch, M.A., Toole, T., Maitland, C.G., Rider, R.A., 2003. The effects of balance training and high-intensity resistance training on persons with idiopathic Parkinson's disease. Arch Phys Med Rehabil 84, 1109–1117. https://doi.org/10.1016/s0003-9993(03)00046-7
- Hoehn, M.M., Yahr, M.D., 1967. Parkinsonism: onset, progression, and mortality. Neurology 17, 427–442.
- Jacobs, D., Farid, L., Ferré, S., Herraez, K., Gracies, J.-M., Hutin, E., 2021. Evaluation of the Validity and Reliability of Connected Insoles to Measure Gait Parameters in Healthy Adults. Sensors 21, 6543. https://doi.org/10.3390/s21196543

- Jenkinson, C., Fitzpatrick, R., Peto, V., Greenhall, R., Hyman, N., 1997. The PDQ-8: Development and validation of a short-form parkinson's disease questionnaire. Psychology & Health 12, 805–814. https://doi.org/10.1080/08870449708406741
- Keus SHJ, Munneke M, Graziano M, et al. European Physiotherapy Guideline for Parkinson's Disease. 2014; KNGF/ParkinsonNet, the Netherlands
- Laplanche, A., Ferré, S., Jacobs, D., Farid, L., Post, A., Moreau, C., Degos, B., Baille, G., 2021. Self rehabilitation with connected insoles in Parkinson's Disease: results of a pilot study
- Lunardini, F., Malavolti, M., Pedrocchi, A.L.G., Borghese, N.A., Ferrante, S., 2021. A mobile app to transparently distinguish single- from dual-task walking for the ecological monitoring of agerelated changes in daily-life gait. Gait & Posture 86, 27–32. https://doi.org/10.1016/j.gaitpost.2021.02.028
- Mak, M.K., Wong-Yu, I.S., Shen, X., Chung, C.L., 2017. Long-term effects of exercise and physical therapy in people with Parkinson disease. Nat Rev Neurol 13, 689–703. https://doi.org/10.1038/nrneurol.2017.128
- McGinley, J.L., Martin, C., Huxham, F.E., Menz, H.B., Danoudis, M., Murphy, A.T., Watts, J.J., Iansek, R., Morris, M.E., 2011. Feasibility, Safety, and Compliance in a Randomised Controlled Trial of Physical Therapy for Parkinson's Disease. Parkinson's Disease 2012, e795294. https://doi.org/10.1155/2012/795294
- Mehrholz, J., Kugler, J., Storch, A., Pohl, M., Hirsch, K., Elsner, B., 2016. Treadmill training for patients with Parkinson Disease. An abridged version of a Cochrane Review. European journal of physical and rehabilitation medicine 52.
- Millage, B., Vesey, E., Finkelstein, M., Anheluk, M. 2017. "Effect on Gait Speed, Balance, Motor Symptom Rating, and Quality of Life in Those with Stage I Parkinson's Disease Utilizing LSVT BIG®", Rehabilitation Research and Practice, vol. 2017, Article ID 9871070, 8 pages, 2017. https://doi.org/10.1155/2017/9871070
- Muslimović, D., Post, B., Speelman, J.D., Schmand, B., Haan, R.J. de, 2008. Determinants of disability and quality of life in mild to moderate Parkinson disease. Neurology 70, 2241–2247. https://doi.org/10.1212/01.wnl.0000313835.33830.80
- Nasreddine, Z.S., Phillips, N.A., Bédirian, V., Charbonneau, S., Whitehead, V., Collin, I., Cummings, J.L., Chertkow, H., 2005. The Montreal Cognitive Assessment, MoCA: A Brief Screening Tool For Mild Cognitive Impairment. Journal of the American Geriatrics Society 53, 695–699. https://doi.org/10.1111/j.1532-5415.2005.53221.x
- Paul, S.S., Canning, C.G., Sherrington, C., Lord, S.R., Close, J.C.T., Fung, V.S.C., 2013. Three simple clinical tests to accurately predict falls in people with Parkinson's disease: Fall Predictors in PD. Mov Disord. 28, 655–662. https://doi.org/10.1002/mds.25404
- Peto, V., Jenkinson, C., Fitzpatrick, R., Greenhall, R., 1995. The development and validation of a short measure of functioning and well being for individuals with Parkinson's disease. Qual Life Res 4, 241–248. https://doi.org/10.1007/BF02260863
- Pickering, R.M., Grimbergen, Y.A.M., Rigney, U., Ashburn, A., Mazibrada, G., Wood, B., Gray, P., Kerr, G., Bloem, B.R., 2007. A meta-analysis of six prospective studies of falling in Parkinson's disease. Mov Disord 22, 1892–1900. https://doi.org/10.1002/mds.21598
- Poewe, W., Seppi, K., Tanner, C.M., Halliday, G.M., Brundin, P., Volkmann, J., Schrag, A.-E., Lang, A.E., 2017. Parkinson disease. Nat Rev Dis Primers 3, 17013. https://doi.org/10.1038/nrdp.2017.13
- Rennie L, Opheim A, Dietrichs E, Löfgren N, Franzén E. 2021. Highly challenging balance and gait training for individuals with Parkinson's disease improves pace, rhythm and variability domains of gait A secondary analysis from a randomized controlled trial. Clinical Rehabilitation. 35(2):200-212. doi:10.1177/0269215520956503
- Ridgel, A.L., Vitek, J.L., Alberts, J.L., 2009. Forced, Not Voluntary, Exercise Improves Motor Function in Parkinson's Disease Patients. Neurorehabil Neural Repair 23, 600–608. https://doi.org/10.1177/1545968308328726
- Rodríguez-Molinero, A., Herrero-Larrea, A., Miñarro, A., Narvaiza, L., Gálvez-Barrón, C., Gonzalo León, N., Valldosera, E., de Mingo, E., Macho, O., Aivar, D., Pinzón, E., Alba, A., Passarelli, J., Stasi, N., Valverde, R.A., Kruse, L., Felipe, E., Collado, I., Sabater, J.B., 2019. The spatial

- parameters of gait and their association with falls, functional decline and death in older adults: a prospective study. Sci Rep 9, 8813. https://doi.org/10.1038/s41598-019-45113-2
- Rush, A.J., Trivedi, M.H., Ibrahim, H.M., Carmody, T.J., Arnow, B., Klein, D.N., Markowitz, J.C., Ninan, P.T., Kornstein, S., Manber, R., Thase, M.E., Kocsis, J.H., Keller, M.B., 2003. The 16-Item quick inventory of depressive symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biological Psychiatry 54, 573–583. https://doi.org/10.1016/S0006-3223(02)01866-8
- Schwab, R.S., England, A.C., 1969. Projection techniques for evaluating surgery in Parkinson's Disease. Third Symposium on Parkinson's Disease, Royal College of Surgeons in Edinburgh. E. & S. Livingstone Ltd. 152–157.
- Shen, X., Wong-Yu, I.S.K., Mak, M.K.Y., 2016. Effects of Exercise on Falls, Balance, and Gait Ability in Parkinson's Disease: A Meta-analysis. Neurorehabil Neural Repair 30, 512–527. https://doi.org/10.1177/1545968315613447
- Sockeel, P., 2006. The Lille apathy rating scale (LARS), a new instrument for detecting and quantifying apathy: validation in Parkinson's disease. Journal of Neurology, Neurosurgery & Psychiatry 77, 579–584. https://doi.org/10.1136/jnnp.2005.075929
- Spillantini, M.G., Schmidt, M.L., Lee, V.M.-Y., Trojanowski, J.Q., Jakes, R., Goedert, M., 1997. α-Synuclein in Lewy bodies. Nature 388, 839–840. https://doi.org/10.1038/42166
- Spitzer, R.L., Kroenke, K., Williams, J.B.W., Löwe, B., 2006. A Brief Measure for Assessing Generalized Anxiety Disorder: The GAD-7. Arch Intern Med 166, 1092. https://doi.org/10.1001/archinte.166.10.1092
- Tomlinson, C.L., Patel, S., Meek, C., Herd, C.P., Clarke, C.E., Stowe, R., Shah, L., Sackley, C.M., Deane, K.H., Wheatley, K., Ives, N., 2013. Physiotherapy versus placebo or no intervention in Parkinson's disease. Cochrane Database of Systematic Reviews. https://doi.org/10.1002/14651858.CD002817.pub4
- Van Den Eeden, S.K., Tanner, C.M., Bernstein, A.L., Fross, R.D., Leimpeter, A., Bloch, D.A., Nelson, L.M., 2003. Incidence of Parkinson's Disease: Variation by Age, Gender, and Race/Ethnicity. American Journal of Epidemiology 157, 1015–1022. https://doi.org/10.1093/aje/kwg068
- van der Kolk, N.M., King, L.A., 2013. Effects of exercise on mobility in people with Parkinson's disease. Movement Disorders 28, 1587–1596. https://doi.org/10.1002/mds.25658
- Vellata, C., Belli, S., Balsamo, F., Giordano, A., Colombo, R., Maggioni, G., 2021. Effectiveness of Telerehabilitation on Motor Impairments, Non-motor Symptoms and Compliance in Patients With Parkinson's Disease: A Systematic Review. Frontiers in Neurology 12, 1394. https://doi.org/10.3389/fneur.2021.627999
- Verghese, J., Holtzer, R., Lipton, R.B., Wang, C., 2009. Quantitative Gait Markers and Incident Fall Risk in Older Adults. The Journals of Gerontology Series A: Biological Sciences and Medical Sciences 64A, 896–901. https://doi.org/10.1093/gerona/glp033
- Vergier, N., Chaput, H., 2017. Déserts médicaux : comment les définir ? Comment les mesurer ? Les Dossiers de la Drees.
- Wood, B.H., Bilclough, J.A., Bowron, A., Walker, R.W., 2002. Incidence and prediction of falls in Parkinson's disease: a prospective multidisciplinary study. J Neurol Neurosurg Psychiatry 72, 721–725. https://doi.org/10.1136/jnnp.72.6.721
- Yalcin, I., Bump, R.C., 2003. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol 189, 98–101. https://doi.org/10.1067/mob.2003.379
- Yogev, G., Giladi, N., Peretz, C., Springer, S., Simon, E.S., Hausdorff, J.M., 2005. Dual tasking, gait rhythmicity, and Parkinson's disease: Which aspects of gait are attention demanding? European Journal of Neuroscience 22, 1248–1256. https://doi.org/10.1111/j.1460-9568.2005.04298.x